CLINICAL TRIAL: NCT03622580
Title: A Phase III, Multicenter, Randomized, Double-Masked, Active Comparator-Controlled Study to Evaluate the Efficacy and Safety of Faricimab (RO6867461) in Patients With Diabetic Macular Edema (YOSEMITE)
Brief Title: A Study to Evaluate the Efficacy and Safety of Faricimab (RO6867461) in Participants With Diabetic Macular Edema (YOSEMITE)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GR40349; 2017-005104-10 (EudraCT Number)
Record Dates: First submitted 2018-08-01; First posted 2018-08-09 (Actual); Results first posted 2022-03-22 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — aflibercept; faricimab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- A: Faricimab 6 mg Q8W (Experimental): Participants randomized to Arm A received 6 milligrams (mg) faricimab intravitreal (IVT) injections once every 4 weeks (Q4W) to Week 20, followed by 6 mg faricimab IVT injections once every 8 weeks (Q8W) to Week 96, followed by the final study visit at Week 100.
  Interventions: Drug: Faricimab; Procedure: Sham Procedure
- B: Faricimab 6 mg PTI (Experimental): Participants randomized to Arm B received 6 milligrams (mg) faricimab intravitreal (IVT) injections Q4W to at least Week 12, followed by a personalized treatment interval (PTI) dosing of 6 mg faricimab IVT injections once every 4 weeks (Q4W), 8 weeks (Q8W), 12 weeks (Q12W), or 16 weeks (Q16W) up to Week 96, followed by the final study visit at Week 100.
  Interventions: Drug: Faricimab; Procedure: Sham Procedure
- C: Aflibercept 2 mg Q8W (Active Comparator): Participants randomized to Arm C received 2 milligrams (mg) aflibercept intravitreal (IVT) injections Q4W to Week 16, followed by 2 mg aflibercept IVT injections Q8W to Week 96, followed by the final study visit at Week 100.
  Interventions: Drug: Aflibercept; Procedure: Sham Procedure

INTERVENTIONS:
Drug: Aflibercept — Aflibercept 2 mg was administered by intravitreal (IVT) injection into the study eye once every 8 weeks (Q8W).
  Other Names: Eylea
  Arms: C: Aflibercept 2 mg Q8W
Drug: Faricimab — Faricimab 6 mg was administered by IVT injection into the study eye either once every 8 weeks (Q8W) in arm A or according to a personalized treatment interval (PTI) in arm B.
  Other Names: VABYSMO™; RO6867461; RG7716
  Arms: A: Faricimab 6 mg Q8W; B: Faricimab 6 mg PTI
Procedure: Sham Procedure — The sham is a procedure that mimics an IVT injection and involves the blunt end of an empty syringe (without a needle) being pressed against the anesthetized eye. It was administered to participants in all three treatments arms at applicable clinic visits to maintain masking among treatment arms.

SUMMARY:
This study will evaluate the efficacy, safety, and pharmacokinetics of faricimab administered at 8-week intervals or as specified in the protocol following treatment initiation, compared with aflibercept once every 8 weeks (Q8W), in participants with diabetic macular edema (DME).

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of diabetes mellitus (Type 1 or Type 2)
* Hemoglobin A1c (HbA1c) of less than or equal to (≤) 10% within 2 months prior to Day 1
* Macular thickening secondary to diabetic macular edema (DME) involving the center of the fovea
* Decreased visual acuity attributable primarily to DME
* Ability and willingness to undertake all scheduled visits and assessments
* For women of childbearing potential: agreement to remain abstinent or use acceptable contraceptive methods that result in a failure rate of <1% per year during the treatment period and for at least 3 months after the final dose of study treatment

Exclusion Criteria:

* Currently untreated diabetes mellitus or previously untreated patients who initiated oral or injectable anti-diabetic medication within 3 months prior to Day 1
* Uncontrolled blood pressure, defined as a systolic value greater than (>)180 millimeters of mercury (mmHg) and/or a diastolic value >100 mmHg while a patient is at rest
* Currently pregnant or breastfeeding, or intend to become pregnant during the study
* Treatment with panretinal photocoagulation or macular laser within 3 months prior to Day 1 to the study eye
* Any intraocular or periocular corticosteroid treatment within the past 6 months prior to Day 1 to the study eye
* Prior administration of IVT faricimab in either eye
* Active intraocular or periocular infection or active intraocular inflammation in the study eye
* Any current or history of ocular disease other than DME that may confound assessment of the macula or affect central vision in the study eye
* Any current ocular condition which, in the opinion of the investigator, is currently causing or could be expected to contribute to irreversible vision loss due to a cause other than DME in the study eye
* Other protocol-specified inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 940 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2021-09-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (185):
- United States (85):
  - Barnet Dulaney Perkins Eye Center, Mesa, Arizona
  - Arizona Retina and Vitreous Consultants, Phoenix, Arizona
  - Retina Associates Southwest PC, Tucson, Arizona
  - Retinal Diagnostic Center, Campbell, California
  - Eye Medical Center, Fresno, California
  - East Bay Retina Consultants, Oakland, California
  - Southern CA Desert Retina Cons, Palm Desert, California
  - California Eye Specialists Medical group Inc., Pasadena, California
  - Retina Consultants, San Diego, Poway, California
  - Retina Consultants of Southern California, Redlands, California
  - Kaiser Permanente Riverside Medical Center, Riverside, California
  - University of California, Davis, Eye Center, Sacramento, California
  - W Coast Retina Med Group Inc, San Francisco, California
  - Orange County Retina Med Group, Santa Ana, California
  - Colorado Retina Associates, PC, Lakewood, Colorado
  - Rand Eye, Deerfield Beach, Florida
  - Retina Care Specialists, Palm Beach Gardens, Florida
  - Retina Specialty Institute, Pensacola, Florida
  - Southern Vitreoretinal Assoc, Tallahassee, Florida
  - Retina Associates of Florida, LLC, Tampa, Florida
  - University of South Florida, Tampa, Florida
  - Georgia Retina PC, Marietta, Georgia
  - Retina Consultants of Hawaii, ‘Aiea, Hawaii
  - Midwest Eye Institute, Indianapolis, Indiana
  - Wolfe Eye Clinic, West Des Moines, Iowa
  - Retina Associates, Lenexa, Kansas
  - Vitreo-Retinal Consultants, Wichita, Kansas
  - Retina Associates of Kentucky, Lexington, Kentucky
  - Paducah Retinal Center, Paducah, Kentucky
  - Maine Eye Center, Portland, Maine
  - The Retina Care Center, Baltimore, Maryland
  - Johns Hopkins Med; Wilmer Eye Inst, Baltimore, Maryland
  - Retina Group of Washington, Chevy Chase, Maryland
  - Cumberland Valley Retina PC, Hagerstown, Maryland
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Beetham Eye Institute, Joslin Diabetes Center, Boston, Massachusetts
  - Vitreo-Retinal Associates, PC, Worcester, Massachusetts
  - Foundation for Vision Research, Grand Rapids, Michigan
  - Assoc Retinal Consultants PC, Royal Oak, Michigan
  - Associated Retinal Consultants, P.C., Traverse City, Michigan
  - Vitreoretinal Surgery, Edina, Minnesota
  - Midwest Vision Research Foundation, Chesterfield, Missouri
  - Sierra Eye Associates, Reno, Nevada
  - Mid Atlantic Retina - Wills Eye Hospital, Cherry Hill, New Jersey
  - NJ Retina, Edison, New Jersey
  - Retinal & Ophthalmic Cons PC, Northfield, New Jersey
  - Retina Associates of NJ, Teaneck, New Jersey
  - University of New Mexico, Albuquerque, New Mexico
  - Capital Region Retina, Albany, New York
  - Long Is. Vitreoretinal Consult, Great Neck, New York
  - Retina Vit Surgeons/Central NY, Liverpool, New York
  - MaculaCare, PLLC, New York, New York
  - Island Retina, Shirley, New York
  - Western Carolina Retinal Associate PA, Asheville, North Carolina
  - Char Eye Ear &Throat Assoc, Charlotte, North Carolina
  - Graystone Eye, Hickory, North Carolina
  - Carolina Eye Associates, Southern Pines, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - Retina Assoc of Cleveland Inc, Cleveland, Ohio
  - OSU Eye Physicians & Surgeons, Columbus, Ohio
  - Midwest Retina, Dublin, Ohio
  - Retina Vitreous Center, Edmond, Oklahoma
  - Retina Northwest, Portland, Oregon
  - Black Hills Eye Institute, Rapid City, South Dakota
  - Charles Retina Institute, Memphis, Tennessee
  - Retina Res Institute of Texas, Abilene, Texas
  - Austin Clinical Research LLC, Austin, Texas
  - Retina Consultants of Texas, Bellaire, Texas
  - Texas Retina Associates, Dallas, Texas
  - Retina Specialists, DeSoto, Texas
  - Valley Retina Institute P.A., Harlingen, Texas
  - Retina & Vitreous of Texas, Houston, Texas
  - Med Center Ophthalmology Assoc, San Antonio, Texas
  - Eye Care Assoc of East Texas, Tyler, Texas
  - Strategic Clinical Research Group, LLC, Willow Park, Texas
  - Retina Associates of Utah, Salt Lake City, Utah
  - University of Utah; Division of Gastroenterology/Hepatology, Salt Lake City, Utah
  - University of Vermont Medical Center; Investigational Drug Service, Pharmacy Department/Baird 1, Burlington, Vermont
  - Emerson Clinical Research Institute, Falls Church, Virginia
  - Piedmont Eye Center, Lynchburg, Virginia
  - Wagner Macula & Retina Center, Norfolk, Virginia
  - Spokane Eye Clinical Research, Spokane, Washington
  - West Virginia University Eye Institute, Morgantown, West Virginia
  - University of Wisconsin, Madison, Wisconsin
- Austria (4):
  - LKH-Univ.Klinikum Graz; Universitäts-Augenklinik, Graz
  - Kepler Universitätskliniken GmbH - Med Campus III; Abt. für Augenheilkunde, Linz
  - Medizinische Universität Wien; Universitätsklinik für Augenheilkunde und Optometrie, Vienna
  - Hanusch Krankenhaus; Abteilung für Augenkrankheiten mit Augen-Tagesklinik, Vienna
- Bulgaria (5):
  - Medical Center for Eye Health - Focus Ltd, Sofia
  - Pentagram Eye Hospital (Medical Center "Pentagram"), Sofia
  - Spec. Ophth. Hospital for Active Treatment- Academic Pashev, Sofia
  - Specialized Hospital for Active Treatment of Eye Diseases Zora, Sofia
  - Ambulatory - Medical Center for Specialized Medical Assistance - "Eye Clinic Sveta Petka" Ltd, Varna
- France (6):
  - Hopital Pellegrin; Ophtalmologie, Bordeaux
  - Pole Vision Val d'Ouest; Ophtalmologie, Écully
  - Centre Paradis Monticelli; Ophtalmologie, Marseille
  - CHU Nantes - Hôtel Dieu; Ophthalmology, Nantes
  - Centre Odeon; Exploration Ophtalmologique, Paris
  - Hopital Lariboisiere; Ophtalmologie, Paris
- Germany (6):
  - Universitäts-Augenklinik Bonn, Bonn
  - Universitätsmedizin Göttingen Georg-August-Universität; Klinik für Augenheilkunde 3.B1.266, Göttingen
  - Medizinische Hochschule Hannover, Klinik für Augenheilkunde, Hanover
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Augenklinik und Poliklinik, Mainz
  - Augenabteilung am St. Franziskus-Hospital, Münster
  - Universitätsklinikum Münster; Augenheilkunde, Münster
- Hungary (6):
  - Budapest Retina Associates Kft., Budapest
  - Debreceni Egyetem Klinikai Kozpont; Szemeszeti Klinika, Debrecen
  - Ganglion Medial Center, Pécs
  - Szegedi Tudományegyetem ÁOK; Department of Ophtalmology, Szeged
  - Markusovszky Egyetemi Oktatokorhaz ; SZEMESZET, Szombathely
  - Zala Megyei Kórház; SZEMESZET, Zalaegerszeg
- Israel (5):
  - Rambam Medical Center; Opthalmology, Haifa
  - Hadassah MC; Ophtalmology, Jerusalem
  - Rabin MC; Ophtalmology, Petah Tikva
  - Kaplan Medical Center, Rehovot
  - Tel Aviv Sourasky MC; Ophtalmology, Tel Aviv
- Italy (6):
  - Ospedale Clinicizzato SS Annunziata; Clinica Oftalmologica, Chieti, Abruzzo
  - Fondazione G.B. Bietti Per Lo Studio E La Ricerca in Oftalmologia-Presidio Ospedaliero Britannico, Rome, Lazio
  - UNIVERSITA' DEGLI STUDI DI GENOVA - Di.N.O.G.;CLINICA OCULISTICA, Genoa, Liguria
  - Fondazione Irccs Ca' Granda Ospedale Maggiore Policlinico-Clinica Regina Elena;U.O.C Oculistica, Milan, Lombardy
  - Irccs Ospedale San Raffaele;U.O. Oculistica, Milan, Lombardy
  - Azienda Ospedaliera di Perugia Ospedale S. Maria Della Misericordia; Clinica Oculistica, Perugia, Umbria
- Japan (27):
  - Sugita Eye Hospital, Aichi
  - Nagoya University Hospital, Aichi
  - Nagoya City University Hospital, Aichi
  - Aichi Medical University Hospital, Aichi
  - Toho University Sakura Medical Center, Chiba
  - Hayashi Eye Hospital, Fukuoka
  - Kurume University Hospital, Fukuoka
  - Hokkaido University Hospital, Hokkaido
  - Asahikawa Medical University Hospital, Hokkaido
  - Hyogo Prefectural Amagasaki General Medical Center (Hyogo AGMC), Hyōgo
  - Kozawa eye hospital and diabetes center, Ibaraki
  - St. Marianna University Hospital, Kanagawa
  - Ideta Eye Hospital, Kumamoto
  - Kyoto University Hospital, Kyoto
  - Mie University Hospital, Mie
  - University of Miyazaki Hospital, Miyazaki
  - Nara Medical University Hospital, Nara
  - Kitano Hospital, Osaka
  - Osaka City University Hospital, Osaka
  - National Defense Medical College Hospital, Saitama
  - Shiga University Of Medical Science Hospital, Shiga
  - Seirei Hamamatsu General Hospital, Shizuoka
  - Tokushima University Hospital, Tokushima
  - Tokyo Women's Medical University Hospital, Tokyo
  - Kyorin University Hospital, Tokyo
  - Tokyo Medical University Hachioji Medical Center, Tokyo
  - Yamaguchi University Hospital, Yamaguchi
- Mexico (4):
  - Centro Oftalmológico Mira, S.C, Cuauhtémoc, Mexico CITY (federal District)
  - Macula Retina Consultores, México
  - Hospital de la Ceguera APEC, México
  - Instituto Mexicano de Oftalmologia I.A.P., Querétaro
- Peru (4):
  - Mácula D&T, Lima
  - Oftalmosalud Srl, Lima
  - TG Laser Oftalmica, Lima
  - Oftalmolaser, Lima
- Poland (8):
  - Szpital sw. Lukasza, Bielsko-Biala
  - Szpital Specjalistyczny nr 1; Oddzial Okulistyki, Bytom
  - Dobry Wzrok Sp Z O O, Gdansk
  - Gabinet Okulistyczny Prof Edward Wylegala, Katowice
  - Centrum Medyczne UNO-MED, Krakow
  - Optomed Sp. z o.o., Rybnik
  - Kliniczny Szpital Wojewodzki nr 1 im. F. Chopina; Klinika Okulistyki, Rzeszów
  - SPEKTRUM Osrodek Okulistyki Klinicznej, Wroclaw
- Russia (3):
  - Clinic Optimed, Ufa, Bashkortostan Republic
  - FSBI "Scientific Research Institute of Eye Diseases" of Russian Academy of medical Sciences, Moscow
  - Medical Military Academy n.a S.M.Kirov, Saint Petersburg
- Slovakia (3):
  - Nemocnica s poliklinikou Trebišov, a.s., Trebišov
  - Fakultna nemocnica Trencin Ocna klinika, Trenčín
  - Fakultna nemocnica s poliklinikou Zilina; Ocne oddelenie, Žilina
- Spain (10):
  - Instituto Oftalmologico Gomez Ulla; Servicio de Oftalmologia, Santiago de Compostela, LA Coruña
  - Hospital Universitario de Gran Canaria; Servicio de oftalmologia, Las Palmas de Gran Canaria, LAS Palmas
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Clinica Universitaria de Navarra; Servicio de Oftalmologia, Pamplona, Navarre
  - Complejo Hospitalario Universitario Albacete; Servicio de oftalmologia, Albacete
  - VISSUM Instituto Oftalmológico de Alicante, Alicante
  - Centro de Oftalmologia Barraquer; Servicio Oftalmologia, Barcelona
  - Hospital Clinic de Barcelona; Consultas Externas Oftalmologia, Barcelona
  - Hospital de Santa Creu I Sant Pau; Servicio de Oftalmologia, Barcelona
  - Clinica Universitaria de Navarra; Servicio de Oftalmologia, Madrid
- Turkey (Türkiye) (3):
  - Hacettepe University Medical Faculty; Department of Ophthalmology, Ankara
  - Ege University Medical Faculty; Department of Ophthalmology, Izmir
  - Selcuk University Faculty of Medicine; Department Of Ophthalmology, Konya

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Result] Wong TY, Haskova Z, Asik K, Baumal CR, Csaky KG, Eter N, Ives JA, Jaffe GJ, Korobelnik JF, Lin H, Murata T, Ruamviboonsuk P, Schlottmann PG, Seres AI, Silverman D, Sun X, Tang Y, Wells JA, Yoon YH, Wykoff CC; YOSEMITE and RHINE Investigators. Faricimab Treat-and-Extend for Diabetic Macular Edema: Two-Year Results from the Randomized Phase 3 YOSEMITE and RHINE Trials. Ophthalmology. 2024 Jun;131(6):708-723. doi: 10.1016/j.ophtha.2023.12.026. Epub 2023 Dec 28. PMID 38158159
- [Derived] Jaffe GJ, Deak G, Gibson K, Khurana RN, Nudleman E, Ogura Y, Schmidt-Erfurth U, Wang T, Westenskow PD, Wong D, Yiu G, Willis JR. IMPACT OF FARICIMAB VERSUS AFLIBERCEPT ON EPIRETINAL MEMBRANE FORMATION OVER 2 YEARS IN PATIENTS WITH DIABETIC MACULAR EDEMA IN THE PHASE 3 YOSEMITE AND RHINE TRIALS. Retina. 2025 Nov 1;45(11):2003-2011. doi: 10.1097/IAE.0000000000004572. PMID 40668667
- [Derived] Gamble A, Khan T, Hughes A, Guo Y, Vasaitis S, Bidwell J, Christman B. Telehealth Diabetes Prevention Program for Adults With Prediabetes in an Academic Medical Center Setting: Protocol for a Hybrid Type III Trial. JMIR Res Protoc. 2023 Nov 13;12:e50183. doi: 10.2196/50183. PMID 37955955
- [Derived] Stockwell AD, Chang MC, Mahajan A, Forrest W, Anegondi N, Pendergrass RK, Selvaraj S, Reeder J, Wei E, Iglesias VA, Creps NM, Macri L, Neeranjan AN, van der Brug MP, Scales SJ, McCarthy MI, Yaspan BL. Multi-ancestry GWAS analysis identifies two novel loci associated with diabetic eye disease and highlights APOL1 as a high risk locus in patients with diabetic macular edema. PLoS Genet. 2023 Aug 16;19(8):e1010609. doi: 10.1371/journal.pgen.1010609. eCollection 2023 Aug. PMID 37585454
- [Derived] Shimura M, Kitano S, Ogata N, Mitamura Y, Oh H, Ochi H, Ohsawa S, Hirakata A; YOSEMITE and RHINE Investigators. Efficacy, durability, and safety of faricimab with extended dosing up to every 16 weeks in Japanese patients with diabetic macular edema: 1-year results from the Japan subgroup of the phase 3 YOSEMITE trial. Jpn J Ophthalmol. 2023 May;67(3):264-279. doi: 10.1007/s10384-023-00979-8. Epub 2023 Mar 10. PMID 36897413
- [Derived] Eter N, Singh RP, Abreu F, Asik K, Basu K, Baumal C, Chang A, Csaky KG, Haskova Z, Lin H, Ruiz CQ, Ruamviboonsuk P, Silverman D, Wykoff CC, Willis JR. YOSEMITE and RHINE: Phase 3 Randomized Clinical Trials of Faricimab for Diabetic Macular Edema: Study Design and Rationale. Ophthalmol Sci. 2021 Dec 30;2(1):100111. doi: 10.1016/j.xops.2021.100111. eCollection 2022 Mar. PMID 36246184
- [Derived] Wykoff CC, Abreu F, Adamis AP, Basu K, Eichenbaum DA, Haskova Z, Lin H, Loewenstein A, Mohan S, Pearce IA, Sakamoto T, Schlottmann PG, Silverman D, Sun JK, Wells JA, Willis JR, Tadayoni R; YOSEMITE and RHINE Investigators. Efficacy, durability, and safety of intravitreal faricimab with extended dosing up to every 16 weeks in patients with diabetic macular oedema (YOSEMITE and RHINE): two randomised, double-masked, phase 3 trials. Lancet. 2022 Feb 19;399(10326):741-755. doi: 10.1016/S0140-6736(22)00018-6. Epub 2022 Jan 24. PMID 35085503

RESULTS

PARTICIPANT FLOW:
Groups:
- B: Faricimab 6 mg PTI: Participants randomized to Arm B received 6 milligrams (mg) faricimab intravitreal (IVT) injections Q4W to at least Week 12, followed by a personalized treatment interval (PTI) dosing of 6 mg faricimab IVT injections up to once every 16 weeks (Q16W) through Week 96, followed by the final study visit at Week 100.
Period: Overall Study
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Started (Intent-to-Treat (ITT) Population) | 315 | 313 | 312
Received at Least One Dose of Study Drug (Safety-Evaluable Population) | 313 | 313 | 311
Completed up to Week 56 (Primary Completion Date Cutoff) | 291 | 289 | 292
Completed | 263 | 269 | 260
Not Completed | 52 | 44 | 52
Not completed — Death | 16 | 21 | 13
Not completed — Adverse Event | 6 | 6 | 5
Not completed — Withdrawal by Subject | 12 | 7 | 19
Not completed — Lost to Follow-up | 12 | 9 | 9
Not completed — Protocol Violation | 1 | 0 | 1
Not completed — Physician Decision | 3 | 0 | 1
Not completed — Pregnancy | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 0 | 1
Not completed — Other | 2 | 0 | 3

BASELINE CHARACTERISTICS:
Population: The overall number of baseline participants (940) comprises the Intent-to-Treat (ITT) Population, which includes all global participants who were randomized in the study, grouped according to the treatment assigned at randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W | Total
Number analyzed (Participants) | 315 | 313 | 312 | 940
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: The ITT and Treatment-Naive (TN) Populations are grouped according to treatment assigned at randomization. The ITT Population (940) includes all global participants randomized in the study. The TN Population (725), a subset of ITT, includes randomized participants who had not received any IVT anti-VEGF agents in the study eye before randomization.
  Years
    ITT Population | 61.6 (9.5) | 62.8 (10.0) | 62.2 (9.6) | 62.2 (9.7)
    Treatment-Naive Population: number analyzed (Participants) | 238 | 245 | 242 | 725
    Treatment-Naive Population | 61.0 (9.6) | 62.5 (10.3) | 62.2 (9.9) | 61.9 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The ITT and Treatment-Naive (TN) Populations are grouped according to treatment assigned at randomization. The ITT Population (940) includes all global participants randomized in the study. The TN Population (725), a subset of ITT, includes randomized participants who had not received any IVT anti-VEGF agents in the study eye before randomization.
  Participants
    ITT Population: Female | 128 | 116 | 134 | 378
    ITT Population: Male | 187 | 197 | 178 | 562
    Treatment-Naive Population: number analyzed (Participants) | 238 | 245 | 242 | 725
    Treatment-Naive Population: Female | 93 | 91 | 108 | 292
    Treatment-Naive Population: Male | 145 | 154 | 134 | 433
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The ITT and Treatment-Naive (TN) Populations are grouped according to treatment assigned at randomization. The ITT Population (940) includes all global participants randomized in the study. The TN Population (725), a subset of ITT, includes randomized participants who had not received any IVT anti-VEGF agents in the study eye before randomization.
  Participants
    ITT Population: Hispanic or Latino | 37 | 40 | 37 | 114
    ITT Population: Not Hispanic or Latino | 273 | 268 | 272 | 813
    ITT Population: Unknown or Not Reported | 5 | 5 | 3 | 13
    Treatment-Naive Population: number analyzed (Participants) | 238 | 245 | 242 | 725
    Treatment-Naive Population: Hispanic or Latino | 31 | 32 | 31 | 94
    Treatment-Naive Population: Not Hispanic or Latino | 202 | 210 | 208 | 620
    Treatment-Naive Population: Unknown or Not Reported | 5 | 3 | 3 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The ITT and Treatment-Naive (TN) Populations are grouped according to treatment assigned at randomization. The ITT Population (940) includes all global participants randomized in the study. The TN Population (725), a subset of ITT, includes randomized participants who had not received any IVT anti-VEGF agents in the study eye before randomization.
  Participants
    ITT Population: American Indian or Alaska Native | 6 | 5 | 7 | 18
    ITT Population: Asian | 31 | 26 | 27 | 84
    ITT Population: Native Hawaiian or Other Pacific Islander | 2 | 0 | 3 | 5
    ITT Population: Black or African American | 22 | 25 | 12 | 59
    ITT Population: White | 241 | 240 | 253 | 734
    ITT Population: More than one race | 0 | 1 | 0 | 1
    ITT Population: Unknown or Not Reported | 13 | 16 | 10 | 39
    Treatment-Naive Population: number analyzed (Participants) | 238 | 245 | 242 | 725
    Treatment-Naive Population: American Indian or Alaska Native | 4 | 3 | 6 | 13
    Treatment-Naive Population: Asian | 21 | 18 | 20 | 59
    Treatment-Naive Population: Native Hawaiian or Other Pacific Islander | 2 | 0 | 2 | 4
    Treatment-Naive Population: Black or African American | 17 | 24 | 9 | 50
    Treatment-Naive Population: White | 181 | 186 | 196 | 563
    Treatment-Naive Population: More than one race | 0 | 1 | 0 | 1
    Treatment-Naive Population: Unknown or Not Reported | 13 | 13 | 9 | 35
Number of Participants by Previous Treatment Status with Intravitreal Anti-VEGF Agents [Count of Participants; unit: Participants] — The Treatment-Naive Population was defined as all participants randomized in the study who had not received any intravitreal (IVT) anti-VEGF agents in the study eye prior to randomization.
  Participants
    Treatment-Naive | 238 | 245 | 242 | 725
    Previously Treated | 77 | 68 | 70 | 215
Region of Enrollment [Count of Participants; unit: Participants] — Population: The ITT and Treatment-Naive (TN) Populations are grouped according to treatment assigned at randomization. The ITT Population (940) includes all global participants randomized in the study. The TN Population (725), a subset of ITT, includes randomized participants who had not received any IVT anti-VEGF agents in the study eye before randomization.
  Participants
    ITT Population: United States and Canada | 167 | 168 | 168 | 503
    ITT Population: Asia | 21 | 19 | 20 | 60
    ITT Population: Rest of the World | 127 | 126 | 124 | 377
    Treatment-Naive Population: number analyzed (Participants) | 238 | 245 | 242 | 725
    Treatment-Naive Population: United States and Canada | 130 | 134 | 135 | 399
    Treatment-Naive Population: Asia | 14 | 14 | 15 | 43
    Treatment-Naive Population: Rest of the World | 94 | 97 | 92 | 283
Number of Participants by the Eye Chosen as the Study Eye (Left or Right) [Count of Participants; unit: Participants] — Population: The ITT and Treatment-Naive (TN) Populations are grouped according to treatment assigned at randomization. The ITT Population (940) includes all global participants randomized in the study. The TN Population (725), a subset of ITT, includes randomized participants who had not received any IVT anti-VEGF agents in the study eye before randomization.
  Participants
    ITT Population: Left Eye | 150 | 172 | 151 | 473
    ITT Population: Right Eye | 165 | 141 | 161 | 467
    Treatment-Naive Population: number analyzed (Participants) | 238 | 245 | 242 | 725
    Treatment-Naive Population: Left Eye | 117 | 130 | 117 | 364
    Treatment-Naive Population: Right Eye | 121 | 115 | 125 | 361
Baseline Best Corrected Visual Acuity (BCVA) Letter Score in the Study Eye [Mean (Standard Deviation); unit: ETDRS Letters] — Best corrected visual acuity (BCVA) was measured at a starting test distance of 4 meters using a set of three Precision VisionTM or Lighthouse distance acuity charts (modified ETDRS Charts 1, 2, and R). The BCVA letter score ranges from 0 to 100 (best score attainable), with a higher score indicating better visual acuity. Population: The ITT and Treatment-Naive (TN) Populations are grouped according to treatment assigned at randomization. The ITT Population (940) includes all global participants randomized in the study. The TN Population (725), a subset of ITT, includes randomized participants who had not received any IVT anti-VEGF agents in the study eye before randomization.
  ETDRS Letters
    ITT Population | 62.0 (9.9) | 61.9 (10.2) | 62.2 (9.5) | 62.0 (9.9)
    Treatment-Naive Population: number analyzed (Participants) | 238 | 245 | 242 | 725
    Treatment-Naive Population | 62.3 (9.9) | 61.8 (10.7) | 62.6 (9.2) | 62.2 (9.9)
Number of Participants by the Baseline BCVA Letter Score Categories in the Study Eye [Count of Participants; unit: Participants] — Best corrected visual acuity (BCVA) was measured at a starting test distance of 4 meters using a set of three Precision VisionTM or Lighthouse distance acuity charts (modified ETDRS Charts 1, 2, and R). The BCVA letter score ranges from 0 to 100 (best score attainable), with a higher score indicating better visual acuity. Population: The ITT and Treatment-Naive (TN) Populations are grouped according to treatment assigned at randomization. The ITT Population (940) includes all global participants randomized in the study. The TN Population (725), a subset of ITT, includes randomized participants who had not received any IVT anti-VEGF agents in the study eye before randomization.
  Participants
    ITT Population: ≤38 Letters | 15 | 12 | 12 | 39
    ITT Population: 39 to 63 Letters | 132 | 126 | 132 | 390
    ITT Population: ≥64 Letters | 168 | 175 | 168 | 511
    ITT Population: Missing/Invalid BCVA | 0 | 0 | 0 | 0
    Treatment-Naive Population: number analyzed (Participants) | 238 | 245 | 242 | 725
    Treatment-Naive Population: ≤38 Letters | 10 | 11 | 8 | 29
    Treatment-Naive Population: 39 to 63 Letters | 98 | 95 | 100 | 293
    Treatment-Naive Population: ≥64 Letters | 130 | 139 | 134 | 403
    Treatment-Naive Population: Missing/Invalid BCVA | 0 | 0 | 0 | 0
Number of Participants by Baseline Diabetic Retinopathy Severity (DRS) Status in the Study Eye [Count of Participants; unit: Participants] — The Early Treatment Diabetic Retinopathy Study (ETDRS) Diabetic Retinopathy Severity Scale (DRSS) classifies diabetic retinopathy into 12 severity steps ranging from absence of retinopathy to advanced proliferative diabetic retinopathy. Ocular imaging assessments were made independently by a central reading center. Population: The ITT and Treatment-Naive (TN) Populations are grouped according to treatment assigned at randomization. The ITT Population (940) includes all global participants randomized in the study. The TN Population (725), a subset of ITT, includes randomized participants who had not received any IVT anti-VEGF agents in the study eye before randomization.
  Participants
    ITT Population: 1 - Diabetic Retinopathy (DR) Absent | 2 | 3 | 4 | 9
    ITT Population: 2 - DR Questionable / Microaneurysms Only | 4 | 6 | 10 | 20
    ITT Population: 3 - Mild Non-Proliferative Diabetic Retinopathy (NPDR) | 84 | 92 | 83 | 259
    ITT Population: 4 - Moderate NPDR | 84 | 86 | 85 | 255
    ITT Population: 5 - Moderately Severe NPDR | 67 | 59 | 54 | 180
    ITT Population: 6 - Severe NPDR | 46 | 40 | 49 | 135
    ITT Population: 7 - Mild Proliferative Diabetic Retinopathy (PDR) | 16 | 11 | 9 | 36
    ITT Population: 8 - Moderate PDR | 6 | 9 | 7 | 22
    ITT Population: 9 - High Risk PDR (DRS Level 71) | 0 | 1 | 2 | 3
    ITT Population: 10 - High Risk PDR (DRS Level 75) | 0 | 0 | 0 | 0
    ITT Population: 11 - Advanced PDR (DRS Level 81) | 0 | 0 | 0 | 0
    ITT Population: 12 - Advanced PDR (DRS Level 85) | 0 | 0 | 0 | 0
    ITT Population: Cannot Grade | 4 | 5 | 7 | 16
    ITT Population: Missing | 2 | 1 | 2 | 5
    Treatment-Naive Population: number analyzed (Participants) | 238 | 245 | 242 | 725
    Treatment-Naive Population: 1 - Diabetic Retinopathy (DR) Absent | 2 | 3 | 2 | 7
    Treatment-Naive Population: 2 - DR Questionable / Microaneurysms Only | 1 | 4 | 4 | 9
    Treatment-Naive Population: 3 - Mild Non-Proliferative Diabetic Retinopathy (NPDR) | 65 | 66 | 57 | 188
    Treatment-Naive Population: 4 - Moderate NPDR | 56 | 58 | 65 | 179
    Treatment-Naive Population: 5 - Moderately Severe NPDR | 50 | 52 | 48 | 150
    Treatment-Naive Population: 6 - Severe NPDR | 40 | 38 | 46 | 124
    Treatment-Naive Population: 7 - Mild Proliferative Diabetic Retinopathy (PDR) | 13 | 9 | 6 | 28
    Treatment-Naive Population: 8 - Moderate PDR | 6 | 9 | 6 | 21
    Treatment-Naive Population: 9 - High Risk PDR (DRS Level 71) | 0 | 0 | 2 | 2
    Treatment-Naive Population: 10 - High Risk PDR (DRS Level 75) | 0 | 0 | 0 | 0
    Treatment-Naive Population: 11 - Advanced PDR (DRS Level 81) | 0 | 0 | 0 | 0
    Treatment-Naive Population: 12 - Advanced PDR (DRS Level 85) | 0 | 0 | 0 | 0
    Treatment-Naive Population: Cannot Grade | 4 | 5 | 5 | 14
    Treatment-Naive Population: Missing | 1 | 1 | 1 | 3
Baseline Central Subfield Thickness in the Study Eye [Mean (Standard Deviation); unit: microns] — Central subfield thickness (CST) was defined as the distance between the internal limiting membrane (ILM) and Bruch's membrane (BM) as assessed by a central reading center. Population: The ITT Population (940) includes all global participants randomized in the study. The TN Population (725), ITT subset, includes randomized participants who had not received any IVT anti-VEGF agents in the study eye before randomization. 8 participants in the ITT (3, 1, and 4 in Arms A, B, and C) were excluded for missing or ungradable assessments.
  microns
    ITT Population: number analyzed (Participants) | 312 | 312 | 308 | 932
    ITT Population | 492.3 (135.8) | 485.8 (130.8) | 484.5 (131.1) | 487.5 (132.5)
    Treatment-Naive Population: number analyzed (Participants) | 235 | 244 | 238 | 717
    Treatment-Naive Population | 488.8 (136.8) | 483.5 (127.3) | 486.8 (130.4) | 486.3 (131.3)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in BCVA in the Study Eye Averaged Over Weeks 48, 52, and 56, ITT and Treatment-Naive Populations
Description: Best Corrected Visual Acuity (BCVA) was measured on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart at a starting distance of 4 meters. The BCVA letter score ranges from 0 to 100 (best score), and a gain in BCVA letter score from baseline indicates an improvement in visual acuity. For the Mixed Model for Repeated Measures (MMRM) analysis, the model adjusted for treatment arm, visit, visit-by-treatment arm interaction, baseline BCVA (continuous), baseline BCVA (<64 vs. ≥64 letters), prior intravitreal anti-VEGF therapy (yes vs. no), and region of enrollment. An unstructured covariance structure was used. Treatment policy strategy (i.e., all observed values used) and hypothetical strategy (i.e., all values censored after the occurrence of the intercurrent event) were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were implicitly imputed by MMRM. Invalid BCVA values were excluded. 97.5% CI is a rounding of 97.52% CI.
Time Frame: From Baseline through Week 56
Population: ITT Population and Treatment-Naive Population
Measure: Mean (97.5% Confidence Interval); unit: ETDRS Letters
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 315 | 313 | 312
ETDRS Letters
  ITT Population | 10.7 [9.4 to 12.0] | 11.6 [10.3 to 12.9] | 10.9 [9.6 to 12.2]
  Treatment-Naive Population: number analyzed (Participants) | 238 | 245 | 242
  Treatment-Naive Population | 10.6 [9.1 to 12.1] | 11.4 [9.9 to 12.8] | 11.3 [9.8 to 12.8]
Statistical Analysis 1: Comparison: A: Faricimab 6 mg Q8W vs C: Aflibercept 2 mg Q8W; Three hypotheses were tested in order for each faricimab arm (Q8W or PTI) separately against the aflibercept arm using a graph-based testing procedure. The analysis presented here is for the non-inferiority of Arm A: Faricimab 6 mg Q8W compared with Arm C: Aflibercept 2 mg Q8W in the ITT Population; Test type: Non-Inferiority — If the lower bound of the two-sided 97.52% confidence interval for the difference in adjusted means for the faricimab 6 mg Q8W and the active comparator (aflibercept 2 mg Q8W) arms was greater than -4 letters, then faricimab 6 mg Q8W was considered non-inferior to aflibercept 2 mg Q8W. Non-inferiority was tested one-sided at a significance level of α = 0.0248; Adjusted mean difference = -0.2, 97.5% CI 2-sided [-2.0 to 1.6], Standard Error of Mean 0.79 — The difference in adjusted means was calculated as Arm A: Faricimab 6 mg Q8W minus Arm C: Aflibercept 2 mg Q8W in the ITT Population
Statistical Analysis 2: Comparison: B: Faricimab 6 mg PTI vs C: Aflibercept 2 mg Q8W; Three hypotheses were tested in order for each faricimab arm (Q8W or PTI) separately against the aflibercept arm using a graph-based testing procedure. The analysis presented here is for the non-inferiority of Arm B: Faricimab 6 mg PTI compared with Arm C: Aflibercept 2 mg Q8W in the ITT Population; Test type: Non-Inferiority — If the lower bound of the two-sided 97.52% confidence interval for the difference in adjusted means for the faricimab 6 mg PTI and the active comparator (aflibercept 2 mg Q8W) arms was greater than -4 letters, then faricimab 6 mg PTI was considered non-inferior to aflibercept 2 mg Q8W. Non-inferiority was tested one-sided at a significance level of α = 0.0248; Adjusted mean difference = 0.7, 97.5% CI 2-sided [-1.1 to 2.5], Standard Error of Mean 0.79 — The difference in adjusted means was calculated as Arm B: Faricimab 6 mg PTI minus Arm C: Aflibercept 2 mg Q8W in the ITT Population
Statistical Analysis 3: Comparison: A: Faricimab 6 mg Q8W vs C: Aflibercept 2 mg Q8W; Three hypotheses were tested in order for each faricimab arm (Q8W or PTI) separately against the aflibercept arm using a graph-based testing procedure. The analysis presented here is for the superiority of Arm A: Faricimab 6 mg Q8W compared with Arm C: Aflibercept 2 mg Q8W in the Treatment-Naive Population; Test type: Superiority; p = 0.4699, Mixed Model for Repeated Measures — Tested at an overall significance level of α = 0.0248; Adjusted mean difference = -0.7, 97.5% CI 2-sided [-2.8 to 1.4], Standard Error of Mean 0.95 — The difference in adjusted means was calculated as Arm A: Faricimab 6 mg Q8W minus Arm C: Aflibercept 2 mg Q8W in the Treatment-Naive Population
Statistical Analysis 4: Comparison: B: Faricimab 6 mg PTI vs C: Aflibercept 2 mg Q8W; Three hypotheses were tested in order for each faricimab arm (Q8W or PTI) separately against the aflibercept arm using a graph-based testing procedure. The analysis presented here is for the superiority of Arm B: Faricimab 6 mg PTI compared with Arm C: Aflibercept 2 mg Q8W in the Treatment-Naive Population; Test type: Superiority; p = 0.9650, Mixed Model for Repeated Measures — Tested at an overall significance level of α = 0.0248; Adjusted mean difference = 0.0, 97.5% CI 2-sided [-2.1 to 2.2], Standard Error of Mean 0.94 — The difference in adjusted means was calculated as Arm B: Faricimab 6 mg PTI minus Arm C: Aflibercept 2 mg Q8W in the Treatment-Naive Population
Statistical Analysis 5: Comparison: A: Faricimab 6 mg Q8W vs C: Aflibercept 2 mg Q8W; Three hypotheses were tested in order for each faricimab arm (Q8W or PTI) separately against the aflibercept arm using a graph-based testing procedure. The analysis presented here is for the superiority of Arm A: Faricimab 6 mg Q8W compared with Arm C: Aflibercept 2 mg Q8W in the ITT Population; Test type: Superiority; p = 0.7967, Mixed Model for Repeated Measures — Tested at an overall significance level of α = 0.0248; Adjusted mean difference = -0.2, 97.5% CI 2-sided [-2.0 to 1.6], Standard Error of Mean 0.79 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: B: Faricimab 6 mg PTI vs C: Aflibercept 2 mg Q8W; Three hypotheses were tested in order for each faricimab arm (Q8W or PTI) separately against the aflibercept arm using a graph-based testing procedure. The analysis presented here is for the superiority of Arm B: Faricimab 6 mg PTI compared with Arm C: Aflibercept 2 mg Q8W in the ITT Population; Test type: Superiority; p = 0.3772, Mixed Model for Repeated Measures — Tested at an overall significance level of α = 0.0248; Adjusted mean difference = 0.7, 97.5% CI 2-sided [-1.1 to 2.5], Standard Error of Mean 0.79 — [estimate comment as in outcome 1, analysis 2]

2. Secondary Outcome: Percentage of Participants With a ≥2-Step Diabetic Retinopathy Severity Improvement From Baseline on the ETDRS Diabetic Retinopathy Severity Scale at Week 52, ITT and Treatment-Naive Populations
Description: The Early Treatment Diabetic Retinopathy Study (ETDRS) Diabetic Retinopathy Severity Scale (DRSS) classifies diabetic retinopathy into 12 severity steps ranging from absence of retinopathy to advanced proliferative diabetic retinopathy. Ocular imaging assessments were made independently by a central reading center. The weighted estimates of the percentage of participants were based on the Cochran-Mantel Haenszel (CMH) weights stratified by baseline BCVA (≥64 vs. <64 letters), prior IVT anti-VEGF therapy (yes vs. no), and region (U.S. and Canada vs. rest of the world; Asia and rest of the world regions were combined). Treatment policy strategy (i.e., all observed values used) and hypothetical strategy (i.e., all values censored after the occurrence of the intercurrent event) were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were not imputed. 97.5% confidence interval (CI) is a rounding of 97.52% CI.
Time Frame: Baseline and Week 52
Population: ITT Population and Treatment-Naive Population. Only participants with non-missing, valid assessments at Baseline and Week 52 were included in the analysis.
Measure: Number (97.5% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 237 | 242 | 229
Percentage of participants
  ITT Population | 46.0 [38.8 to 53.1] | 42.5 [35.5 to 49.5] | 35.8 [29.1 to 42.5]
  Treatment-Naive Population: number analyzed (Participants) | 173 | 187 | 179
  Treatment-Naive Population | 49.7 [41.2 to 58.2] | 47.6 [39.5 to 55.8] | 42.5 [34.4 to 50.6]
Statistical Analysis 1: Comparison: A: Faricimab 6 mg Q8W vs C: Aflibercept 2 mg Q8W; The analysis presented here is for the non-inferiority of Arm A: Faricimab 6 mg Q8W compared with Arm C: Aflibercept 2 mg Q8W in the ITT Population; Test type: Non-Inferiority — If the lower bound of the two-sided 97.52% confidence interval for the difference in CMH weighted percentages of participants for the faricimab 6 mg Q8W and the active comparator (aflibercept 2 mg Q8W) arms was greater than -10%, then faricimab 6 mg Q8W was considered non-inferior to aflibercept 2 mg Q8W; Difference in CMH Weighted Percentage = 10.2, 97.5% CI 2-sided [0.3 to 20.0]
Statistical Analysis 2: Comparison: B: Faricimab 6 mg PTI vs C: Aflibercept 2 mg Q8W; The analysis presented here is for the non-inferiority of Arm B: Faricimab 6 mg PTI compared with Arm C: Aflibercept 2 mg Q8W in the ITT Population; Test type: Non-Inferiority — If the lower bound of the two-sided 97.52% confidence interval for the difference in CMH weighted percentages of participants for the faricimab 6 mg PTI and the active comparator (aflibercept 2 mg Q8W) arms was greater than -10%, then faricimab 6 mg PTI was considered non-inferior to aflibercept 2 mg Q8W; Difference in CMH Weighted Percentage = 6.1, 97.5% CI 2-sided [-3.6 to 15.8]
Statistical Analysis 3: Comparison: A: Faricimab 6 mg Q8W vs C: Aflibercept 2 mg Q8W; The analysis presented here is for the superiority of Arm A: Faricimab 6 mg Q8W compared with Arm C: Aflibercept 2 mg Q8W in the Treatment-Naive Population; Test type: Superiority; p = 0.1761, Cochran-Mantel-Haenszel — Tested at an overall significance level of α = 0.0248; Difference in CMH Weighted Percentage = 7.2, 97.5% CI 2-sided [-4.6 to 18.9]
Statistical Analysis 4: Comparison: B: Faricimab 6 mg PTI vs C: Aflibercept 2 mg Q8W; The analysis presented here is for the superiority of Arm B: Faricimab 6 mg PTI compared with Arm C: Aflibercept 2 mg Q8W in the Treatment-Naive Population; Test type: Superiority; p = 0.3539, Cochran-Mantel-Haenszel — Tested at an overall significance level of α = 0.0248; Difference in CMH Weighted Percentage = 4.8, 97.5% CI 2-sided [-6.7 to 16.3]
Statistical Analysis 5: Comparison: A: Faricimab 6 mg Q8W vs C: Aflibercept 2 mg Q8W; The analysis presented here is for the superiority of Arm A: Faricimab 6 mg Q8W compared with Arm C: Aflibercept 2 mg Q8W in the ITT Population; Test type: Superiority; p = 0.0237, Cochran-Mantel-Haenszel — Tested at an overall significance level of α = 0.0248; Difference in CMH Weighted Percentage = 10.2, 97.5% CI 2-sided [0.3 to 20.0]
Statistical Analysis 6: Comparison: B: Faricimab 6 mg PTI vs C: Aflibercept 2 mg Q8W; The analysis presented here is for the superiority of Arm B: Faricimab 6 mg PTI compared with Arm C: Aflibercept 2 mg Q8W in the ITT Population; Test type: Superiority; p = 0.1677, Cochran-Mantel-Haenszel — Tested at an overall significance level of α = 0.0248; Difference in CMH Weighted Percentage = 6.1, 97.5% CI 2-sided [-3.6 to 15.8]

3. Secondary Outcome: Change From Baseline in BCVA in the Study Eye Over Time, ITT Population
Description: Best Corrected Visual Acuity (BCVA) was measured on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart at a starting distance of 4 meters. The BCVA letter score ranges from 0 to 100 (best score), and a gain in BCVA letter score from baseline indicates an improvement in visual acuity. For the Mixed Model for Repeated Measures (MMRM) analysis, the model adjusted for treatment arm, visit, visit-by-treatment arm interaction, baseline BCVA (continuous), baseline BCVA (<64 vs. ≥64 letters), prior intravitreal anti-VEGF therapy (yes vs. no), and region of enrollment. An unstructured covariance structure was used. Treatment policy strategy (i.e., all observed values used) and hypothetical strategy (i.e., all values censored after the occurrence of the intercurrent event) were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were implicitly imputed by MMRM. Invalid BCVA values were excluded. 95% CI is a rounding of 95.04% CI.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96, and 100
Population: ITT Population: all participants who were randomized in the study, grouped according to the treatment assigned at randomization.
Measure: Mean (95% Confidence Interval); unit: ETDRS Letters
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 315 | 313 | 312
ETDRS Letters
  Week 4 | 5.5 [4.8 to 6.3] | 6.7 [6.0 to 7.4] | 6.5 [5.8 to 7.2]
  Week 8 | 7.2 [6.4 to 7.9] | 8.2 [7.4 to 9.0] | 8.1 [7.3 to 8.8]
  Week 12 | 8.2 [7.4 to 9.0] | 9.2 [8.4 to 10.0] | 9.1 [8.3 to 9.9]
  Week 16 | 9.1 [8.2 to 9.9] | 10.0 [9.2 to 10.8] | 9.7 [8.8 to 10.5]
  Week 20 | 9.6 [8.7 to 10.5] | 9.9 [9.0 to 10.8] | 9.8 [8.9 to 10.7]
  Week 24 | 10.2 [9.3 to 11.1] | 11.3 [10.4 to 12.2] | 9.4 [8.5 to 10.3]
  Week 28 | 9.5 [8.6 to 10.5] | 11.0 [10.0 to 11.9] | 10.5 [9.6 to 11.5]
  Week 32 | 10.2 [9.2 to 11.2] | 10.9 [9.9 to 11.9] | 10.2 [9.2 to 11.2]
  Week 36 | 10.1 [9.1 to 11.1] | 11.7 [10.7 to 12.8] | 10.4 [9.4 to 11.4]
  Week 40 | 10.2 [9.1 to 11.2] | 11.4 [10.3 to 12.5] | 10.3 [9.2 to 11.4]
  Week 44 | 9.9 [8.8 to 11.0] | 11.4 [10.3 to 12.5] | 10.7 [9.6 to 11.9]
  Week 48 | 10.5 [9.4 to 11.6] | 11.4 [10.3 to 12.5] | 10.8 [9.7 to 11.9]
  Week 52 | 9.9 [8.7 to 11.1] | 11.0 [9.8 to 12.2] | 10.9 [9.7 to 12.2]
  Week 56 | 10.8 [9.7 to 12.0] | 11.6 [10.4 to 12.8] | 10.6 [9.4 to 11.8]
  Week 60 | 10.3 [9.1 to 11.5] | 12.0 [10.8 to 13.1] | 11.3 [10.1 to 12.5]
  Week 64 | 10.7 [9.5 to 12.0] | 11.5 [10.3 to 12.7] | 10.8 [9.6 to 12.0]
  Week 68 | 10.2 [8.9 to 11.5] | 11.4 [10.1 to 12.6] | 11.3 [10.0 to 12.5]
  Week 72 | 10.4 [9.1 to 11.7] | 11.3 [10.0 to 12.6] | 10.7 [9.4 to 12.0]
  Week 76 | 10.2 [8.8 to 11.6] | 11.5 [10.1 to 12.9] | 11.0 [9.6 to 12.4]
  Week 80 | 10.9 [9.5 to 12.2] | 11.1 [9.8 to 12.4] | 10.9 [9.6 to 12.2]
  Week 84 | 9.9 [8.6 to 11.2] | 11.5 [10.2 to 12.8] | 11.8 [10.5 to 13.1]
  Week 88 | 9.8 [8.4 to 11.2] | 10.9 [9.5 to 12.3] | 11.0 [9.6 to 12.4]
  Week 92 | 10.5 [9.1 to 11.9] | 11.2 [9.9 to 12.6] | 11.5 [10.1 to 12.9]
  Week 96 | 11.1 [9.7 to 12.6] | 10.6 [9.2 to 12.0] | 11.1 [9.7 to 12.5]
  Week 100 | 10.5 [9.1 to 12.0] | 10.4 [9.0 to 11.8] | 11.6 [10.1 to 13.1]

4. Secondary Outcome: Change From Baseline in BCVA in the Study Eye Over Time, Treatment-Naive Population
Description: Best-Corrected Visual Acuity (BCVA) was measured on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart at a starting distance of 4 meters. The BCVA letter score ranges from 0 to 100 (best score attainable), and a gain in BCVA letter score from baseline indicates an improvement in visual acuity. For the Mixed Model for Repeated Measures (MMRM) analysis, the model adjusted for treatment group, visit, visit-by-treatment group interaction, baseline BCVA (continuous), baseline BCVA (<64 vs. ≥64 letters), and region of enrollment. An unstructured covariance structure was used. Treatment policy strategy (i.e., all observed values used) and hypothetical strategy (i.e., all values censored after the occurrence of the intercurrent event) were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were implicitly imputed by MMRM. Invalid BCVA values were excluded from analysis. 95% confidence interval (CI) is a rounding of 95.04% CI.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96, and 100
Population: Treatment-Naive Population: all participants randomized in the study who had not received any intravitreal anti-VEGF agents in the study eye prior to randomization. Participants were grouped according to the treatment assigned at randomization.
Measure: Mean (95% Confidence Interval); unit: ETDRS Letters
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 238 | 245 | 242
ETDRS Letters
  Week 4 | 5.8 [5.0 to 6.7] | 6.8 [6.0 to 7.6] | 6.9 [6.1 to 7.7]
  Week 8 | 7.2 [6.3 to 8.1] | 8.3 [7.4 to 9.2] | 8.7 [7.8 to 9.5]
  Week 12 | 8.5 [7.6 to 9.4] | 9.3 [8.4 to 10.2] | 9.6 [8.7 to 10.5]
  Week 16 | 9.3 [8.4 to 10.3] | 10.0 [9.1 to 10.9] | 10.1 [9.2 to 11.1]
  Week 20 | 9.7 [8.7 to 10.8] | 9.7 [8.6 to 10.7] | 10.3 [9.3 to 11.4]
  Week 24 | 10.5 [9.4 to 11.5] | 11.2 [10.2 to 12.2] | 9.8 [8.7 to 10.8]
  Week 28 | 9.6 [8.5 to 10.7] | 11.0 [9.9 to 12.1] | 11.0 [9.9 to 12.1]
  Week 32 | 10.3 [9.1 to 11.5] | 10.9 [9.8 to 12.1] | 10.6 [9.5 to 11.8]
  Week 36 | 10.3 [9.1 to 11.6] | 11.9 [10.7 to 13.1] | 10.6 [9.4 to 11.8]
  Week 40 | 10.0 [8.7 to 11.3] | 11.4 [10.1 to 12.7] | 10.7 [9.4 to 12.1]
  Week 44 | 10.1 [8.8 to 11.4] | 11.4 [10.1 to 12.7] | 11.3 [10.0 to 12.6]
  Week 48 | 10.3 [9.0 to 11.7] | 11.0 [9.7 to 12.4] | 11.2 [9.8 to 12.5]
  Week 52 | 9.6 [8.2 to 11.1] | 10.7 [9.3 to 12.2] | 11.3 [9.9 to 12.8]
  Week 56 | 10.9 [9.5 to 12.3] | 11.5 [10.1 to 12.8] | 11.0 [9.6 to 12.4]
  Week 60 | 10.1 [8.7 to 11.6] | 12.0 [10.6 to 13.4] | 11.6 [10.2 to 13.0]
  Week 64 | 10.6 [9.1 to 12.1] | 11.5 [10.0 to 13.0] | 11.0 [9.5 to 12.4]
  Week 68 | 10.3 [8.8 to 11.8] | 11.3 [9.8 to 12.8] | 11.4 [9.9 to 12.9]
  Week 72 | 10.2 [8.6 to 11.7] | 11.3 [9.8 to 12.8] | 10.8 [9.3 to 12.4]
  Week 76 | 9.9 [8.2 to 11.6] | 11.4 [9.7 to 13.0] | 10.8 [9.2 to 12.5]
  Week 80 | 10.6 [9.0 to 12.2] | 11.0 [9.4 to 12.6] | 11.1 [9.6 to 12.7]
  Week 84 | 9.6 [8.0 to 11.1] | 11.6 [10.0 to 13.1] | 11.9 [10.3 to 13.4]
  Week 88 | 9.4 [7.7 to 11.1] | 10.8 [9.1 to 12.5] | 10.9 [9.2 to 12.6]
  Week 92 | 10.1 [8.4 to 11.7] | 11.2 [9.5 to 12.8] | 11.6 [10.0 to 13.3]
  Week 96 | 11.1 [9.4 to 12.8] | 10.5 [8.9 to 12.1] | 11.4 [9.7 to 13.0]
  Week 100 | 10.5 [8.8 to 12.3] | 10.5 [8.8 to 12.1] | 11.7 [10.0 to 13.4]

5. Secondary Outcome: Percentage of Participants Gaining Greater Than or Equal to (≥)15, ≥10, ≥5, or ≥0 Letters in BCVA From Baseline in the Study Eye Averaged Over Weeks 48, 52, and 56, ITT Population
Description: BCVA was measured on the ETDRS chart at a starting distance of 4 meters. The BCVA letter score ranges from 0 to 100 (best score), and a gain in BCVA from baseline indicates an improvement in visual acuity. For each participant, an average BCVA value was calculated across the three visits, and this averaged value was then used to determine if the endpoint was met. The results were summarized as the percentage of participants per treatment arm who met the endpoint. The weighted estimates of the percentage of participants were based on the Cochran-Mantel Haenszel (CMH) weights stratified by baseline BCVA (≥64 vs. <64 letters), prior IVT anti-VEGF therapy (yes vs. no), and region (U.S. and Canada vs. rest of the world). Treatment policy strategy and hypothetical strategy were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were not imputed. Invalid BCVA values were excluded. 95% confidence interval (CI) is a rounding of 95.04% CI.
Time Frame: Baseline, average of Weeks 48, 52, and 56
Population: ITT Population: all participants who were randomized in the study, grouped according to the treatment assigned at randomization. Only participants with at least one non-missing, valid assessment at Weeks 48, 52, or 56 were included in the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 271 | 276 | 276
Percentage of participants
  Gaining ≥15 Letters | 29.2 [23.9 to 34.5] | 35.5 [30.1 to 40.9] | 31.8 [26.6 to 37.0]
  Gaining ≥10 Letters | 57.2 [51.3 to 63.1] | 58.3 [52.6 to 64.0] | 57.6 [51.8 to 63.4]
  Gaining ≥5 Letters | 78.9 [74.1 to 83.8] | 79.6 [74.9 to 84.3] | 81.4 [76.9 to 86.0]
  Gaining ≥0 Letters | 91.5 [88.1 to 94.8] | 94.5 [91.8 to 97.2] | 91.4 [88.1 to 94.6]
Statistical Analysis 1: Comparison: A: Faricimab 6 mg Q8W vs C: Aflibercept 2 mg Q8W; This is the difference in percentage of participants gaining ≥15 letters in Arm A: Faricimab 6 mg Q8W minus Arm C: Aflibercept 2 mg Q8W; Test type: Other; Difference in CMH Weighted Percentage = -2.6, 95% CI 2-sided [-10.0 to 4.9]
Statistical Analysis 2: Comparison: B: Faricimab 6 mg PTI vs C: Aflibercept 2 mg Q8W; This is the difference in percentage of participants gaining ≥15 letters in Arm B: Faricimab 6 mg PTI minus Arm C: Aflibercept 2 mg Q8W; Test type: Other; Difference in CMH Weighted Percentage = 3.5, 95% CI 2-sided [-4.0 to 11.1]
Statistical Analysis 3: Comparison: A: Faricimab 6 mg Q8W vs C: Aflibercept 2 mg Q8W; This is the difference in percentage of participants gaining ≥10 letters in Arm A: Faricimab 6 mg Q8W minus Arm C: Aflibercept 2 mg Q8W; Test type: Other; Difference in CMH Weighted Percentage = -0.4, 95% CI 2-sided [-8.6 to 7.9]
Statistical Analysis 4: Comparison: B: Faricimab 6 mg PTI vs C: Aflibercept 2 mg Q8W; This is the difference in percentage of participants gaining ≥10 letters in Arm B: Faricimab 6 mg PTI minus Arm C: Aflibercept 2 mg Q8W; Test type: Other; Difference in CMH Weighted Percentage = 0.7, 95% CI 2-sided [-7.4 to 8.8]
Statistical Analysis 5: Comparison: A: Faricimab 6 mg Q8W vs C: Aflibercept 2 mg Q8W; This is the difference in percentage of participants gaining ≥5 letters in Arm A: Faricimab 6 mg Q8W minus Arm C: Aflibercept 2 mg Q8W; Test type: Other; Difference in CMH Weighted Percentage = -2.5, 95% CI 2-sided [-9.1 to 4.1]
Statistical Analysis 6: Comparison: B: Faricimab 6 mg PTI vs C: Aflibercept 2 mg Q8W; This is the difference in percentage of participants gaining ≥5 letters in Arm B: Faricimab 6 mg PTI minus Arm C: Aflibercept 2 mg Q8W; Test type: Other; Difference in CMH Weighted Percentage = -2.0, 95% CI 2-sided [-8.5 to 4.5]
Statistical Analysis 7: Comparison: A: Faricimab 6 mg Q8W vs C: Aflibercept 2 mg Q8W; This is the difference in percentage of participants gaining ≥0 letters in Arm A: Faricimab 6 mg Q8W minus Arm C: Aflibercept 2 mg Q8W; Test type: Other; Difference in CMH Weighted Percentage = 0.1, 95% CI 2-sided [-4.6 to 4.8]
Statistical Analysis 8: Comparison: B: Faricimab 6 mg PTI vs C: Aflibercept 2 mg Q8W; This is the difference in percentage of participants gaining ≥0 letters in Arm B: Faricimab 6 mg PTI minus Arm C: Aflibercept 2 mg Q8W; Test type: Other; Difference in CMH Weighted Percentage = 3.3, 95% CI 2-sided [-1.0 to 7.5]

6. Secondary Outcome: Percentage of Participants Gaining ≥15 Letters in BCVA From Baseline in the Study Eye Over Time, ITT Population
Description: Best Corrected Visual Acuity (BCVA) was measured on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart at a starting distance of 4 meters. The BCVA letter score ranges from 0 to 100 (best score), and a gain in BCVA letter score from baseline indicates an improvement in visual acuity. The weighted estimates of the percentage of participants were based on the Cochran-Mantel Haenszel (CMH) weights stratified by baseline BCVA (≥64 vs. <64 letters), prior IVT anti-VEGF therapy (yes vs. no), and region (U.S. and Canada vs. rest of the world; Asia and rest of the world were combined). Treatment policy strategy (i.e., all observed values used) and hypothetical strategy (i.e., all values censored after the occurrence of the intercurrent event) were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were not imputed. Invalid BCVA values were excluded from analysis. 95% confidence interval (CI) is a rounding of 95.04% CI.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96, and 100
Population: ITT Population: all participants who were randomized in the study, grouped according to the treatment assigned at randomization. At each timepoint, only participants with non-missing, valid assessments were included in the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 315 | 313 | 312
Percentage of participants
  Week 4: number analyzed (Participants) | 310 | 308 | 306
  Week 4 | 7.7 [4.8 to 10.7] | 13.0 [9.4 to 16.6] | 11.4 [8.0 to 14.9]
  Week 8: number analyzed (Participants) | 309 | 308 | 304
  Week 8 | 13.4 [9.6 to 17.1] | 18.8 [14.8 to 22.9] | 16.7 [12.7 to 20.7]
  Week 12: number analyzed (Participants) | 305 | 303 | 302
  Week 12 | 14.9 [11.0 to 18.9] | 23.1 [18.6 to 27.5] | 22.1 [17.6 to 26.5]
  Week 16: number analyzed (Participants) | 296 | 296 | 299
  Week 16 | 20.4 [15.9 to 24.9] | 27.8 [22.9 to 32.7] | 22.2 [17.7 to 26.8]
  Week 20: number analyzed (Participants) | 294 | 292 | 296
  Week 20 | 25.6 [20.8 to 30.5] | 28.4 [23.4 to 33.4] | 24.0 [19.4 to 28.6]
  Week 24: number analyzed (Participants) | 292 | 293 | 294
  Week 24 | 26.8 [21.8 to 31.8] | 34.2 [29.0 to 39.3] | 25.7 [21.0 to 30.5]
  Week 28: number analyzed (Participants) | 283 | 287 | 284
  Week 28 | 23.5 [18.6 to 28.4] | 31.2 [26.2 to 36.3] | 29.2 [24.3 to 34.2]
  Week 32: number analyzed (Participants) | 267 | 268 | 275
  Week 32 | 28.5 [23.1 to 33.8] | 36.2 [30.7 to 41.7] | 25.8 [21.0 to 30.7]
  Week 36: number analyzed (Participants) | 268 | 268 | 268
  Week 36 | 24.4 [19.3 to 29.5] | 40.2 [34.6 to 45.8] | 32.5 [27.1 to 37.9]
  Week 40: number analyzed (Participants) | 275 | 269 | 263
  Week 40 | 29.7 [24.3 to 35.1] | 37.1 [31.6 to 42.7] | 30.3 [24.9 to 35.6]
  Week 44: number analyzed (Participants) | 268 | 269 | 266
  Week 44 | 29.2 [23.8 to 34.6] | 37.1 [31.7 to 42.6] | 34.9 [29.4 to 40.4]
  Week 48: number analyzed (Participants) | 264 | 266 | 266
  Week 48 | 31.7 [26.1 to 37.2] | 39.6 [33.9 to 45.3] | 34.0 [28.7 to 39.3]
  Week 52: number analyzed (Participants) | 264 | 267 | 253
  Week 52 | 31.2 [25.7 to 36.8] | 37.2 [31.7 to 42.7] | 36.0 [30.3 to 41.6]
  Week 56: number analyzed (Participants) | 260 | 263 | 256
  Week 56 | 38.1 [32.3 to 43.9] | 38.4 [32.7 to 44.0] | 31.5 [26.1 to 36.9]
  Week 60: number analyzed (Participants) | 270 | 261 | 261
  Week 60 | 34.4 [28.8 to 40.0] | 41.3 [35.5 to 47.1] | 35.9 [30.3 to 41.4]
  Week 64: number analyzed (Participants) | 259 | 263 | 263
  Week 64 | 37.5 [31.7 to 43.4] | 41.4 [35.8 to 47.1] | 34.8 [29.1 to 40.5]
  Week 68: number analyzed (Participants) | 251 | 257 | 253
  Week 68 | 37.1 [31.4 to 42.9] | 43.7 [37.9 to 49.6] | 37.1 [31.4 to 42.8]
  Week 72: number analyzed (Participants) | 253 | 257 | 251
  Week 72 | 34.8 [29.1 to 40.6] | 38.2 [32.6 to 43.8] | 35.2 [29.5 to 41.0]
  Week 76: number analyzed (Participants) | 247 | 253 | 251
  Week 76 | 36.6 [30.7 to 42.6] | 44.1 [38.4 to 49.9] | 37.2 [31.3 to 43.1]
  Week 80: number analyzed (Participants) | 247 | 259 | 251
  Week 80 | 39.3 [33.4 to 45.3] | 42.1 [36.5 to 47.8] | 36.9 [31.1 to 42.6]
  Week 84: number analyzed (Participants) | 248 | 260 | 252
  Week 84 | 40.6 [34.5 to 46.6] | 41.5 [35.8 to 47.2] | 38.8 [32.9 to 44.6]
  Week 88: number analyzed (Participants) | 245 | 256 | 247
  Week 88 | 39.2 [33.2 to 45.2] | 39.8 [34.2 to 45.4] | 35.9 [30.1 to 41.6]
  Week 92: number analyzed (Participants) | 248 | 258 | 248
  Week 92 | 39.7 [33.8 to 45.7] | 41.0 [35.3 to 46.6] | 38.8 [33.0 to 44.7]
  Week 96: number analyzed (Participants) | 242 | 259 | 245
  Week 96 | 41.3 [35.1 to 47.4] | 40.2 [34.5 to 45.8] | 38.8 [32.9 to 44.7]
  Week 100: number analyzed (Participants) | 254 | 258 | 247
  Week 100 | 40.2 [34.2 to 46.1] | 40.3 [34.7 to 46.0] | 40.9 [34.9 to 46.9]

7. Secondary Outcome: Percentage of Participants Gaining ≥10 Letters in BCVA From Baseline in the Study Eye Over Time, ITT Population
Description: as for outcome 6
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96, and 100
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 315 | 313 | 312
Percentage of participants
  Week 4: number analyzed (Participants) | 310 | 308 | 306
  Week 4 | 23.9 [19.2 to 28.6] | 31.1 [26.2 to 36.1] | 27.1 [22.2 to 32.0]
  Week 8: number analyzed (Participants) | 309 | 308 | 304
  Week 8 | 30.8 [25.7 to 35.9] | 37.1 [31.8 to 42.3] | 41.0 [35.6 to 46.4]
  Week 12: number analyzed (Participants) | 305 | 303 | 302
  Week 12 | 35.5 [30.2 to 40.8] | 47.5 [42.0 to 53.0] | 46.2 [40.7 to 51.7]
  Week 16: number analyzed (Participants) | 296 | 296 | 299
  Week 16 | 43.7 [38.0 to 49.3] | 48.4 [42.8 to 54.0] | 49.7 [44.1 to 55.3]
  Week 20: number analyzed (Participants) | 294 | 292 | 296
  Week 20 | 45.6 [40.0 to 51.3] | 53.1 [47.6 to 58.6] | 50.3 [44.7 to 56.0]
  Week 24: number analyzed (Participants) | 292 | 293 | 294
  Week 24 | 55.6 [50.0 to 61.2] | 58.6 [53.2 to 64.1] | 48.2 [42.6 to 53.9]
  Week 28: number analyzed (Participants) | 283 | 287 | 284
  Week 28 | 55.6 [49.9 to 61.3] | 57.0 [51.4 to 62.6] | 57.2 [51.6 to 62.9]
  Week 32: number analyzed (Participants) | 267 | 268 | 275
  Week 32 | 56.7 [50.9 to 62.6] | 58.5 [52.8 to 64.2] | 53.1 [47.3 to 58.8]
  Week 36: number analyzed (Participants) | 268 | 268 | 268
  Week 36 | 55.6 [49.7 to 61.5] | 65.5 [60.0 to 71.1] | 55.7 [49.9 to 61.6]
  Week 40: number analyzed (Participants) | 275 | 269 | 263
  Week 40 | 55.7 [49.8 to 61.5] | 60.0 [54.2 to 65.8] | 53.2 [47.2 to 59.2]
  Week 44: number analyzed (Participants) | 268 | 269 | 266
  Week 44 | 55.1 [49.3 to 61.0] | 60.5 [54.7 to 66.2] | 57.2 [51.3 to 63.2]
  Week 48: number analyzed (Participants) | 264 | 266 | 266
  Week 48 | 57.0 [51.0 to 62.9] | 60.2 [54.5 to 65.9] | 61.7 [55.9 to 67.4]
  Week 52: number analyzed (Participants) | 264 | 267 | 253
  Week 52 | 59.9 [54.0 to 65.8] | 59.5 [53.8 to 65.2] | 60.2 [54.3 to 66.2]
  Week 56: number analyzed (Participants) | 260 | 263 | 256
  Week 56 | 63.5 [57.7 to 69.4] | 62.6 [56.9 to 68.3] | 59.0 [53.0 to 64.9]
  Week 60: number analyzed (Participants) | 270 | 261 | 261
  Week 60 | 59.4 [53.5 to 65.2] | 62.6 [56.9 to 68.3] | 60.7 [54.9 to 66.5]
  Week 64: number analyzed (Participants) | 259 | 263 | 263
  Week 64 | 64.9 [59.2 to 70.7] | 60.0 [54.3 to 65.7] | 59.6 [53.8 to 65.5]
  Week 68: number analyzed (Participants) | 251 | 257 | 253
  Week 68 | 60.1 [54.2 to 66.0] | 58.9 [53.1 to 64.7] | 59.4 [53.5 to 65.4]
  Week 72: number analyzed (Participants) | 253 | 257 | 251
  Week 72 | 61.2 [55.2 to 67.1] | 61.0 [55.2 to 66.8] | 56.8 [50.7 to 62.9]
  Week 76: number analyzed (Participants) | 247 | 253 | 251
  Week 76 | 60.1 [54.1 to 66.2] | 67.8 [62.3 to 73.3] | 64.2 [58.3 to 70.0]
  Week 80: number analyzed (Participants) | 247 | 259 | 251
  Week 80 | 64.0 [58.1 to 70.0] | 61.7 [56.1 to 67.4] | 60.5 [54.5 to 66.4]
  Week 84: number analyzed (Participants) | 248 | 260 | 252
  Week 84 | 61.0 [55.0 to 67.0] | 64.4 [58.8 to 70.1] | 64.4 [58.6 to 70.2]
  Week 88: number analyzed (Participants) | 245 | 256 | 247
  Week 88 | 59.6 [53.5 to 65.7] | 59.8 [54.0 to 65.7] | 62.7 [56.9 to 68.5]
  Week 92: number analyzed (Participants) | 248 | 258 | 248
  Week 92 | 63.2 [57.3 to 69.1] | 63.3 [57.6 to 69.0] | 64.6 [58.7 to 70.4]
  Week 96: number analyzed (Participants) | 242 | 259 | 245
  Week 96 | 60.3 [54.1 to 66.4] | 59.7 [53.9 to 65.5] | 62.5 [56.5 to 68.6]
  Week 100: number analyzed (Participants) | 254 | 258 | 247
  Week 100 | 63.0 [57.3 to 68.8] | 60.5 [54.8 to 66.2] | 66.0 [60.1 to 71.8]

8. Secondary Outcome: Percentage of Participants Gaining ≥5 Letters in BCVA From Baseline in the Study Eye Over Time, ITT Population
Description: as for outcome 6
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96, and 100
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 315 | 313 | 312
Percentage of participants
  Week 4: number analyzed (Participants) | 310 | 308 | 306
  Week 4 | 53.6 [48.1 to 59.1] | 62.6 [57.3 to 67.9] | 61.1 [55.7 to 66.5]
  Week 8: number analyzed (Participants) | 309 | 308 | 304
  Week 8 | 64.7 [59.4 to 70.0] | 71.1 [66.1 to 76.0] | 67.6 [62.4 to 72.8]
  Week 12: number analyzed (Participants) | 305 | 303 | 302
  Week 12 | 71.9 [66.9 to 76.9] | 74.3 [69.4 to 79.2] | 75.4 [70.6 to 80.3]
  Week 16: number analyzed (Participants) | 296 | 296 | 299
  Week 16 | 74.9 [70.0 to 79.9] | 81.4 [77.0 to 85.8] | 77.5 [72.7 to 82.2]
  Week 20: number analyzed (Participants) | 294 | 292 | 296
  Week 20 | 78.2 [73.6 to 82.9] | 78.4 [73.7 to 83.1] | 76.4 [71.6 to 81.1]
  Week 24: number analyzed (Participants) | 292 | 293 | 294
  Week 24 | 80.5 [76.0 to 85.0] | 83.3 [79.0 to 87.5] | 71.0 [65.8 to 76.1]
  Week 28: number analyzed (Participants) | 283 | 287 | 284
  Week 28 | 77.4 [72.5 to 82.2] | 81.0 [76.6 to 85.5] | 79.1 [74.4 to 83.8]
  Week 32: number analyzed (Participants) | 267 | 268 | 275
  Week 32 | 79.4 [74.6 to 84.3] | 77.1 [72.2 to 82.0] | 81.3 [76.8 to 85.8]
  Week 36: number analyzed (Participants) | 268 | 268 | 268
  Week 36 | 79.2 [74.4 to 84.1] | 82.6 [78.2 to 87.1] | 78.3 [73.5 to 83.1]
  Week 40: number analyzed (Participants) | 275 | 269 | 263
  Week 40 | 76.3 [71.3 to 81.3] | 84.3 [80.0 to 88.6] | 77.1 [72.0 to 82.2]
  Week 44: number analyzed (Participants) | 268 | 269 | 266
  Week 44 | 80.7 [75.9 to 85.4] | 81.9 [77.3 to 86.4] | 77.9 [73.0 to 82.7]
  Week 48: number analyzed (Participants) | 264 | 266 | 266
  Week 48 | 79.2 [74.4 to 84.1] | 82.0 [77.5 to 86.6] | 79.3 [74.4 to 84.1]
  Week 52: number analyzed (Participants) | 264 | 267 | 253
  Week 52 | 78.4 [73.5 to 83.4] | 78.4 [73.5 to 83.2] | 81.2 [76.4 to 85.9]
  Week 56: number analyzed (Participants) | 260 | 263 | 256
  Week 56 | 83.0 [78.5 to 87.6] | 81.3 [76.6 to 86.0] | 81.4 [76.7 to 86.1]
  Week 60: number analyzed (Participants) | 270 | 261 | 261
  Week 60 | 80.4 [75.7 to 85.1] | 81.3 [76.7 to 85.9] | 81.4 [76.8 to 86.1]
  Week 64: number analyzed (Participants) | 259 | 263 | 263
  Week 64 | 80.2 [75.4 to 85.1] | 80.6 [75.9 to 85.2] | 79.7 [74.9 to 84.5]
  Week 68: number analyzed (Participants) | 251 | 257 | 253
  Week 68 | 79.1 [74.1 to 84.0] | 78.9 [74.0 to 83.8] | 79.1 [74.2 to 84.0]
  Week 72: number analyzed (Participants) | 253 | 257 | 251
  Week 72 | 79.7 [74.8 to 84.6] | 78.1 [73.2 to 83.0] | 80.9 [76.1 to 85.7]
  Week 76: number analyzed (Participants) | 247 | 253 | 251
  Week 76 | 79.9 [74.9 to 84.8] | 78.9 [74.0 to 83.8] | 82.9 [78.3 to 87.5]
  Week 80: number analyzed (Participants) | 247 | 259 | 251
  Week 80 | 81.0 [76.1 to 85.9] | 80.3 [75.5 to 85.0] | 78.3 [73.2 to 83.4]
  Week 84: number analyzed (Participants) | 248 | 260 | 252
  Week 84 | 77.1 [71.9 to 82.3] | 82.0 [77.5 to 86.5] | 82.6 [77.9 to 87.2]
  Week 88: number analyzed (Participants) | 245 | 256 | 247
  Week 88 | 79.3 [74.2 to 84.3] | 80.5 [75.8 to 85.2] | 80.5 [75.6 to 85.5]
  Week 92: number analyzed (Participants) | 248 | 258 | 248
  Week 92 | 81.4 [76.6 to 86.3] | 82.1 [77.5 to 86.7] | 83.2 [78.6 to 87.7]
  Week 96: number analyzed (Participants) | 242 | 259 | 245
  Week 96 | 82.6 [77.8 to 87.3] | 77.4 [72.5 to 82.4] | 81.2 [76.3 to 86.0]
  Week 100: number analyzed (Participants) | 254 | 258 | 247
  Week 100 | 81.1 [76.3 to 85.9] | 77.0 [71.9 to 82.0] | 85.2 [80.9 to 89.6]

9. Secondary Outcome: Percentage of Participants Gaining ≥0 Letters in BCVA From Baseline in the Study Eye Over Time, ITT Population
Description: as for outcome 6
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96, and 100
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 315 | 313 | 312
Percentage of participants
  Week 4: number analyzed (Participants) | 310 | 308 | 306
  Week 4 | 86.1 [82.3 to 90.0] | 90.8 [87.7 to 94.0] | 88.9 [85.4 to 92.3]
  Week 8: number analyzed (Participants) | 309 | 308 | 304
  Week 8 | 89.7 [86.4 to 93.0] | 91.9 [88.8 to 94.9] | 91.1 [87.9 to 94.2]
  Week 12: number analyzed (Participants) | 305 | 303 | 302
  Week 12 | 92.5 [89.6 to 95.4] | 94.7 [92.2 to 97.2] | 92.7 [89.8 to 95.6]
  Week 16: number analyzed (Participants) | 296 | 296 | 299
  Week 16 | 91.2 [88.0 to 94.4] | 94.9 [92.4 to 97.4] | 93.7 [90.9 to 96.4]
  Week 20: number analyzed (Participants) | 294 | 292 | 296
  Week 20 | 93.9 [91.2 to 96.6] | 93.1 [90.2 to 96.0] | 92.2 [89.2 to 95.2]
  Week 24: number analyzed (Participants) | 292 | 293 | 294
  Week 24 | 93.1 [90.2 to 96.0] | 93.8 [91.0 to 96.5] | 89.9 [86.5 to 93.3]
  Week 28: number analyzed (Participants) | 283 | 287 | 284
  Week 28 | 90.4 [87.0 to 93.8] | 94.1 [91.4 to 96.8] | 91.5 [88.3 to 94.6]
  Week 32: number analyzed (Participants) | 267 | 268 | 275
  Week 32 | 92.1 [88.9 to 95.3] | 95.1 [92.6 to 97.7] | 91.3 [88.0 to 94.6]
  Week 36: number analyzed (Participants) | 268 | 268 | 268
  Week 36 | 92.1 [88.9 to 95.3] | 93.2 [90.2 to 96.2] | 90.4 [87.0 to 93.9]
  Week 40: number analyzed (Participants) | 275 | 269 | 263
  Week 40 | 90.9 [87.5 to 94.3] | 94.0 [91.1 to 96.8] | 93.2 [90.2 to 96.2]
  Week 44: number analyzed (Participants) | 268 | 269 | 266
  Week 44 | 91.0 [87.6 to 94.4] | 94.5 [91.8 to 97.2] | 91.0 [87.6 to 94.4]
  Week 48: number analyzed (Participants) | 264 | 266 | 266
  Week 48 | 95.2 [92.6 to 97.7] | 93.7 [90.8 to 96.5] | 91.3 [88.0 to 94.6]
  Week 52: number analyzed (Participants) | 264 | 267 | 253
  Week 52 | 89.8 [86.1 to 93.4] | 91.3 [88.0 to 94.7] | 91.0 [87.5 to 94.5]
  Week 56: number analyzed (Participants) | 260 | 263 | 256
  Week 56 | 91.4 [88.0 to 94.8] | 93.9 [91.0 to 96.7] | 90.6 [87.1 to 94.2]
  Week 60: number analyzed (Participants) | 270 | 261 | 261
  Week 60 | 89.5 [85.9 to 93.2] | 93.5 [90.5 to 96.4] | 92.8 [89.7 to 95.9]
  Week 64: number analyzed (Participants) | 259 | 263 | 263
  Week 64 | 91.3 [87.9 to 94.7] | 92.7 [89.6 to 95.8] | 92.0 [88.7 to 95.2]
  Week 68: number analyzed (Participants) | 251 | 257 | 253
  Week 68 | 92.1 [88.8 to 95.4] | 92.9 [89.8 to 96.0] | 91.9 [88.6 to 95.2]
  Week 72: number analyzed (Participants) | 253 | 257 | 251
  Week 72 | 88.5 [84.6 to 92.5] | 91.9 [88.7 to 95.2] | 90.0 [86.3 to 93.7]
  Week 76: number analyzed (Participants) | 247 | 253 | 251
  Week 76 | 87.8 [83.8 to 91.9] | 91.2 [87.8 to 94.7] | 92.5 [89.4 to 95.7]
  Week 80: number analyzed (Participants) | 247 | 259 | 251
  Week 80 | 89.2 [85.4 to 93.0] | 91.5 [88.1 to 94.9] | 89.6 [85.9 to 93.4]
  Week 84: number analyzed (Participants) | 248 | 260 | 252
  Week 84 | 87.1 [82.9 to 91.2] | 92.4 [89.2 to 95.6] | 93.5 [90.5 to 96.5]
  Week 88: number analyzed (Participants) | 245 | 256 | 247
  Week 88 | 87.3 [83.2 to 91.4] | 90.3 [86.7 to 93.8] | 89.9 [86.1 to 93.7]
  Week 92: number analyzed (Participants) | 248 | 258 | 248
  Week 92 | 89.4 [85.5 to 93.2] | 91.1 [87.6 to 94.6] | 90.8 [87.3 to 94.3]
  Week 96: number analyzed (Participants) | 242 | 259 | 245
  Week 96 | 90.7 [87.0 to 94.4] | 88.9 [85.1 to 92.6] | 90.5 [86.8 to 94.2]
  Week 100: number analyzed (Participants) | 254 | 258 | 247
  Week 100 | 88.3 [84.3 to 92.3] | 86.8 [82.7 to 90.9] | 92.0 [88.7 to 95.4]

10. Secondary Outcome: Percentage of Participants Gaining ≥15, ≥10, ≥5, or ≥0 Letters in BCVA From Baseline in the Study Eye Averaged Over Weeks 48, 52, and 56, Treatment-Naive Population
Description: BCVA was measured on the ETDRS chart at a starting distance of 4 meters. The BCVA letter score ranges from 0 to 100 (best score), and a gain in BCVA from baseline indicates an improvement in visual acuity. For each participant, an average BCVA value was calculated across the three visits, and this averaged value was then used to determine if the endpoint was met. The results were summarized as the percentage of participants per treatment arm who met the endpoint. The weighted estimates of the percentage of participants were based on the Cochran-Mantel Haenszel (CMH) weights stratified by baseline BCVA (≥64 vs. <64 letters) and region (U.S. and Canada vs. rest of the world). Treatment policy strategy and hypothetical strategy were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were not imputed. Invalid BCVA values were excluded. 95% confidence interval (CI) is a rounding of 95.04% CI.
Time Frame: Baseline, average of Weeks 48, 52, and 56
Population: Treatment-Naive Population: all participants randomized in the study who had not received any intravitreal anti-VEGF agents in the study eye prior to randomization. Participants were grouped according to the treatment assigned at randomization. Only participants with at least one non-missing, valid assessment at Weeks 48, 52, or 56 were included in the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 200 | 215 | 212
Percentage of participants
  Gaining ≥15 Letters | 28.6 [22.3 to 34.8] | 35.5 [29.3 to 41.7] | 33.8 [27.7 to 39.9]
  Gaining ≥10 Letters | 57.5 [50.7 to 64.4] | 59.6 [53.2 to 65.9] | 57.5 [50.9 to 64.1]
  Gaining ≥5 Letters | 80.0 [74.4 to 85.5] | 77.2 [71.6 to 82.8] | 84.5 [79.6 to 89.3]
  Gaining ≥0 Letters | 91.5 [87.6 to 95.3] | 93.5 [90.2 to 96.8] | 91.6 [87.9 to 95.3]
Statistical Analysis 1: Comparison: A: Faricimab 6 mg Q8W vs C: Aflibercept 2 mg Q8W; [analysis description as in outcome 5, analysis 1]; Test type: Other; Difference in CMH Weighted Percentage = -5.2, 95% CI 2-sided [-14.0 to 3.5]
Statistical Analysis 2: Comparison: B: Faricimab 6 mg PTI vs C: Aflibercept 2 mg Q8W; [analysis description as in outcome 5, analysis 2]; Test type: Other; Difference in CMH Weighted Percentage = 1.7, 95% CI 2-sided [-7.0 to 10.3]
Statistical Analysis 3: Comparison: A: Faricimab 6 mg Q8W vs C: Aflibercept 2 mg Q8W; [analysis description as in outcome 5, analysis 3]; Test type: Other; Difference in CMH Weighted Percentage = 0.0, 95% CI 2-sided [-9.5 to 9.5]
Statistical Analysis 4: Comparison: B: Faricimab 6 mg PTI vs C: Aflibercept 2 mg Q8W; [analysis description as in outcome 5, analysis 4]; Test type: Other; Difference in CMH Weighted Percentage = 2.1, 95% CI 2-sided [-7.1 to 11.3]
Statistical Analysis 5: Comparison: A: Faricimab 6 mg Q8W vs C: Aflibercept 2 mg Q8W; [analysis description as in outcome 5, analysis 5]; Test type: Other; Difference in CMH Weighted Percentage = -4.5, 95% CI 2-sided [-11.9 to 2.9]
Statistical Analysis 6: Comparison: B: Faricimab 6 mg PTI vs C: Aflibercept 2 mg Q8W; [analysis description as in outcome 5, analysis 6]; Test type: Other; Difference in CMH Weighted Percentage = -7.2, 95% CI 2-sided [-14.6 to 0.2]
Statistical Analysis 7: Comparison: A: Faricimab 6 mg Q8W vs C: Aflibercept 2 mg Q8W; [analysis description as in outcome 5, analysis 7]; Test type: Other; Difference in CMH Weighted Percentage = -0.2, 95% CI 2-sided [-5.5 to 5.2]
Statistical Analysis 8: Comparison: B: Faricimab 6 mg PTI vs C: Aflibercept 2 mg Q8W; [analysis description as in outcome 5, analysis 8]; Test type: Other; Difference in CMH Weighted Percentage = 2.0, 95% CI 2-sided [-3.0 to 7.0]

11. Secondary Outcome: Percentage of Participants Gaining ≥15 Letters in BCVA From Baseline in the Study Eye Over Time, Treatment-Naive Population
Description: Best Corrected Visual Acuity (BCVA) was measured on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart at a starting distance of 4 meters. The BCVA letter score ranges from 0 to 100 (best score), and a gain in BCVA letter score from baseline indicates an improvement in visual acuity. The weighted estimates of the percentage of participants were based on the Cochran-Mantel Haenszel (CMH) weights stratified by baseline BCVA (≥64 vs. <64 letters) and region (U.S. and Canada vs. rest of the world; Asia and rest of the world were combined). Treatment policy strategy (i.e., all observed values used) and hypothetical strategy (i.e., all values censored after the occurrence of the intercurrent event) were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were not imputed. Invalid BCVA values were excluded from analysis. 95% confidence interval (CI) is a rounding of 95.04% CI.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96, and 100
Population: Treatment-Naive Population: all participants randomized in the study who had not received any intravitreal anti-VEGF agents in the study eye prior to randomization. Participants were grouped according to the treatment assigned at randomization. At each timepoint, only participants with non-missing, valid assessments were included in the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 238 | 245 | 242
Percentage of participants
  Week 4: number analyzed (Participants) | 234 | 241 | 236
  Week 4 | 8.9 [5.3 to 12.5] | 14.9 [10.6 to 19.3] | 12.7 [8.6 to 16.9]
  Week 8: number analyzed (Participants) | 232 | 240 | 234
  Week 8 | 14.3 [9.9 to 18.8] | 19.2 [14.6 to 23.8] | 17.8 [13.1 to 22.6]
  Week 12: number analyzed (Participants) | 230 | 235 | 235
  Week 12 | 15.7 [11.1 to 20.3] | 22.2 [17.2 to 27.1] | 24.2 [19.0 to 29.5]
  Week 16: number analyzed (Participants) | 222 | 229 | 232
  Week 16 | 21.3 [16.0 to 26.6] | 28.2 [22.6 to 33.8] | 24.0 [18.6 to 29.3]
  Week 20: number analyzed (Participants) | 223 | 227 | 229
  Week 20 | 26.5 [20.8 to 32.2] | 27.7 [22.2 to 33.3] | 26.2 [20.7 to 31.6]
  Week 24: number analyzed (Participants) | 219 | 228 | 228
  Week 24 | 27.1 [21.3 to 32.9] | 34.3 [28.4 to 40.2] | 27.5 [22.0 to 33.1]
  Week 28: number analyzed (Participants) | 212 | 224 | 217
  Week 28 | 21.5 [16.0 to 27.0] | 30.7 [25.0 to 36.4] | 32.8 [26.8 to 38.7]
  Week 32: number analyzed (Participants) | 195 | 205 | 209
  Week 32 | 27.2 [21.0 to 33.5] | 37.5 [31.2 to 43.8] | 29.5 [23.6 to 35.4]
  Week 36: number analyzed (Participants) | 194 | 205 | 205
  Week 36 | 23.5 [17.6 to 29.5] | 41.9 [35.5 to 48.2] | 34.9 [28.6 to 41.2]
  Week 40: number analyzed (Participants) | 202 | 204 | 200
  Week 40 | 27.6 [21.5 to 33.8] | 37.7 [31.2 to 44.1] | 33.5 [27.0 to 39.9]
  Week 44: number analyzed (Participants) | 199 | 209 | 202
  Week 44 | 27.2 [21.1 to 33.4] | 39.7 [33.3 to 46.0] | 37.0 [30.6 to 43.4]
  Week 48: number analyzed (Participants) | 195 | 210 | 203
  Week 48 | 32.5 [26.0 to 39.1] | 39.6 [33.1 to 46.0] | 36.3 [30.1 to 42.5]
  Week 52: number analyzed (Participants) | 197 | 209 | 196
  Week 52 | 30.7 [24.3 to 37.1] | 35.9 [29.6 to 42.1] | 37.4 [30.9 to 43.9]
  Week 56: number analyzed (Participants) | 194 | 207 | 198
  Week 56 | 37.7 [31.0 to 44.5] | 38.8 [32.3 to 45.2] | 34.3 [27.9 to 40.8]
  Week 60: number analyzed (Participants) | 200 | 198 | 199
  Week 60 | 33.1 [26.6 to 39.6] | 42.2 [35.6 to 48.9] | 38.9 [32.4 to 45.5]
  Week 64: number analyzed (Participants) | 191 | 202 | 200
  Week 64 | 37.9 [31.1 to 44.7] | 43.5 [37.0 to 50.0] | 36.0 [29.5 to 42.6]
  Week 68: number analyzed (Participants) | 187 | 197 | 193
  Week 68 | 37.4 [30.7 to 44.2] | 45.4 [38.7 to 52.1] | 39.0 [32.4 to 45.5]
  Week 72: number analyzed (Participants) | 186 | 196 | 189
  Week 72 | 35.6 [28.8 to 42.4] | 39.6 [33.1 to 46.0] | 36.6 [29.8 to 43.3]
  Week 76: number analyzed (Participants) | 180 | 195 | 189
  Week 76 | 37.6 [30.6 to 44.6] | 45.3 [38.8 to 51.8] | 37.2 [30.5 to 43.9]
  Week 80: number analyzed (Participants) | 177 | 203 | 190
  Week 80 | 39.7 [32.7 to 46.8] | 43.2 [36.8 to 49.7] | 40.5 [33.6 to 47.3]
  Week 84: number analyzed (Participants) | 181 | 203 | 192
  Week 84 | 40.7 [33.7 to 47.8] | 43.2 [36.8 to 49.7] | 41.2 [34.3 to 48.1]
  Week 88: number analyzed (Participants) | 179 | 196 | 185
  Week 88 | 39.1 [32.1 to 46.2] | 40.7 [34.4 to 47.1] | 38.0 [31.2 to 44.8]
  Week 92: number analyzed (Participants) | 180 | 199 | 188
  Week 92 | 40.2 [33.2 to 47.3] | 42.1 [35.7 to 48.5] | 40.4 [33.6 to 47.3]
  Week 96: number analyzed (Participants) | 174 | 201 | 187
  Week 96 | 42.9 [35.6 to 50.2] | 41.2 [34.9 to 47.6] | 40.1 [33.2 to 47.0]
  Week 100: number analyzed (Participants) | 185 | 199 | 186
  Week 100 | 41.7 [34.6 to 48.7] | 42.5 [36.1 to 48.9] | 41.2 [34.3 to 48.1]

12. Secondary Outcome: Percentage of Participants Gaining ≥10 Letters in BCVA From Baseline in the Study Eye Over Time, Treatment-Naive Population
Description: as for outcome 11
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96, and 100
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 238 | 245 | 242
Percentage of participants
  Week 4: number analyzed (Participants) | 234 | 241 | 236
  Week 4 | 25.2 [19.7 to 30.7] | 32.0 [26.3 to 37.7] | 29.2 [23.5 to 35.0]
  Week 8: number analyzed (Participants) | 232 | 240 | 234
  Week 8 | 31.1 [25.2 to 37.1] | 37.2 [31.3 to 43.1] | 43.9 [37.7 to 50.2]
  Week 12: number analyzed (Participants) | 230 | 235 | 235
  Week 12 | 36.9 [30.8 to 43.1] | 46.5 [40.3 to 52.6] | 48.9 [42.6 to 55.2]
  Week 16: number analyzed (Participants) | 222 | 229 | 232
  Week 16 | 43.8 [37.3 to 50.3] | 47.8 [41.4 to 54.1] | 49.8 [43.5 to 56.2]
  Week 20: number analyzed (Participants) | 223 | 227 | 229
  Week 20 | 44.9 [38.4 to 51.4] | 53.7 [47.5 to 59.9] | 51.5 [45.1 to 57.9]
  Week 24: number analyzed (Participants) | 219 | 228 | 228
  Week 24 | 57.6 [51.1 to 64.1] | 57.9 [51.7 to 64.2] | 49.9 [43.5 to 56.3]
  Week 28: number analyzed (Participants) | 212 | 224 | 217
  Week 28 | 55.3 [48.6 to 61.9] | 56.6 [50.3 to 62.9] | 57.4 [50.8 to 63.9]
  Week 32: number analyzed (Participants) | 195 | 205 | 209
  Week 32 | 59.0 [52.2 to 65.9] | 59.6 [53.1 to 66.0] | 53.1 [46.5 to 59.7]
  Week 36: number analyzed (Participants) | 194 | 205 | 205
  Week 36 | 59.0 [52.1 to 65.9] | 66.3 [60.0 to 72.5] | 55.8 [49.1 to 62.5]
  Week 40: number analyzed (Participants) | 202 | 204 | 200
  Week 40 | 55.5 [48.7 to 62.4] | 59.7 [53.1 to 66.4] | 54.5 [47.7 to 61.4]
  Week 44: number analyzed (Participants) | 199 | 209 | 202
  Week 44 | 55.0 [48.1 to 61.9] | 59.2 [52.7 to 65.7] | 58.1 [51.3 to 64.8]
  Week 48: number analyzed (Participants) | 195 | 210 | 203
  Week 48 | 57.1 [50.2 to 64.0] | 58.5 [52.0 to 65.0] | 62.6 [56.0 to 69.2]
  Week 52: number analyzed (Participants) | 197 | 209 | 196
  Week 52 | 60.0 [53.1 to 66.8] | 58.8 [52.2 to 65.3] | 61.0 [54.2 to 67.8]
  Week 56: number analyzed (Participants) | 194 | 207 | 198
  Week 56 | 65.0 [58.3 to 71.7] | 62.9 [56.5 to 69.3] | 60.1 [53.4 to 66.8]
  Week 60: number analyzed (Participants) | 200 | 198 | 199
  Week 60 | 61.5 [54.7 to 68.2] | 63.4 [56.9 to 69.9] | 61.3 [54.5 to 68.0]
  Week 64: number analyzed (Participants) | 191 | 202 | 200
  Week 64 | 67.7 [61.1 to 74.3] | 59.8 [53.3 to 66.2] | 59.7 [53.0 to 66.4]
  Week 68: number analyzed (Participants) | 187 | 197 | 193
  Week 68 | 64.1 [57.4 to 70.8] | 60.7 [54.2 to 67.2] | 60.6 [53.9 to 67.3]
  Week 72: number analyzed (Participants) | 186 | 196 | 189
  Week 72 | 62.6 [55.8 to 69.5] | 62.5 [56.0 to 69.0] | 56.7 [49.8 to 63.7]
  Week 76: number analyzed (Participants) | 180 | 195 | 189
  Week 76 | 61.8 [54.8 to 68.9] | 66.8 [60.5 to 73.0] | 66.2 [59.6 to 72.9]
  Week 80: number analyzed (Participants) | 177 | 203 | 190
  Week 80 | 66.7 [59.8 to 73.5] | 62.4 [56.0 to 68.8] | 62.8 [56.0 to 69.6]
  Week 84: number analyzed (Participants) | 181 | 203 | 192
  Week 84 | 63.2 [56.3 to 70.1] | 65.3 [59.0 to 71.6] | 67.1 [60.5 to 73.6]
  Week 88: number analyzed (Participants) | 179 | 196 | 185
  Week 88 | 60.2 [53.2 to 67.3] | 60.9 [54.3 to 67.6] | 61.9 [55.1 to 68.7]
  Week 92: number analyzed (Participants) | 180 | 199 | 188
  Week 92 | 63.2 [56.2 to 70.2] | 65.1 [58.7 to 71.5] | 65.0 [58.2 to 71.7]
  Week 96: number analyzed (Participants) | 174 | 201 | 187
  Week 96 | 58.8 [51.5 to 66.0] | 60.6 [54.0 to 67.1] | 63.8 [56.9 to 70.6]
  Week 100: number analyzed (Participants) | 185 | 199 | 186
  Week 100 | 64.0 [57.3 to 70.7] | 62.4 [56.0 to 68.8] | 64.8 [58.0 to 71.6]

13. Secondary Outcome: Percentage of Participants Gaining ≥5 Letters in BCVA From Baseline in the Study Eye Over Time, Treatment-Naive Population
Description: as for outcome 11
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96, and 100
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 238 | 245 | 242
Percentage of participants
  Week 4: number analyzed (Participants) | 234 | 241 | 236
  Week 4 | 53.8 [47.5 to 60.2] | 63.1 [57.1 to 69.1] | 62.8 [56.7 to 68.9]
  Week 8: number analyzed (Participants) | 232 | 240 | 234
  Week 8 | 63.4 [57.2 to 69.6] | 70.5 [64.8 to 76.2] | 70.4 [64.6 to 76.2]
  Week 12: number analyzed (Participants) | 230 | 235 | 235
  Week 12 | 72.7 [66.9 to 78.4] | 75.4 [69.9 to 80.8] | 77.0 [71.6 to 82.4]
  Week 16: number analyzed (Participants) | 222 | 229 | 232
  Week 16 | 75.6 [70.0 to 81.3] | 81.3 [76.3 to 86.3] | 79.3 [74.1 to 84.5]
  Week 20: number analyzed (Participants) | 223 | 227 | 229
  Week 20 | 79.0 [73.6 to 84.3] | 79.3 [74.0 to 84.6] | 78.2 [72.9 to 83.5]
  Week 24: number analyzed (Participants) | 219 | 228 | 228
  Week 24 | 81.7 [76.6 to 86.8] | 82.9 [78.1 to 87.7] | 71.4 [65.5 to 77.2]
  Week 28: number analyzed (Participants) | 212 | 224 | 217
  Week 28 | 76.9 [71.2 to 82.5] | 81.7 [76.6 to 86.7] | 80.0 [74.8 to 85.3]
  Week 32: number analyzed (Participants) | 195 | 205 | 209
  Week 32 | 80.0 [74.4 to 85.6] | 77.6 [72.0 to 83.1] | 83.7 [78.8 to 88.7]
  Week 36: number analyzed (Participants) | 194 | 205 | 205
  Week 36 | 80.5 [74.9 to 86.1] | 82.9 [77.9 to 88.0] | 79.6 [74.1 to 85.1]
  Week 40: number analyzed (Participants) | 202 | 204 | 200
  Week 40 | 77.1 [71.3 to 82.8] | 85.3 [80.5 to 90.1] | 80.0 [74.5 to 85.6]
  Week 44: number analyzed (Participants) | 199 | 209 | 202
  Week 44 | 81.4 [76.0 to 86.8] | 82.5 [77.4 to 87.6] | 80.8 [75.4 to 86.2]
  Week 48: number analyzed (Participants) | 195 | 210 | 203
  Week 48 | 79.5 [73.8 to 85.2] | 80.0 [74.6 to 85.4] | 80.8 [75.4 to 86.2]
  Week 52: number analyzed (Participants) | 197 | 209 | 196
  Week 52 | 78.7 [72.9 to 84.4] | 75.3 [69.5 to 81.1] | 82.3 [77.1 to 87.6]
  Week 56: number analyzed (Participants) | 194 | 207 | 198
  Week 56 | 84.0 [78.9 to 89.2] | 81.2 [75.9 to 86.4] | 81.9 [76.6 to 87.1]
  Week 60: number analyzed (Participants) | 200 | 198 | 199
  Week 60 | 81.0 [75.5 to 86.4] | 80.5 [75.2 to 85.8] | 80.0 [74.5 to 85.5]
  Week 64: number analyzed (Participants) | 191 | 202 | 200
  Week 64 | 80.7 [75.1 to 86.3] | 80.2 [74.9 to 85.6] | 80.3 [74.8 to 85.7]
  Week 68: number analyzed (Participants) | 187 | 197 | 193
  Week 68 | 82.0 [76.5 to 87.5] | 78.3 [72.6 to 83.9] | 79.7 [74.1 to 85.2]
  Week 72: number analyzed (Participants) | 186 | 196 | 189
  Week 72 | 81.5 [76.0 to 87.0] | 77.3 [71.6 to 82.9] | 80.9 [75.4 to 86.5]
  Week 76: number analyzed (Participants) | 180 | 195 | 189
  Week 76 | 79.5 [73.7 to 85.4] | 78.0 [72.4 to 83.6] | 83.8 [78.6 to 88.9]
  Week 80: number analyzed (Participants) | 177 | 203 | 190
  Week 80 | 82.0 [76.3 to 87.7] | 80.5 [75.2 to 85.8] | 80.0 [74.3 to 85.7]
  Week 84: number analyzed (Participants) | 181 | 203 | 192
  Week 84 | 78.6 [72.6 to 84.6] | 83.0 [78.0 to 87.9] | 81.8 [76.4 to 87.3]
  Week 88: number analyzed (Participants) | 179 | 196 | 185
  Week 88 | 77.9 [71.8 to 83.9] | 80.7 [75.4 to 86.1] | 80.6 [74.9 to 86.2]
  Week 92: number analyzed (Participants) | 180 | 199 | 188
  Week 92 | 80.5 [74.8 to 86.3] | 82.1 [76.8 to 87.3] | 82.5 [77.2 to 87.9]
  Week 96: number analyzed (Participants) | 174 | 201 | 187
  Week 96 | 82.7 [77.1 to 88.3] | 76.9 [71.2 to 82.5] | 82.4 [76.9 to 87.8]
  Week 100: number analyzed (Participants) | 185 | 199 | 186
  Week 100 | 80.0 [74.3 to 85.8] | 78.2 [72.6 to 83.9] | 85.7 [80.8 to 90.7]

14. Secondary Outcome: Percentage of Participants Gaining ≥0 Letters in BCVA From Baseline in the Study Eye Over Time, Treatment-Naive Population
Description: as for outcome 11
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96, and 100
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 238 | 245 | 242
Percentage of participants
  Week 4: number analyzed (Participants) | 234 | 241 | 236
  Week 4 | 86.3 [81.9 to 90.7] | 90.9 [87.3 to 94.5] | 90.2 [86.5 to 94.0]
  Week 8: number analyzed (Participants) | 232 | 240 | 234
  Week 8 | 91.4 [87.8 to 95.0] | 93.3 [90.2 to 96.5] | 93.1 [89.9 to 96.4]
  Week 12: number analyzed (Participants) | 230 | 235 | 235
  Week 12 | 93.5 [90.4 to 96.6] | 96.2 [93.7 to 98.6] | 92.8 [89.4 to 96.1]
  Week 16: number analyzed (Participants) | 222 | 229 | 232
  Week 16 | 91.5 [87.8 to 95.1] | 94.7 [91.9 to 97.6] | 94.5 [91.6 to 97.4]
  Week 20: number analyzed (Participants) | 223 | 227 | 229
  Week 20 | 94.2 [91.2 to 97.2] | 92.5 [89.1 to 95.9] | 92.1 [88.6 to 95.6]
  Week 24: number analyzed (Participants) | 219 | 228 | 228
  Week 24 | 94.0 [90.9 to 97.1] | 93.4 [90.2 to 96.6] | 89.0 [85.0 to 93.1]
  Week 28: number analyzed (Participants) | 212 | 224 | 217
  Week 28 | 90.9 [87.0 to 94.8] | 94.2 [91.1 to 97.2] | 92.6 [89.1 to 96.1]
  Week 32: number analyzed (Participants) | 195 | 205 | 209
  Week 32 | 92.3 [88.5 to 96.0] | 94.2 [91.0 to 97.3] | 91.4 [87.7 to 95.2]
  Week 36: number analyzed (Participants) | 194 | 205 | 205
  Week 36 | 93.1 [89.5 to 96.7] | 93.7 [90.4 to 97.0] | 89.4 [85.2 to 93.6]
  Week 40: number analyzed (Participants) | 202 | 204 | 200
  Week 40 | 91.0 [87.0 to 94.9] | 93.6 [90.3 to 97.0] | 92.5 [88.9 to 96.2]
  Week 44: number analyzed (Participants) | 199 | 209 | 202
  Week 44 | 91.8 [88.0 to 95.6] | 93.4 [90.0 to 96.7] | 91.6 [87.8 to 95.4]
  Week 48: number analyzed (Participants) | 195 | 210 | 203
  Week 48 | 95.5 [92.6 to 98.4] | 91.9 [88.2 to 95.6] | 93.1 [89.7 to 96.6]
  Week 52: number analyzed (Participants) | 197 | 209 | 196
  Week 52 | 89.8 [85.6 to 94.0] | 89.5 [85.4 to 93.6] | 90.9 [87.0 to 94.9]
  Week 56: number analyzed (Participants) | 194 | 207 | 198
  Week 56 | 91.7 [87.8 to 95.6] | 92.7 [89.2 to 96.3] | 90.9 [86.9 to 94.9]
  Week 60: number analyzed (Participants) | 200 | 198 | 199
  Week 60 | 89.9 [85.7 to 94.1] | 93.5 [90.1 to 96.9] | 91.9 [88.2 to 95.7]
  Week 64: number analyzed (Participants) | 191 | 202 | 200
  Week 64 | 92.0 [88.1 to 95.9] | 92.6 [89.1 to 96.1] | 92.4 [88.7 to 96.1]
  Week 68: number analyzed (Participants) | 187 | 197 | 193
  Week 68 | 92.0 [88.1 to 95.8] | 93.4 [90.0 to 96.8] | 91.8 [88.0 to 95.6]
  Week 72: number analyzed (Participants) | 186 | 196 | 189
  Week 72 | 88.7 [84.1 to 93.2] | 92.0 [88.4 to 95.6] | 89.3 [84.9 to 93.7]
  Week 76: number analyzed (Participants) | 180 | 195 | 189
  Week 76 | 86.8 [81.8 to 91.7] | 90.8 [86.8 to 94.8] | 91.6 [87.8 to 95.5]
  Week 80: number analyzed (Participants) | 177 | 203 | 190
  Week 80 | 89.5 [85.0 to 94.0] | 90.7 [86.7 to 94.7] | 90.1 [85.8 to 94.3]
  Week 84: number analyzed (Participants) | 181 | 203 | 192
  Week 84 | 87.4 [82.6 to 92.3] | 92.2 [88.5 to 95.8] | 92.5 [88.9 to 96.1]
  Week 88: number analyzed (Participants) | 179 | 196 | 185
  Week 88 | 85.6 [80.4 to 90.7] | 88.8 [84.5 to 93.2] | 89.2 [84.7 to 93.7]
  Week 92: number analyzed (Participants) | 180 | 199 | 188
  Week 92 | 88.8 [84.2 to 93.4] | 90.5 [86.5 to 94.6] | 91.0 [86.9 to 95.1]
  Week 96: number analyzed (Participants) | 174 | 201 | 187
  Week 96 | 90.1 [85.7 to 94.6] | 87.2 [82.6 to 91.7] | 90.3 [86.1 to 94.6]
  Week 100: number analyzed (Participants) | 185 | 199 | 186
  Week 100 | 87.8 [83.1 to 92.6] | 86.1 [81.4 to 90.8] | 92.0 [88.1 to 95.9]

15. Secondary Outcome: Percentage of Participants Avoiding a Loss of ≥15, ≥10, or ≥5 Letters in BCVA From Baseline in the Study Eye Averaged Over Weeks 48, 52, and 56, ITT Population
Description: Best Corrected Visual Acuity (BCVA) was measured on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart at a starting distance of 4 meters. For each participant, an average BCVA value was calculated across the three visits, and this averaged value was then used to determine if the endpoint was met. The results were summarized as the percentage of participants per treatment arm who met the endpoint. The weighted estimates of the percentage of participants were based on the Cochran-Mantel Haenszel (CMH) weights stratified by baseline BCVA (≥64 vs. <64 letters), prior IVT anti-VEGF therapy (yes vs. no), and region (U.S. and Canada vs. rest of the world; Asia and rest of the world were combined). Treatment policy strategy and hypothetical strategy were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were not imputed. Invalid BCVA values were excluded. 95% confidence interval (CI) is a rounding of 95.04% CI.
Time Frame: Baseline, average of Weeks 48, 52, and 56
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 271 | 276 | 276
Percentage of participants
  Avoiding a Loss of ≥15 Letters | 98.1 [96.5 to 99.7] | 98.6 [97.2 to 100.0] | 98.9 [97.6 to 100.0]
  Avoiding a Loss of ≥10 Letters | 96.3 [94.1 to 98.5] | 98.2 [96.6 to 99.8] | 98.1 [96.5 to 99.7]
  Avoiding a Loss of ≥5 Letters | 95.2 [92.7 to 97.7] | 96.7 [94.7 to 98.8] | 96.3 [94.1 to 98.5]
Statistical Analysis 1: Comparison: A: Faricimab 6 mg Q8W vs C: Aflibercept 2 mg Q8W; This is the difference in percentage of participants avoiding a loss of ≥15 letters in Arm A: Faricimab 6 mg Q8W minus Arm C: Aflibercept 2 mg Q8W; Test type: Other; Difference in CMH Weighted Percentage = -0.8, 95% CI 2-sided [-2.8 to 1.3]
Statistical Analysis 2: Comparison: B: Faricimab 6 mg PTI vs C: Aflibercept 2 mg Q8W; This is the difference in percentage of participants avoiding a loss of ≥15 letters in Arm B: Faricimab 6 mg PTI minus Arm C: Aflibercept 2 mg Q8W; Test type: Other; Difference in CMH Weighted Percentage = -0.3, 95% CI 2-sided [-2.2 to 1.5]
Statistical Analysis 3: Comparison: A: Faricimab 6 mg Q8W vs C: Aflibercept 2 mg Q8W; This is the difference in percentage of participants avoiding a loss of ≥10 letters in Arm A: Faricimab 6 mg Q8W minus Arm C: Aflibercept 2 mg Q8W; Test type: Other; Difference in CMH Weighted Percentage = -1.8, 95% CI 2-sided [-4.6 to 0.9]
Statistical Analysis 4: Comparison: B: Faricimab 6 mg PTI vs C: Aflibercept 2 mg Q8W; This is the difference in percentage of participants avoiding a loss of ≥10 letters in Arm B: Faricimab 6 mg PTI minus Arm C: Aflibercept 2 mg Q8W; Test type: Other; Difference in CMH Weighted Percentage = 0.0, 95% CI 2-sided [-2.2 to 2.2]
Statistical Analysis 5: Comparison: A: Faricimab 6 mg Q8W vs C: Aflibercept 2 mg Q8W; This is the difference in percentage of participants avoiding a loss of ≥5 letters in Arm A: Faricimab 6 mg Q8W minus Arm C: Aflibercept 2 mg Q8W; Test type: Other; Difference in CMH Weighted Percentage = -1.1, 95% CI 2-sided [-4.5 to 2.2]
Statistical Analysis 6: Comparison: B: Faricimab 6 mg PTI vs C: Aflibercept 2 mg Q8W; This is the difference in percentage of participants avoiding a loss of ≥5 letters in Arm B: Faricimab 6 mg PTI minus Arm C: Aflibercept 2 mg Q8W; Test type: Other; Difference in CMH Weighted Percentage = 0.4, 95% CI 2-sided [-2.6 to 3.4]

16. Secondary Outcome: Percentage of Participants Avoiding a Loss of ≥15 Letters in BCVA From Baseline in the Study Eye Over Time, ITT Population
Description: Best Corrected Visual Acuity (BCVA) was measured on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart at a starting distance of 4 meters. The weighted estimates of the percentage of participants avoiding a loss of letters in BCVA from baseline were based on the Cochran-Mantel Haenszel (CMH) weights stratified by baseline BCVA (≥64 vs. <64 letters), prior IVT anti-VEGF therapy (yes vs. no), and region (U.S. and Canada vs. rest of the world; Asia and rest of the world were combined). Treatment policy strategy (i.e., all observed values used) and hypothetical strategy (i.e., all values censored after the occurrence of the intercurrent event) were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were not imputed. Invalid BCVA values were excluded from analysis. 95% confidence interval (CI) is a rounding of 95.04% CI.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96, and 100
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 315 | 313 | 312
Percentage of participants
  Week 4: number analyzed (Participants) | 310 | 308 | 306
  Week 4 | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0]
  Week 8: number analyzed (Participants) | 309 | 308 | 304
  Week 8 | 99.7 [99.0 to 100.0] | 100.0 [100.0 to 100.0] | 99.3 [98.4 to 100.0]
  Week 12: number analyzed (Participants) | 305 | 303 | 302
  Week 12 | 99.3 [98.5 to 100.0] | 100.0 [100.0 to 100.0] | 99.7 [99.0 to 100.0]
  Week 16: number analyzed (Participants) | 296 | 296 | 299
  Week 16 | 99.7 [99.0 to 100.0] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0]
  Week 20: number analyzed (Participants) | 294 | 292 | 296
  Week 20 | 99.3 [98.4 to 100.0] | 99.3 [98.4 to 100.0] | 99.6 [99.0 to 100.0]
  Week 24: number analyzed (Participants) | 292 | 293 | 294
  Week 24 | 99.6 [98.9 to 100.0] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0]
  Week 28: number analyzed (Participants) | 283 | 287 | 284
  Week 28 | 99.3 [98.2 to 100.0] | 99.7 [99.0 to 100.0] | 99.6 [99.0 to 100.0]
  Week 32: number analyzed (Participants) | 267 | 268 | 275
  Week 32 | 99.6 [98.8 to 100.0] | 100.0 [100.0 to 100.0] | 99.3 [98.3 to 100.0]
  Week 36: number analyzed (Participants) | 268 | 268 | 268
  Week 36 | 99.2 [98.0 to 100.0] | 99.2 [98.2 to 100.0] | 99.6 [98.8 to 100.0]
  Week 40: number analyzed (Participants) | 275 | 269 | 263
  Week 40 | 98.8 [97.5 to 100.0] | 99.3 [98.2 to 100.0] | 99.6 [98.8 to 100.0]
  Week 44: number analyzed (Participants) | 268 | 269 | 266
  Week 44 | 98.8 [97.5 to 100.0] | 98.9 [97.7 to 100.0] | 100.0 [100.0 to 100.0]
  Week 48: number analyzed (Participants) | 264 | 266 | 266
  Week 48 | 98.4 [96.9 to 100.0] | 98.1 [96.5 to 99.7] | 99.3 [98.3 to 100.0]
  Week 52: number analyzed (Participants) | 264 | 267 | 253
  Week 52 | 97.2 [95.2 to 99.2] | 98.1 [96.5 to 99.7] | 98.4 [96.8 to 99.9]
  Week 56: number analyzed (Participants) | 260 | 263 | 256
  Week 56 | 98.4 [96.9 to 99.9] | 98.5 [97.0 to 100.0] | 98.4 [96.9 to 99.9]
  Week 60: number analyzed (Participants) | 270 | 261 | 261
  Week 60 | 98.1 [96.4 to 99.7] | 98.5 [97.0 to 99.9] | 99.2 [98.1 to 100.0]
  Week 64: number analyzed (Participants) | 259 | 263 | 263
  Week 64 | 98.8 [97.4 to 100.0] | 97.7 [95.8 to 99.5] | 98.8 [97.5 to 100.0]
  Week 68: number analyzed (Participants) | 251 | 257 | 253
  Week 68 | 99.1 [98.0 to 100.0] | 98.0 [96.3 to 99.7] | 98.8 [97.5 to 100.0]
  Week 72: number analyzed (Participants) | 253 | 257 | 251
  Week 72 | 97.2 [95.1 to 99.2] | 98.8 [97.5 to 100.0] | 98.8 [97.5 to 100.0]
  Week 76: number analyzed (Participants) | 247 | 253 | 251
  Week 76 | 96.6 [94.4 to 98.9] | 98.0 [96.3 to 99.7] | 98.0 [96.3 to 99.7]
  Week 80: number analyzed (Participants) | 247 | 259 | 251
  Week 80 | 97.6 [95.7 to 99.5] | 96.9 [94.8 to 99.0] | 99.1 [98.0 to 100.0]
  Week 84: number analyzed (Participants) | 248 | 260 | 252
  Week 84 | 97.1 [95.0 to 99.2] | 98.1 [96.5 to 99.7] | 99.1 [98.0 to 100.0]
  Week 88: number analyzed (Participants) | 245 | 256 | 247
  Week 88 | 97.1 [95.0 to 99.2] | 97.2 [95.2 to 99.2] | 97.9 [96.1 to 99.7]
  Week 92: number analyzed (Participants) | 248 | 258 | 248
  Week 92 | 97.1 [95.0 to 99.2] | 97.4 [95.5 to 99.3] | 98.3 [96.6 to 99.9]
  Week 96: number analyzed (Participants) | 242 | 259 | 245
  Week 96 | 97.4 [95.3 to 99.4] | 96.6 [94.4 to 98.8] | 97.8 [95.9 to 99.7]
  Week 100: number analyzed (Participants) | 254 | 258 | 247
  Week 100 | 96.3 [93.9 to 98.7] | 97.0 [94.9 to 99.0] | 98.4 [96.8 to 99.9]

17. Secondary Outcome: Percentage of Participants Avoiding a Loss of ≥10 Letters in BCVA From Baseline in the Study Eye Over Time, ITT Population
Description: as for outcome 16
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96, and 100
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 315 | 313 | 312
Percentage of participants
  Week 4: number analyzed (Participants) | 310 | 308 | 306
  Week 4 | 98.7 [97.5 to 99.9] | 100.0 [100.0 to 100.0] | 99.4 [98.5 to 100.0]
  Week 8: number analyzed (Participants) | 309 | 308 | 304
  Week 8 | 98.4 [97.0 to 99.8] | 100.0 [100.0 to 100.0] | 99.0 [97.9 to 100.0]
  Week 12: number analyzed (Participants) | 305 | 303 | 302
  Week 12 | 98.7 [97.4 to 100.0] | 100.0 [100.0 to 100.0] | 99.3 [98.4 to 100.0]
  Week 16: number analyzed (Participants) | 296 | 296 | 299
  Week 16 | 99.3 [98.4 to 100.0] | 99.3 [98.4 to 100.0] | 99.7 [99.0 to 100.0]
  Week 20: number analyzed (Participants) | 294 | 292 | 296
  Week 20 | 99.0 [97.8 to 100.0] | 98.6 [97.3 to 100.0] | 99.3 [98.4 to 100.0]
  Week 24: number analyzed (Participants) | 292 | 293 | 294
  Week 24 | 98.6 [97.2 to 100.0] | 99.7 [99.0 to 100.0] | 99.3 [98.4 to 100.0]
  Week 28: number analyzed (Participants) | 283 | 287 | 284
  Week 28 | 97.4 [95.6 to 99.3] | 99.0 [97.8 to 100.0] | 98.6 [97.2 to 100.0]
  Week 32: number analyzed (Participants) | 267 | 268 | 275
  Week 32 | 99.2 [98.1 to 100.0] | 98.5 [97.0 to 99.9] | 98.5 [97.1 to 99.9]
  Week 36: number analyzed (Participants) | 268 | 268 | 268
  Week 36 | 98.4 [96.9 to 99.9] | 98.9 [97.6 to 100.0] | 99.2 [98.2 to 100.0]
  Week 40: number analyzed (Participants) | 275 | 269 | 263
  Week 40 | 97.7 [95.9 to 99.5] | 99.3 [98.2 to 100.0] | 98.5 [97.0 to 99.9]
  Week 44: number analyzed (Participants) | 268 | 269 | 266
  Week 44 | 97.3 [95.4 to 99.3] | 98.2 [96.6 to 99.8] | 99.2 [98.2 to 100.0]
  Week 48: number analyzed (Participants) | 264 | 266 | 266
  Week 48 | 98.1 [96.4 to 99.7] | 97.8 [96.0 to 99.5] | 98.5 [97.1 to 99.9]
  Week 52: number analyzed (Participants) | 264 | 267 | 253
  Week 52 | 95.3 [92.8 to 97.9] | 97.0 [95.0 to 99.0] | 96.8 [94.6 to 99.0]
  Week 56: number analyzed (Participants) | 260 | 263 | 256
  Week 56 | 97.2 [95.2 to 99.2] | 98.1 [96.5 to 99.7] | 96.5 [94.3 to 98.7]
  Week 60: number analyzed (Participants) | 270 | 261 | 261
  Week 60 | 96.9 [94.8 to 99.0] | 97.3 [95.4 to 99.3] | 98.1 [96.4 to 99.7]
  Week 64: number analyzed (Participants) | 259 | 263 | 263
  Week 64 | 98.0 [96.3 to 99.7] | 96.5 [94.2 to 98.7] | 98.1 [96.4 to 99.7]
  Week 68: number analyzed (Participants) | 251 | 257 | 253
  Week 68 | 96.9 [94.7 to 99.0] | 97.6 [95.8 to 99.5] | 98.4 [96.9 to 100.0]
  Week 72: number analyzed (Participants) | 253 | 257 | 251
  Week 72 | 96.0 [93.6 to 98.4] | 98.0 [96.4 to 99.7] | 97.6 [95.7 to 99.5]
  Week 76: number analyzed (Participants) | 247 | 253 | 251
  Week 76 | 95.9 [93.4 to 98.4] | 95.6 [93.1 to 98.1] | 97.6 [95.7 to 99.5]
  Week 80: number analyzed (Participants) | 247 | 259 | 251
  Week 80 | 96.3 [94.0 to 98.7] | 96.2 [93.8 to 98.5] | 97.6 [95.9 to 99.5]
  Week 84: number analyzed (Participants) | 248 | 260 | 252
  Week 84 | 95.5 [93.0 to 98.1] | 97.0 [95.0 to 99.0] | 99.1 [98.0 to 100.0]
  Week 88: number analyzed (Participants) | 245 | 256 | 247
  Week 88 | 95.0 [92.3 to 97.7] | 95.6 [93.1 to 98.1] | 96.7 [94.5 to 98.9]
  Week 92: number analyzed (Participants) | 248 | 258 | 248
  Week 92 | 95.9 [93.3 to 98.4] | 96.5 [94.3 to 98.7] | 97.5 [95.5 to 99.5]
  Week 96: number analyzed (Participants) | 242 | 259 | 245
  Week 96 | 96.9 [94.7 to 99.2] | 94.3 [91.5 to 97.1] | 96.6 [94.3 to 98.9]
  Week 100: number analyzed (Participants) | 254 | 258 | 247
  Week 100 | 94.3 [91.5 to 97.2] | 94.6 [91.8 to 97.3] | 97.1 [95.1 to 99.2]

18. Secondary Outcome: Percentage of Participants Avoiding a Loss of ≥5 Letters in BCVA From Baseline in the Study Eye Over Time, ITT Population
Description: as for outcome 16
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96, and 100
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 315 | 313 | 312
Percentage of participants
  Week 4: number analyzed (Participants) | 310 | 308 | 306
  Week 4 | 97.7 [96.1 to 99.4] | 97.4 [95.6 to 99.1] | 96.4 [94.4 to 98.4]
  Week 8: number analyzed (Participants) | 309 | 308 | 304
  Week 8 | 96.4 [94.4 to 98.5] | 98.7 [97.5 to 100.0] | 97.3 [95.5 to 99.1]
  Week 12: number analyzed (Participants) | 305 | 303 | 302
  Week 12 | 98.0 [96.5 to 99.6] | 98.0 [96.4 to 99.6] | 98.4 [97.0 to 99.8]
  Week 16: number analyzed (Participants) | 296 | 296 | 299
  Week 16 | 97.3 [95.5 to 99.1] | 98.6 [97.3 to 100.0] | 98.7 [97.4 to 100.0]
  Week 20: number analyzed (Participants) | 294 | 292 | 296
  Week 20 | 96.9 [95.0 to 98.9] | 97.2 [95.4 to 99.1] | 97.3 [95.4 to 99.1]
  Week 24: number analyzed (Participants) | 292 | 293 | 294
  Week 24 | 96.9 [94.9 to 98.9] | 96.9 [94.9 to 98.9] | 96.6 [94.6 to 98.7]
  Week 28: number analyzed (Participants) | 283 | 287 | 284
  Week 28 | 96.4 [94.2 to 98.6] | 97.6 [95.8 to 99.3] | 96.1 [93.9 to 98.4]
  Week 32: number analyzed (Participants) | 267 | 268 | 275
  Week 32 | 96.6 [94.4 to 98.8] | 97.4 [95.5 to 99.3] | 97.5 [95.6 to 99.3]
  Week 36: number analyzed (Participants) | 268 | 268 | 268
  Week 36 | 96.2 [93.9 to 98.5] | 97.3 [95.4 to 99.3] | 97.7 [96.0 to 99.5]
  Week 40: number analyzed (Participants) | 275 | 269 | 263
  Week 40 | 95.2 [92.6 to 97.7] | 95.8 [93.4 to 98.2] | 97.7 [95.9 to 99.5]
  Week 44: number analyzed (Participants) | 268 | 269 | 266
  Week 44 | 95.2 [92.6 to 97.7] | 96.7 [94.6 to 98.8] | 95.8 [93.4 to 98.2]
  Week 48: number analyzed (Participants) | 264 | 266 | 266
  Week 48 | 96.6 [94.4 to 98.8] | 96.7 [94.5 to 98.8] | 96.9 [94.9 to 99.0]
  Week 52: number analyzed (Participants) | 264 | 267 | 253
  Week 52 | 94.2 [91.4 to 97.0] | 95.9 [93.5 to 98.3] | 94.9 [92.2 to 97.6]
  Week 56: number analyzed (Participants) | 260 | 263 | 256
  Week 56 | 96.0 [93.7 to 98.4] | 96.2 [93.8 to 98.5] | 95.0 [92.4 to 97.6]
  Week 60: number analyzed (Participants) | 270 | 261 | 261
  Week 60 | 94.0 [91.2 to 96.8] | 96.2 [93.8 to 98.5] | 97.0 [94.9 to 99.0]
  Week 64: number analyzed (Participants) | 259 | 263 | 263
  Week 64 | 95.7 [93.2 to 98.2] | 96.1 [93.8 to 98.5] | 96.1 [93.8 to 98.4]
  Week 68: number analyzed (Participants) | 251 | 257 | 253
  Week 68 | 94.8 [92.1 to 97.6] | 96.4 [94.1 to 98.7] | 96.1 [93.8 to 98.5]
  Week 72: number analyzed (Participants) | 253 | 257 | 251
  Week 72 | 93.3 [90.3 to 96.4] | 95.3 [92.7 to 97.9] | 94.4 [91.5 to 97.2]
  Week 76: number analyzed (Participants) | 247 | 253 | 251
  Week 76 | 92.6 [89.4 to 95.9] | 94.8 [92.0 to 97.5] | 95.2 [92.6 to 97.8]
  Week 80: number analyzed (Participants) | 247 | 259 | 251
  Week 80 | 94.0 [91.0 to 96.9] | 93.4 [90.4 to 96.4] | 94.0 [91.1 to 96.9]
  Week 84: number analyzed (Participants) | 248 | 260 | 252
  Week 84 | 92.8 [89.6 to 96.0] | 95.8 [93.4 to 98.2] | 97.2 [95.1 to 99.2]
  Week 88: number analyzed (Participants) | 245 | 256 | 247
  Week 88 | 89.8 [86.0 to 93.5] | 92.6 [89.4 to 95.8] | 94.7 [91.9 to 97.5]
  Week 92: number analyzed (Participants) | 248 | 258 | 248
  Week 92 | 93.8 [90.8 to 96.8] | 92.7 [89.5 to 95.8] | 96.7 [94.4 to 98.9]
  Week 96: number analyzed (Participants) | 242 | 259 | 245
  Week 96 | 94.9 [92.0 to 97.7] | 92.3 [89.1 to 95.5] | 95.0 [92.3 to 97.8]
  Week 100: number analyzed (Participants) | 254 | 258 | 247
  Week 100 | 91.1 [87.6 to 94.6] | 88.9 [85.1 to 92.6] | 96.4 [94.1 to 98.6]

19. Secondary Outcome: Percentage of Participants Avoiding a Loss of ≥15, ≥10, or ≥5 Letters in BCVA From Baseline in the Study Eye Averaged Over Weeks 48, 52, and 56, Treatment-Naive Population
Description: Best Corrected Visual Acuity (BCVA) was measured on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart at a starting distance of 4 meters. For each participant, an average BCVA value was calculated across the three visits, and this averaged value was then used to determine if the endpoint was met. The results were summarized as the percentage of participants per treatment arm who met the endpoint. The weighted estimates of the percentage of participants were based on the Cochran-Mantel Haenszel (CMH) weights stratified by baseline BCVA (≥64 vs. <64 letters) and region (U.S. and Canada vs. rest of the world; Asia and rest of the world were combined). Treatment policy strategy and hypothetical strategy were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were not imputed. Invalid BCVA values were excluded. 95% confidence interval (CI) is a rounding of 95.04% CI.
Time Frame: Baseline, average of Weeks 48, 52, and 56
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 200 | 215 | 212
Percentage of participants
  Avoiding a Loss of ≥15 Letters | 97.9 [96.0 to 99.9] | 98.1 [96.3 to 99.9] | 99.0 [97.7 to 100.0]
  Avoiding a Loss of ≥10 Letters | 96.5 [93.9 to 99.0] | 97.7 [95.7 to 99.7] | 98.6 [97.0 to 100.0]
  Avoiding a Loss of ≥5 Letters | 95.0 [91.9 to 98.0] | 95.8 [93.1 to 98.5] | 96.2 [93.6 to 98.8]
Statistical Analysis 1: Comparison: A: Faricimab 6 mg Q8W vs C: Aflibercept 2 mg Q8W; [analysis description as in outcome 15, analysis 1]; Test type: Other; Difference in CMH Weighted Percentage = -1.1, 95% CI 2-sided [-3.5 to 1.3]
Statistical Analysis 2: Comparison: B: Faricimab 6 mg PTI vs C: Aflibercept 2 mg Q8W; [analysis description as in outcome 15, analysis 2]; Test type: Other; Difference in CMH Weighted Percentage = -0.9, 95% CI 2-sided [-3.1 to 1.3]
Statistical Analysis 3: Comparison: A: Faricimab 6 mg Q8W vs C: Aflibercept 2 mg Q8W; [analysis description as in outcome 15, analysis 3]; Test type: Other; Difference in CMH Weighted Percentage = -2.1, 95% CI 2-sided [-5.1 to 0.9]
Statistical Analysis 4: Comparison: B: Faricimab 6 mg PTI vs C: Aflibercept 2 mg Q8W; [analysis description as in outcome 15, analysis 4]; Test type: Other; Difference in CMH Weighted Percentage = -0.9, 95% CI 2-sided [-3.5 to 1.6]
Statistical Analysis 5: Comparison: A: Faricimab 6 mg Q8W vs C: Aflibercept 2 mg Q8W; [analysis description as in outcome 15, analysis 5]; Test type: Other; Difference in CMH Weighted Percentage = -1.2, 95% CI 2-sided [-5.2 to 2.8]
Statistical Analysis 6: Comparison: B: Faricimab 6 mg PTI vs C: Aflibercept 2 mg Q8W; [analysis description as in outcome 15, analysis 6]; Test type: Other; Difference in CMH Weighted Percentage = -0.4, 95% CI 2-sided [-4.1 to 3.3]

20. Secondary Outcome: Percentage of Participants Avoiding a Loss of ≥15 Letters in BCVA From Baseline in the Study Eye Over Time, Treatment-Naive Population
Description: Best Corrected Visual Acuity (BCVA) was measured on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart at a starting distance of 4 meters. The weighted estimates of the percentage of participants avoiding a loss of letters in BCVA from baseline were based on the Cochran-Mantel Haenszel (CMH) weights stratified by baseline BCVA (≥64 vs. <64 letters) and region (U.S. and Canada vs. rest of the world; Asia and rest of the world were combined). Treatment policy strategy (i.e., all observed values used) and hypothetical strategy (i.e., all values censored after the occurrence of the intercurrent event) were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were not imputed. Invalid BCVA values were excluded from analysis. 95% confidence interval (CI) is a rounding of 95.04% CI.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96, and 100
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 238 | 245 | 242
Percentage of participants
  Week 4: number analyzed (Participants) | 234 | 241 | 236
  Week 4 | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0]
  Week 8: number analyzed (Participants) | 232 | 240 | 234
  Week 8 | 99.6 [98.7 to 100.0] | 100.0 [100.0 to 100.0] | 99.6 [98.8 to 100.0]
  Week 12: number analyzed (Participants) | 230 | 235 | 235
  Week 12 | 99.6 [98.7 to 100.0] | 100.0 [100.0 to 100.0] | 99.6 [98.7 to 100.0]
  Week 16: number analyzed (Participants) | 222 | 229 | 232
  Week 16 | 99.6 [98.7 to 100.0] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0]
  Week 20: number analyzed (Participants) | 223 | 227 | 229
  Week 20 | 99.1 [97.9 to 100.0] | 99.1 [97.9 to 100.0] | 100.0 [100.0 to 100.0]
  Week 24: number analyzed (Participants) | 219 | 228 | 228
  Week 24 | 99.5 [98.6 to 100.0] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0]
  Week 28: number analyzed (Participants) | 212 | 224 | 217
  Week 28 | 99.0 [97.6 to 100.0] | 99.6 [98.7 to 100.0] | 99.5 [98.6 to 100.0]
  Week 32: number analyzed (Participants) | 195 | 205 | 209
  Week 32 | 99.5 [98.4 to 100.0] | 100.0 [100.0 to 100.0] | 99.0 [97.7 to 100.0]
  Week 36: number analyzed (Participants) | 194 | 205 | 205
  Week 36 | 98.9 [97.3 to 100.0] | 99.0 [97.6 to 100.0] | 99.5 [98.4 to 100.0]
  Week 40: number analyzed (Participants) | 202 | 204 | 200
  Week 40 | 98.4 [96.6 to 100.0] | 99.0 [97.7 to 100.0] | 99.5 [98.4 to 100.0]
  Week 44: number analyzed (Participants) | 199 | 209 | 202
  Week 44 | 98.9 [97.5 to 100.0] | 98.6 [97.0 to 100.0] | 100.0 [100.0 to 100.0]
  Week 48: number analyzed (Participants) | 195 | 210 | 203
  Week 48 | 98.4 [96.6 to 100.0] | 97.6 [95.5 to 99.7] | 99.0 [97.7 to 100.0]
  Week 52: number analyzed (Participants) | 197 | 209 | 196
  Week 52 | 96.8 [94.3 to 99.3] | 97.6 [95.5 to 99.7] | 98.4 [96.6 to 100.0]
  Week 56: number analyzed (Participants) | 194 | 207 | 198
  Week 56 | 98.4 [96.7 to 100.0] | 98.1 [96.2 to 99.9] | 98.5 [96.7 to 100.0]
  Week 60: number analyzed (Participants) | 200 | 198 | 199
  Week 60 | 97.4 [95.2 to 99.6] | 98.0 [96.1 to 99.9] | 99.0 [97.5 to 100.0]
  Week 64: number analyzed (Participants) | 191 | 202 | 200
  Week 64 | 98.4 [96.5 to 100.0] | 97.0 [94.6 to 99.4] | 98.4 [96.7 to 100.0]
  Week 68: number analyzed (Participants) | 187 | 197 | 193
  Week 68 | 98.9 [97.3 to 100.0] | 97.4 [95.2 to 99.6] | 98.4 [96.7 to 100.0]
  Week 72: number analyzed (Participants) | 186 | 196 | 189
  Week 72 | 96.2 [93.4 to 98.9] | 98.5 [96.8 to 100.0] | 98.4 [96.6 to 100.0]
  Week 76: number analyzed (Participants) | 180 | 195 | 189
  Week 76 | 95.5 [92.4 to 98.5] | 97.4 [95.2 to 99.6] | 97.9 [95.9 to 99.9]
  Week 80: number analyzed (Participants) | 177 | 203 | 190
  Week 80 | 96.7 [94.1 to 99.3] | 96.6 [94.1 to 99.1] | 98.8 [97.3 to 100.0]
  Week 84: number analyzed (Participants) | 181 | 203 | 192
  Week 84 | 96.1 [93.3 to 98.9] | 98.0 [96.1 to 99.9] | 99.5 [98.4 to 100.0]
  Week 88: number analyzed (Participants) | 179 | 196 | 185
  Week 88 | 96.1 [93.2 to 98.9] | 97.5 [95.3 to 99.6] | 97.7 [95.5 to 99.9]
  Week 92: number analyzed (Participants) | 180 | 199 | 188
  Week 92 | 96.1 [93.2 to 98.9] | 97.0 [94.7 to 99.3] | 98.3 [96.4 to 100.0]
  Week 96: number analyzed (Participants) | 174 | 201 | 187
  Week 96 | 97.1 [94.6 to 99.6] | 96.1 [93.4 to 98.7] | 98.9 [97.3 to 100.0]
  Week 100: number analyzed (Participants) | 185 | 199 | 186
  Week 100 | 96.1 [93.3 to 98.9] | 97.1 [94.8 to 99.4] | 98.4 [96.6 to 100.0]

21. Secondary Outcome: Percentage of Participants Avoiding a Loss of ≥10 Letters in BCVA From Baseline in the Study Eye Over Time, Treatment-Naive Population
Description: as for outcome 20
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96, and 100
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 238 | 245 | 242
Percentage of participants
  Week 4: number analyzed (Participants) | 234 | 241 | 236
  Week 4 | 99.6 [98.7 to 100.0] | 100.0 [100.0 to 100.0] | 99.2 [98.0 to 100.0]
  Week 8: number analyzed (Participants) | 232 | 240 | 234
  Week 8 | 98.3 [96.6 to 100.0] | 100.0 [100.0 to 100.0] | 99.6 [98.8 to 100.0]
  Week 12: number analyzed (Participants) | 230 | 235 | 235
  Week 12 | 99.1 [97.9 to 100.0] | 100.0 [100.0 to 100.0] | 99.6 [98.7 to 100.0]
  Week 16: number analyzed (Participants) | 222 | 229 | 232
  Week 16 | 99.1 [97.9 to 100.0] | 99.1 [97.9 to 100.0] | 100.0 [100.0 to 100.0]
  Week 20: number analyzed (Participants) | 223 | 227 | 229
  Week 20 | 99.1 [97.9 to 100.0] | 98.3 [96.6 to 99.9] | 100.0 [100.0 to 100.0]
  Week 24: number analyzed (Participants) | 219 | 228 | 228
  Week 24 | 99.1 [97.8 to 100.0] | 99.6 [98.7 to 100.0] | 99.1 [97.9 to 100.0]
  Week 28: number analyzed (Participants) | 212 | 224 | 217
  Week 28 | 98.0 [96.1 to 99.9] | 98.7 [97.2 to 100.0] | 98.6 [97.1 to 100.0]
  Week 32: number analyzed (Participants) | 195 | 205 | 209
  Week 32 | 99.5 [98.4 to 100.0] | 98.0 [96.1 to 99.9] | 98.1 [96.2 to 99.9]
  Week 36: number analyzed (Participants) | 194 | 205 | 205
  Week 36 | 97.9 [95.8 to 99.9] | 98.5 [96.8 to 100.0] | 99.0 [97.6 to 100.0]
  Week 40: number analyzed (Participants) | 202 | 204 | 200
  Week 40 | 96.9 [94.5 to 99.3] | 99.0 [97.7 to 100.0] | 97.9 [95.9 to 99.9]
  Week 44: number analyzed (Participants) | 199 | 209 | 202
  Week 44 | 97.4 [95.2 to 99.6] | 97.6 [95.6 to 99.7] | 99.0 [97.6 to 100.0]
  Week 48: number analyzed (Participants) | 195 | 210 | 203
  Week 48 | 97.9 [95.9 to 99.9] | 97.1 [94.9 to 99.4] | 98.5 [96.9 to 100.0]
  Week 52: number analyzed (Participants) | 197 | 209 | 196
  Week 52 | 95.3 [92.3 to 98.3] | 96.2 [93.6 to 98.8] | 96.8 [94.4 to 99.3]
  Week 56: number analyzed (Participants) | 194 | 207 | 198
  Week 56 | 97.4 [95.2 to 99.6] | 97.6 [95.5 to 99.7] | 96.4 [93.9 to 99.0]
  Week 60: number analyzed (Participants) | 200 | 198 | 199
  Week 60 | 96.4 [93.8 to 99.0] | 96.5 [93.9 to 99.0] | 97.9 [95.9 to 99.9]
  Week 64: number analyzed (Participants) | 191 | 202 | 200
  Week 64 | 97.3 [95.0 to 99.6] | 96.5 [94.0 to 99.1] | 97.4 [95.2 to 99.6]
  Week 68: number analyzed (Participants) | 187 | 197 | 193
  Week 68 | 96.8 [94.3 to 99.3] | 96.9 [94.6 to 99.3] | 97.9 [95.9 to 99.9]
  Week 72: number analyzed (Participants) | 186 | 196 | 189
  Week 72 | 95.1 [92.0 to 98.2] | 98.0 [96.1 to 99.9] | 97.3 [95.0 to 99.6]
  Week 76: number analyzed (Participants) | 180 | 195 | 189
  Week 76 | 94.9 [91.7 to 98.2] | 94.3 [91.1 to 97.6] | 97.4 [95.1 to 99.6]
  Week 80: number analyzed (Participants) | 177 | 203 | 190
  Week 80 | 95.0 [91.8 to 98.2] | 95.6 [92.8 to 98.4] | 97.3 [94.9 to 99.6]
  Week 84: number analyzed (Participants) | 181 | 203 | 192
  Week 84 | 94.0 [90.5 to 97.4] | 97.1 [94.7 to 99.4] | 99.5 [98.4 to 100.0]
  Week 88: number analyzed (Participants) | 179 | 196 | 185
  Week 88 | 93.9 [90.4 to 97.4] | 95.4 [92.5 to 98.3] | 96.1 [93.3 to 98.9]
  Week 92: number analyzed (Participants) | 180 | 199 | 188
  Week 92 | 95.0 [91.8 to 98.2] | 96.5 [94.0 to 99.0] | 97.2 [94.9 to 99.6]
  Week 96: number analyzed (Participants) | 174 | 201 | 187
  Week 96 | 96.5 [93.7 to 99.3] | 93.6 [90.2 to 97.0] | 97.2 [94.8 to 99.6]
  Week 100: number analyzed (Participants) | 185 | 199 | 186
  Week 100 | 93.9 [90.4 to 97.4] | 94.6 [91.5 to 97.7] | 97.3 [94.9 to 99.6]

22. Secondary Outcome: Percentage of Participants Avoiding a Loss of ≥5 Letters in BCVA From Baseline in the Study Eye Over Time, Treatment-Naive Population
Description: as for outcome 20
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96, and 100
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 238 | 245 | 242
Percentage of participants
  Week 4: number analyzed (Participants) | 234 | 241 | 236
  Week 4 | 98.7 [97.3 to 100.0] | 97.5 [95.5 to 99.5] | 97.0 [94.9 to 99.2]
  Week 8: number analyzed (Participants) | 232 | 240 | 234
  Week 8 | 96.5 [94.2 to 98.8] | 99.2 [98.1 to 100.0] | 98.3 [96.6 to 99.9]
  Week 12: number analyzed (Participants) | 230 | 235 | 235
  Week 12 | 98.3 [96.6 to 99.9] | 98.7 [97.3 to 100.0] | 98.7 [97.3 to 100.0]
  Week 16: number analyzed (Participants) | 222 | 229 | 232
  Week 16 | 97.8 [95.8 to 99.7] | 98.3 [96.6 to 99.9] | 98.7 [97.3 to 100.0]
  Week 20: number analyzed (Participants) | 223 | 227 | 229
  Week 20 | 97.3 [95.2 to 99.4] | 96.5 [94.2 to 98.9] | 97.8 [95.9 to 99.7]
  Week 24: number analyzed (Participants) | 219 | 228 | 228
  Week 24 | 97.7 [95.7 to 99.7] | 96.1 [93.5 to 98.6] | 96.5 [94.1 to 98.9]
  Week 28: number analyzed (Participants) | 212 | 224 | 217
  Week 28 | 96.6 [94.1 to 99.0] | 97.3 [95.2 to 99.4] | 96.8 [94.5 to 99.1]
  Week 32: number analyzed (Participants) | 195 | 205 | 209
  Week 32 | 97.4 [95.1 to 99.6] | 96.6 [94.1 to 99.1] | 97.6 [95.5 to 99.7]
  Week 36: number analyzed (Participants) | 194 | 205 | 205
  Week 36 | 96.3 [93.6 to 99.0] | 97.6 [95.4 to 99.7] | 98.1 [96.2 to 99.9]
  Week 40: number analyzed (Participants) | 202 | 204 | 200
  Week 40 | 94.5 [91.3 to 97.6] | 95.6 [92.7 to 98.4] | 96.9 [94.5 to 99.3]
  Week 44: number analyzed (Participants) | 199 | 209 | 202
  Week 44 | 95.9 [93.2 to 98.7] | 95.8 [93.1 to 98.5] | 96.5 [93.9 to 99.0]
  Week 48: number analyzed (Participants) | 195 | 210 | 203
  Week 48 | 96.4 [93.8 to 99.0] | 95.7 [93.0 to 98.5] | 97.5 [95.4 to 99.7]
  Week 52: number analyzed (Participants) | 197 | 209 | 196
  Week 52 | 94.3 [91.1 to 97.6] | 94.8 [91.7 to 97.8] | 94.4 [91.2 to 97.6]
  Week 56: number analyzed (Participants) | 194 | 207 | 198
  Week 56 | 95.8 [93.0 to 98.6] | 95.6 [92.9 to 98.4] | 94.4 [91.3 to 97.6]
  Week 60: number analyzed (Participants) | 200 | 198 | 199
  Week 60 | 94.4 [91.2 to 97.6] | 96.0 [93.3 to 98.7] | 96.9 [94.6 to 99.3]
  Week 64: number analyzed (Participants) | 191 | 202 | 200
  Week 64 | 95.2 [92.2 to 98.3] | 96.0 [93.3 to 98.7] | 95.8 [93.0 to 98.6]
  Week 68: number analyzed (Participants) | 187 | 197 | 193
  Week 68 | 94.6 [91.4 to 97.9] | 95.9 [93.2 to 98.7] | 96.4 [93.8 to 99.0]
  Week 72: number analyzed (Participants) | 186 | 196 | 189
  Week 72 | 92.6 [88.8 to 96.3] | 95.9 [93.2 to 98.7] | 94.7 [91.4 to 97.9]
  Week 76: number analyzed (Participants) | 180 | 195 | 189
  Week 76 | 91.1 [86.9 to 95.3] | 93.8 [90.5 to 97.2] | 94.7 [91.5 to 97.9]
  Week 80: number analyzed (Participants) | 177 | 203 | 190
  Week 80 | 92.8 [89.0 to 96.6] | 92.6 [89.1 to 96.2] | 94.2 [90.9 to 97.5]
  Week 84: number analyzed (Participants) | 181 | 203 | 192
  Week 84 | 91.9 [87.9 to 95.8] | 96.1 [93.4 to 98.7] | 96.9 [94.4 to 99.3]
  Week 88: number analyzed (Participants) | 179 | 196 | 185
  Week 88 | 88.3 [83.6 to 93.0] | 91.9 [88.1 to 95.7] | 93.5 [89.9 to 97.0]
  Week 92: number analyzed (Participants) | 180 | 199 | 188
  Week 92 | 92.7 [88.9 to 96.5] | 92.5 [88.9 to 96.2] | 96.7 [94.1 to 99.3]
  Week 96: number analyzed (Participants) | 174 | 201 | 187
  Week 96 | 94.8 [91.4 to 98.1] | 91.5 [87.7 to 95.4] | 95.2 [92.1 to 98.3]
  Week 100: number analyzed (Participants) | 185 | 199 | 186
  Week 100 | 90.6 [86.4 to 94.9] | 88.1 [83.7 to 92.5] | 96.8 [94.2 to 99.3]

23. Secondary Outcome: Percentage of Participants Gaining ≥15 Letters in BCVA From Baseline or Achieving BCVA Snellen Equivalent of 20/20 or Better (BCVA ≥84 Letters) in the Study Eye Averaged Over Weeks 48, 52, and 56, ITT and Treatment-Naive Populations
Description: as for outcome 5
Time Frame: Baseline, average of Weeks 48, 52, and 56
Population: ITT Population and Treatment-Naive Population. Only participants with at least one non-missing, valid assessment at Weeks 48, 52, or 56 were included in the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 271 | 276 | 276
Percentage of participants
  ITT Population | 32.1 [26.6 to 37.6] | 39.1 [33.5 to 44.7] | 37.0 [31.5 to 42.5]
  Treatment-Naive Population: number analyzed (Participants) | 200 | 215 | 212
  Treatment-Naive Population | 31.5 [25.1 to 38.0] | 39.2 [32.8 to 45.5] | 40.2 [33.7 to 46.6]
Statistical Analysis 1: Comparison: A: Faricimab 6 mg Q8W vs C: Aflibercept 2 mg Q8W; This is the difference in percentage of participants in Arm A: Faricimab 6 mg Q8W minus Arm C: Aflibercept 2 mg Q8W for the ITT Population; Test type: Other; Difference in CMH Weighted Percentage = -4.9, 95% CI 2-sided [-12.6 to 2.9]
Statistical Analysis 2: Comparison: B: Faricimab 6 mg PTI vs C: Aflibercept 2 mg Q8W; This is the difference in percentage of participants in Arm B: Faricimab 6 mg PTI minus Arm C: Aflibercept 2 mg Q8W for the ITT Population; Test type: Other; Difference in CMH Weighted Percentage = 2.0, 95% CI 2-sided [-5.9 to 9.8]
Statistical Analysis 3: Comparison: A: Faricimab 6 mg Q8W vs C: Aflibercept 2 mg Q8W; This is the difference in percentage of participants in Arm A: Faricimab 6 mg Q8W minus Arm C: Aflibercept 2 mg Q8W for the Treatment-Naive Population; Test type: Other; Difference in CMH Weighted Percentage = -8.6, 95% CI 2-sided [-17.8 to 0.5]
Statistical Analysis 4: Comparison: B: Faricimab 6 mg PTI vs C: Aflibercept 2 mg Q8W; This is the difference in percentage of participants in Arm B: Faricimab 6 mg PTI minus Arm C: Aflibercept 2 mg Q8W for the Treatment-Naive Population; Test type: Other; Difference in CMH Weighted Percentage = -0.9, 95% CI 2-sided [-9.9 to 8.2]

24. Secondary Outcome: Percentage of Participants Gaining ≥15 Letters in BCVA From Baseline or Achieving BCVA Snellen Equivalent of 20/20 or Better (BCVA ≥84 Letters) in the Study Eye Over Time, ITT Population
Description: as for outcome 6
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96, and 100
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 315 | 313 | 312
Percentage of participants
  Week 4: number analyzed (Participants) | 310 | 308 | 306
  Week 4 | 8.7 [5.6 to 11.8] | 14.6 [10.8 to 18.4] | 13.3 [9.6 to 17.0]
  Week 8: number analyzed (Participants) | 309 | 308 | 304
  Week 8 | 15.3 [11.3 to 19.3] | 20.1 [15.9 to 24.4] | 19.9 [15.6 to 24.3]
  Week 12: number analyzed (Participants) | 305 | 303 | 302
  Week 12 | 17.9 [13.6 to 22.1] | 25.7 [21.1 to 30.4] | 25.3 [20.6 to 30.0]
  Week 16: number analyzed (Participants) | 296 | 296 | 299
  Week 16 | 24.1 [19.2 to 28.9] | 29.1 [24.2 to 34.0] | 25.2 [20.5 to 30.0]
  Week 20: number analyzed (Participants) | 294 | 292 | 296
  Week 20 | 30.1 [24.9 to 35.2] | 30.8 [25.6 to 35.9] | 27.7 [22.8 to 32.6]
  Week 24: number analyzed (Participants) | 292 | 293 | 294
  Week 24 | 31.3 [26.0 to 36.5] | 37.8 [32.5 to 43.2] | 30.9 [25.7 to 36.0]
  Week 28: number analyzed (Participants) | 283 | 287 | 284
  Week 28 | 28.3 [23.1 to 33.5] | 32.6 [27.4 to 37.8] | 35.0 [29.7 to 40.4]
  Week 32: number analyzed (Participants) | 267 | 268 | 275
  Week 32 | 33.7 [28.0 to 39.3] | 38.8 [33.2 to 44.4] | 31.0 [25.8 to 36.2]
  Week 36: number analyzed (Participants) | 268 | 268 | 268
  Week 36 | 29.6 [24.1 to 35.0] | 42.4 [36.8 to 48.1] | 35.6 [30.0 to 41.1]
  Week 40: number analyzed (Participants) | 275 | 269 | 263
  Week 40 | 32.9 [27.4 to 38.5] | 40.4 [34.7 to 46.2] | 33.8 [28.2 to 39.4]
  Week 44: number analyzed (Participants) | 268 | 269 | 266
  Week 44 | 32.1 [26.5 to 37.7] | 39.7 [34.1 to 45.3] | 39.9 [34.2 to 45.7]
  Week 48: number analyzed (Participants) | 264 | 266 | 266
  Week 48 | 35.7 [30.0 to 41.5] | 41.8 [36.1 to 47.6] | 41.7 [36.0 to 47.4]
  Week 52: number analyzed (Participants) | 264 | 267 | 253
  Week 52 | 35.7 [29.9 to 41.4] | 40.2 [34.5 to 45.8] | 41.7 [35.8 to 47.6]
  Week 56: number analyzed (Participants) | 260 | 263 | 256
  Week 56 | 43.1 [37.1 to 49.1] | 42.6 [36.7 to 48.4] | 35.7 [30.1 to 41.4]
  Week 60: number analyzed (Participants) | 270 | 261 | 261
  Week 60 | 39.5 [33.7 to 45.3] | 45.0 [39.1 to 51.0] | 40.6 [34.8 to 46.3]
  Week 64: number analyzed (Participants) | 259 | 263 | 263
  Week 64 | 42.1 [36.1 to 48.1] | 44.0 [38.2 to 49.8] | 37.9 [32.1 to 43.7]
  Week 68: number analyzed (Participants) | 251 | 257 | 253
  Week 68 | 42.2 [36.2 to 48.2] | 45.6 [39.7 to 51.6] | 40.3 [34.5 to 46.2]
  Week 72: number analyzed (Participants) | 253 | 257 | 251
  Week 72 | 39.8 [33.9 to 45.8] | 40.5 [34.8 to 46.2] | 37.7 [31.8 to 43.6]
  Week 76: number analyzed (Participants) | 247 | 253 | 251
  Week 76 | 42.2 [36.1 to 48.4] | 47.7 [41.8 to 53.5] | 42.9 [36.8 to 49.0]
  Week 80: number analyzed (Participants) | 247 | 259 | 251
  Week 80 | 42.9 [36.8 to 49.0] | 44.8 [39.0 to 50.5] | 41.9 [35.9 to 47.8]
  Week 84: number analyzed (Participants) | 248 | 260 | 252
  Week 84 | 42.4 [36.3 to 48.5] | 43.0 [37.2 to 48.7] | 42.9 [36.9 to 48.9]
  Week 88: number analyzed (Participants) | 245 | 256 | 247
  Week 88 | 41.2 [35.1 to 47.3] | 41.7 [36.1 to 47.4] | 40.0 [34.1 to 46.0]
  Week 92: number analyzed (Participants) | 248 | 258 | 248
  Week 92 | 42.5 [36.4 to 48.5] | 43.6 [37.8 to 49.4] | 42.7 [36.7 to 48.7]
  Week 96: number analyzed (Participants) | 242 | 259 | 245
  Week 96 | 44.9 [38.7 to 51.1] | 42.4 [36.6 to 48.1] | 42.7 [36.6 to 48.7]
  Week 100: number analyzed (Participants) | 254 | 258 | 247
  Week 100 | 43.5 [37.5 to 49.6] | 41.8 [36.1 to 47.5] | 44.7 [38.6 to 50.8]

25. Secondary Outcome: Percentage of Participants Gaining ≥15 Letters in BCVA From Baseline or Achieving BCVA Snellen Equivalent of 20/20 or Better (BCVA ≥84 Letters) in the Study Eye Over Time, Treatment-Naive Population
Description: as for outcome 11
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96, and 100
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 238 | 245 | 242
Percentage of participants
  Week 4: number analyzed (Participants) | 234 | 241 | 236
  Week 4 | 9.8 [6.0 to 13.5] | 17.0 [12.4 to 21.6] | 15.2 [10.7 to 19.8]
  Week 8: number analyzed (Participants) | 232 | 240 | 234
  Week 8 | 16.0 [11.3 to 20.7] | 20.9 [16.1 to 25.7] | 22.2 [16.9 to 27.4]
  Week 12: number analyzed (Participants) | 230 | 235 | 235
  Week 12 | 19.2 [14.1 to 24.2] | 25.6 [20.3 to 30.9] | 28.5 [22.9 to 34.1]
  Week 16: number analyzed (Participants) | 222 | 229 | 232
  Week 16 | 24.9 [19.2 to 30.5] | 29.5 [23.8 to 35.2] | 27.9 [22.2 to 33.6]
  Week 20: number analyzed (Participants) | 223 | 227 | 229
  Week 20 | 31.0 [25.0 to 37.0] | 30.4 [24.6 to 36.1] | 30.6 [24.8 to 36.4]
  Week 24: number analyzed (Participants) | 219 | 228 | 228
  Week 24 | 32.5 [26.3 to 38.7] | 38.2 [32.1 to 44.3] | 33.3 [27.3 to 39.4]
  Week 28: number analyzed (Participants) | 212 | 224 | 217
  Week 28 | 26.9 [20.9 to 32.9] | 32.0 [26.2 to 37.8] | 38.5 [32.2 to 44.8]
  Week 32: number analyzed (Participants) | 195 | 205 | 209
  Week 32 | 33.3 [26.7 to 39.9] | 40.5 [34.0 to 46.9] | 35.4 [29.0 to 41.7]
  Week 36: number analyzed (Participants) | 194 | 205 | 205
  Week 36 | 29.5 [23.1 to 36.0] | 44.8 [38.3 to 51.3] | 38.4 [31.9 to 44.8]
  Week 40: number analyzed (Participants) | 202 | 204 | 200
  Week 40 | 31.5 [25.1 to 37.9] | 41.1 [34.5 to 47.7] | 37.1 [30.4 to 43.7]
  Week 44: number analyzed (Participants) | 199 | 209 | 202
  Week 44 | 31.1 [24.7 to 37.6] | 42.9 [36.4 to 49.5] | 42.7 [36.0 to 49.4]
  Week 48: number analyzed (Participants) | 195 | 210 | 203
  Week 48 | 37.5 [30.7 to 44.3] | 41.9 [35.3 to 48.5] | 44.9 [38.2 to 51.6]
  Week 52: number analyzed (Participants) | 197 | 209 | 196
  Week 52 | 35.5 [28.9 to 42.2] | 39.2 [32.8 to 45.6] | 43.8 [36.9 to 50.6]
  Week 56: number analyzed (Participants) | 194 | 207 | 198
  Week 56 | 43.3 [36.3 to 50.3] | 43.1 [36.5 to 49.7] | 38.9 [32.2 to 45.5]
  Week 60: number analyzed (Participants) | 200 | 198 | 199
  Week 60 | 39.4 [32.6 to 46.2] | 46.7 [39.9 to 53.5] | 43.6 [36.8 to 50.4]
  Week 64: number analyzed (Participants) | 191 | 202 | 200
  Week 64 | 43.0 [36.0 to 50.0] | 46.4 [39.8 to 53.1] | 38.7 [32.0 to 45.3]
  Week 68: number analyzed (Participants) | 187 | 197 | 193
  Week 68 | 43.7 [36.6 to 50.7] | 47.9 [41.1 to 54.7] | 42.2 [35.4 to 49.0]
  Week 72: number analyzed (Participants) | 186 | 196 | 189
  Week 72 | 40.7 [33.7 to 47.8] | 42.1 [35.5 to 48.7] | 39.3 [32.5 to 46.2]
  Week 76: number analyzed (Participants) | 180 | 195 | 189
  Week 76 | 44.6 [37.3 to 51.8] | 49.9 [43.3 to 56.6] | 43.8 [36.8 to 50.8]
  Week 80: number analyzed (Participants) | 177 | 203 | 190
  Week 80 | 44.6 [37.3 to 51.8] | 46.6 [40.1 to 53.2] | 46.1 [39.1 to 53.1]
  Week 84: number analyzed (Participants) | 181 | 203 | 192
  Week 84 | 42.7 [35.6 to 49.9] | 45.2 [38.6 to 51.7] | 45.7 [38.7 to 52.7]
  Week 88: number analyzed (Participants) | 179 | 196 | 185
  Week 88 | 41.3 [34.2 to 48.5] | 42.7 [36.3 to 49.2] | 42.5 [35.5 to 49.6]
  Week 92: number analyzed (Participants) | 180 | 199 | 188
  Week 92 | 43.4 [36.3 to 50.6] | 45.5 [38.9 to 52.1] | 43.9 [36.9 to 50.8]
  Week 96: number analyzed (Participants) | 174 | 201 | 187
  Week 96 | 46.7 [39.3 to 54.1] | 43.6 [37.2 to 50.1] | 44.7 [37.7 to 51.8]
  Week 100: number analyzed (Participants) | 185 | 199 | 186
  Week 100 | 44.1 [37.0 to 51.3] | 44.4 [37.9 to 50.9] | 45.8 [38.8 to 52.9]

26. Secondary Outcome: Percentage of Participants With BCVA Snellen Equivalent of 20/40 or Better (BCVA ≥69 Letters) in the Study Eye Averaged Over Weeks 48, 52, and 56, ITT and Treatment-Naive Populations
Description: BCVA was measured on the ETDRS chart at a starting distance of 4 meters. The BCVA letter score ranges from 0 to 100 (best score), and a gain in BCVA from baseline indicates an improvement in visual acuity. For each participant, an average BCVA value was calculated across the three visits, and this averaged value was then used to determine if the endpoint was met. The results were summarized as the percentage of participants per treatment arm who met the endpoint. The weighted estimates of the percentage of participants were based on the Cochran-Mantel Haenszel (CMH) weights stratified by baseline BCVA (≥69 vs. <69 letters), prior IVT anti-VEGF therapy (yes vs. no), and region (U.S. and Canada vs. rest of the world). Treatment policy strategy and hypothetical strategy were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were not imputed. Invalid BCVA values were excluded. 95% confidence interval (CI) is a rounding of 95.04% CI.
Time Frame: Baseline, average of Weeks 48, 52, and 56
Population: as for outcome 23
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 271 | 276 | 276
Percentage of participants
  ITT Population | 71.6 [66.5 to 76.6] | 77.1 [72.4 to 81.8] | 74.8 [69.9 to 79.6]
  Treatment-Naive Population: number analyzed (Participants) | 200 | 215 | 212
  Treatment-Naive Population | 72.7 [66.9 to 78.5] | 75.7 [70.3 to 81.1] | 77.4 [72.2 to 82.7]
Statistical Analysis 1: Comparison: A: Faricimab 6 mg Q8W vs C: Aflibercept 2 mg Q8W; [analysis description as in outcome 23, analysis 1]; Test type: Other; Difference in CMH Weighted Percentage = -3.2, 95% CI 2-sided [-10.2 to 3.8]
Statistical Analysis 2: Comparison: B: Faricimab 6 mg PTI vs C: Aflibercept 2 mg Q8W; [analysis description as in outcome 23, analysis 2]; Test type: Other; Difference in CMH Weighted Percentage = 2.4, 95% CI 2-sided [-4.3 to 9.2]
Statistical Analysis 3: Comparison: A: Faricimab 6 mg Q8W vs C: Aflibercept 2 mg Q8W; [analysis description as in outcome 23, analysis 3]; Test type: Other; Difference in CMH Weighted Percentage = -4.7, 95% CI 2-sided [-12.6 to 3.1]
Statistical Analysis 4: Comparison: B: Faricimab 6 mg PTI vs C: Aflibercept 2 mg Q8W; [analysis description as in outcome 23, analysis 4]; Test type: Other; Difference in CMH Weighted Percentage = -1.3, 95% CI 2-sided [-8.9 to 6.4]

27. Secondary Outcome: Percentage of Participants With BCVA Snellen Equivalent of 20/40 or Better (BCVA ≥69 Letters) in the Study Eye Over Time, ITT Population
Description: Best Corrected Visual Acuity (BCVA) was measured on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart at a starting distance of 4 meters. The BCVA letter score ranges from 0 to 100 (best score), and a gain in BCVA letter score from baseline indicates an improvement in visual acuity. The weighted estimates of the percentage of participants were based on the Cochran-Mantel Haenszel (CMH) weights stratified by baseline BCVA (≥69 vs. <69 letters), prior IVT anti-VEGF therapy (yes vs. no), and region (U.S. and Canada vs. rest of the world; Asia and rest of the world were combined). Treatment policy strategy (i.e., all observed values used) and hypothetical strategy (i.e., all values censored after the occurrence of the intercurrent event) were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were not imputed. Invalid BCVA values were excluded. 95% confidence interval (CI) is a rounding of 95.04% CI.
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96, and 100
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 315 | 313 | 312
Percentage of participants
  Week 4: number analyzed (Participants) | 310 | 308 | 306
  Week 4 | 53.3 [48.4 to 58.1] | 60.0 [55.1 to 64.8] | 57.5 [52.6 to 62.4]
  Week 8: number analyzed (Participants) | 309 | 308 | 304
  Week 8 | 60.0 [55.1 to 64.9] | 65.5 [60.8 to 70.1] | 66.1 [61.4 to 70.8]
  Week 12: number analyzed (Participants) | 305 | 303 | 302
  Week 12 | 64.4 [59.4 to 69.3] | 69.3 [64.6 to 74.0] | 68.8 [64.1 to 73.6]
  Week 16: number analyzed (Participants) | 296 | 296 | 299
  Week 16 | 66.1 [61.1 to 71.2] | 70.6 [65.8 to 75.3] | 74.7 [70.1 to 79.2]
  Week 20: number analyzed (Participants) | 294 | 292 | 296
  Week 20 | 70.3 [65.4 to 75.3] | 69.7 [64.9 to 74.6] | 70.3 [65.5 to 75.1]
  Week 24: number analyzed (Participants) | 292 | 293 | 294
  Week 24 | 71.0 [66.1 to 76.0] | 76.0 [71.4 to 80.6] | 71.0 [66.3 to 75.8]
  Week 28: number analyzed (Participants) | 283 | 287 | 284
  Week 28 | 71.5 [66.5 to 76.4] | 74.5 [69.9 to 79.1] | 75.1 [70.4 to 79.8]
  Week 32: number analyzed (Participants) | 267 | 268 | 275
  Week 32 | 71.4 [66.3 to 76.5] | 74.1 [69.2 to 79.0] | 74.9 [70.1 to 79.7]
  Week 36: number analyzed (Participants) | 268 | 268 | 268
  Week 36 | 71.8 [66.8 to 76.9] | 79.4 [74.7 to 84.1] | 73.2 [68.1 to 78.2]
  Week 40: number analyzed (Participants) | 275 | 269 | 263
  Week 40 | 69.3 [64.2 to 74.4] | 75.1 [70.2 to 80.1] | 73.6 [68.5 to 78.7]
  Week 44: number analyzed (Participants) | 268 | 269 | 266
  Week 44 | 70.6 [65.4 to 75.7] | 77.7 [72.9 to 82.5] | 73.4 [68.3 to 78.4]
  Week 48: number analyzed (Participants) | 264 | 266 | 266
  Week 48 | 73.4 [68.4 to 78.4] | 78.3 [73.6 to 83.0] | 72.7 [67.6 to 77.8]
  Week 52: number analyzed (Participants) | 264 | 267 | 253
  Week 52 | 69.3 [63.9 to 74.6] | 76.6 [71.7 to 81.4] | 75.2 [70.2 to 80.2]
  Week 56: number analyzed (Participants) | 260 | 263 | 256
  Week 56 | 74.9 [69.9 to 79.9] | 79.5 [74.8 to 84.2] | 72.2 [67.0 to 77.4]
  Week 60: number analyzed (Participants) | 270 | 261 | 261
  Week 60 | 71.8 [66.6 to 76.9] | 76.6 [71.6 to 81.5] | 75.9 [70.9 to 80.9]
  Week 64: number analyzed (Participants) | 259 | 263 | 263
  Week 64 | 74.9 [69.8 to 79.9] | 76.2 [71.4 to 81.0] | 71.4 [66.3 to 76.5]
  Week 68: number analyzed (Participants) | 251 | 257 | 253
  Week 68 | 74.4 [69.2 to 79.7] | 78.0 [73.2 to 82.8] | 73.9 [68.9 to 78.9]
  Week 72: number analyzed (Participants) | 253 | 257 | 251
  Week 72 | 73.9 [68.6 to 79.1] | 76.8 [72.0 to 81.7] | 71.0 [65.8 to 76.1]
  Week 76: number analyzed (Participants) | 247 | 253 | 251
  Week 76 | 72.6 [67.2 to 78.0] | 77.0 [72.0 to 82.0] | 76.0 [71.1 to 81.0]
  Week 80: number analyzed (Participants) | 247 | 259 | 251
  Week 80 | 74.6 [69.3 to 79.9] | 77.5 [72.5 to 82.4] | 73.8 [68.7 to 78.9]
  Week 84: number analyzed (Participants) | 248 | 260 | 252
  Week 84 | 73.7 [68.4 to 79.1] | 77.2 [72.3 to 82.1] | 77.3 [72.5 to 82.2]
  Week 88: number analyzed (Participants) | 245 | 256 | 247
  Week 88 | 72.2 [66.7 to 77.7] | 76.2 [71.2 to 81.3] | 73.3 [68.0 to 78.5]
  Week 92: number analyzed (Participants) | 248 | 258 | 248
  Week 92 | 75.3 [70.0 to 80.6] | 78.4 [73.4 to 83.3] | 77.4 [72.6 to 82.2]
  Week 96: number analyzed (Participants) | 242 | 259 | 245
  Week 96 | 75.9 [70.6 to 81.2] | 74.3 [69.0 to 79.5] | 73.4 [68.3 to 78.5]
  Week 100: number analyzed (Participants) | 254 | 258 | 247
  Week 100 | 75.9 [70.7 to 81.1] | 70.3 [64.9 to 75.7] | 75.7 [70.8 to 80.7]

28. Secondary Outcome: Percentage of Participants With BCVA Snellen Equivalent of 20/40 or Better (BCVA ≥69 Letters) in the Study Eye Over Time, Treatment-Naive Population
Description: Best Corrected Visual Acuity (BCVA) was measured on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart at a starting distance of 4 meters. The BCVA letter score ranges from 0 to 100 (best score), and a gain in BCVA letter score from baseline indicates an improvement in visual acuity. The weighted estimates of the percentage of participants were based on the Cochran-Mantel Haenszel (CMH) weights stratified by baseline BCVA (≥69 vs. <69 letters) and region (U.S. and Canada vs. rest of the world; Asia and rest of the world were combined). Treatment policy strategy (i.e., all observed values used) and hypothetical strategy (i.e., all values censored after the occurrence of the intercurrent event) were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were not imputed. Invalid BCVA values were excluded from analysis. 95% confidence interval (CI) is a rounding of 95.04% CI.
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96, and 100
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 238 | 245 | 242
Percentage of participants
  Week 4: number analyzed (Participants) | 234 | 241 | 236
  Week 4 | 55.7 [50.1 to 61.2] | 60.4 [55.0 to 65.8] | 60.4 [54.9 to 65.9]
  Week 8: number analyzed (Participants) | 232 | 240 | 234
  Week 8 | 62.0 [56.5 to 67.6] | 66.5 [61.3 to 71.6] | 69.6 [64.3 to 74.8]
  Week 12: number analyzed (Participants) | 230 | 235 | 235
  Week 12 | 66.2 [60.5 to 71.8] | 69.3 [64.1 to 74.5] | 70.6 [65.3 to 75.9]
  Week 16: number analyzed (Participants) | 222 | 229 | 232
  Week 16 | 68.5 [62.8 to 74.2] | 68.5 [63.1 to 74.0] | 75.8 [70.8 to 80.9]
  Week 20: number analyzed (Participants) | 223 | 227 | 229
  Week 20 | 72.7 [67.1 to 78.2] | 67.8 [62.2 to 73.4] | 72.0 [66.7 to 77.3]
  Week 24: number analyzed (Participants) | 219 | 228 | 228
  Week 24 | 73.7 [68.2 to 79.3] | 74.5 [69.2 to 79.8] | 72.6 [67.3 to 77.9]
  Week 28: number analyzed (Participants) | 212 | 224 | 217
  Week 28 | 73.7 [68.2 to 79.3] | 73.1 [67.8 to 78.4] | 77.0 [71.8 to 82.2]
  Week 32: number analyzed (Participants) | 195 | 205 | 209
  Week 32 | 71.8 [65.8 to 77.7] | 72.4 [66.7 to 78.1] | 75.8 [70.4 to 81.2]
  Week 36: number analyzed (Participants) | 194 | 205 | 205
  Week 36 | 74.7 [68.9 to 80.5] | 79.4 [74.0 to 84.7] | 73.4 [67.6 to 79.1]
  Week 40: number analyzed (Participants) | 202 | 204 | 200
  Week 40 | 70.6 [64.7 to 76.6] | 74.6 [68.9 to 80.3] | 75.8 [70.2 to 81.4]
  Week 44: number analyzed (Participants) | 199 | 209 | 202
  Week 44 | 71.1 [65.2 to 77.1] | 76.9 [71.3 to 82.4] | 76.4 [70.8 to 82.0]
  Week 48: number analyzed (Participants) | 195 | 210 | 203
  Week 48 | 74.3 [68.6 to 80.0] | 75.7 [70.2 to 81.2] | 75.3 [69.8 to 80.9]
  Week 52: number analyzed (Participants) | 197 | 209 | 196
  Week 52 | 71.7 [65.6 to 77.7] | 74.4 [68.7 to 80.1] | 77.5 [71.9 to 83.0]
  Week 56: number analyzed (Participants) | 194 | 207 | 198
  Week 56 | 76.9 [71.3 to 82.5] | 77.9 [72.4 to 83.4] | 74.0 [68.2 to 79.7]
  Week 60: number analyzed (Participants) | 200 | 198 | 199
  Week 60 | 73.4 [67.5 to 79.3] | 75.2 [69.4 to 81.0] | 78.3 [72.8 to 83.8]
  Week 64: number analyzed (Participants) | 191 | 202 | 200
  Week 64 | 77.0 [71.2 to 82.7] | 75.5 [69.9 to 81.0] | 74.4 [68.9 to 80.0]
  Week 68: number analyzed (Participants) | 187 | 197 | 193
  Week 68 | 77.6 [71.7 to 83.5] | 77.9 [72.4 to 83.3] | 75.5 [69.9 to 81.0]
  Week 72: number analyzed (Participants) | 186 | 196 | 189
  Week 72 | 76.7 [70.7 to 82.6] | 75.9 [70.3 to 81.4] | 74.5 [68.9 to 80.1]
  Week 76: number analyzed (Participants) | 180 | 195 | 189
  Week 76 | 72.7 [66.3 to 79.1] | 75.8 [70.1 to 81.5] | 78.0 [72.6 to 83.3]
  Week 80: number analyzed (Participants) | 177 | 203 | 190
  Week 80 | 76.4 [70.2 to 82.6] | 76.8 [71.2 to 82.5] | 76.5 [70.9 to 82.1]
  Week 84: number analyzed (Participants) | 181 | 203 | 192
  Week 84 | 75.7 [69.5 to 81.9] | 77.8 [72.3 to 83.3] | 77.8 [72.4 to 83.2]
  Week 88: number analyzed (Participants) | 179 | 196 | 185
  Week 88 | 71.8 [65.2 to 78.3] | 75.7 [69.9 to 81.5] | 76.0 [70.1 to 81.9]
  Week 92: number analyzed (Participants) | 180 | 199 | 188
  Week 92 | 75.9 [69.7 to 82.1] | 77.7 [71.9 to 83.4] | 79.9 [74.7 to 85.2]
  Week 96: number analyzed (Participants) | 174 | 201 | 187
  Week 96 | 77.3 [71.1 to 83.4] | 73.5 [67.4 to 79.5] | 75.5 [69.9 to 81.2]
  Week 100: number analyzed (Participants) | 185 | 199 | 186
  Week 100 | 77.6 [71.6 to 83.6] | 70.8 [64.6 to 76.9] | 77.0 [71.4 to 82.5]

29. Secondary Outcome: Percentage of Participants With BCVA Snellen Equivalent of 20/200 or Worse (BCVA ≤38 Letters) in the Study Eye Averaged Over Weeks 48, 52, and 56, ITT and Treatment-Naive Populations
Description: as for outcome 5
Time Frame: Baseline, average of Weeks 48, 52, and 56
Population: as for outcome 23
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 271 | 276 | 276
Percentage of participants
  ITT Population | 2.3 [0.5 to 4.1] | 1.9 [0.3 to 3.5] | 1.7 [0.3 to 3.2]
  Treatment-Naive Population: number analyzed (Participants) | 200 | 215 | 212
  Treatment-Naive Population | 2.6 [0.4 to 4.8] | 1.9 [0.1 to 3.7] | 1.8 [0.1 to 3.5]
Statistical Analysis 1: Comparison: A: Faricimab 6 mg Q8W vs C: Aflibercept 2 mg Q8W; [analysis description as in outcome 23, analysis 1]; Test type: Other; Difference in CMH Weighted Percentage = 0.6, 95% CI 2-sided [-1.8 to 2.9]
Statistical Analysis 2: Comparison: B: Faricimab 6 mg PTI vs C: Aflibercept 2 mg Q8W; [analysis description as in outcome 23, analysis 2]; Test type: Other; Difference in CMH Weighted Percentage = 0.0, 95% CI 2-sided [-2.2 to 2.3]
Statistical Analysis 3: Comparison: A: Faricimab 6 mg Q8W vs C: Aflibercept 2 mg Q8W; [analysis description as in outcome 23, analysis 3]; Test type: Other; Difference in CMH Weighted Percentage = 0.8, 95% CI 2-sided [-2.0 to 3.6]
Statistical Analysis 4: Comparison: B: Faricimab 6 mg PTI vs C: Aflibercept 2 mg Q8W; [analysis description as in outcome 23, analysis 4]; Test type: Other; Difference in CMH Weighted Percentage = 0.0, 95% CI 2-sided [-2.6 to 2.5]

30. Secondary Outcome: Percentage of Participants With BCVA Snellen Equivalent of 20/200 or Worse (BCVA ≤38 Letters) in the Study Eye Over Time, ITT Population
Description: Best Corrected Visual Acuity (BCVA) was measured on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart at a starting distance of 4 meters. The BCVA letter score ranges from 0 to 100 (best score), and a gain in BCVA letter score from baseline indicates an improvement invisual acuity. The weighted estimates of the percentage of participants were based on the Cochran-Mantel Haenszel (CMH) weights stratified by baseline BCVA (≥64 vs. <64 letters), prior IVT anti-VEGF therapy (yes vs. no), and region (U.S. and Canada vs. rest of the world; Asia and rest of the world were combined). Treatment policy strategy (i.e., all observed values used) and hypothetical strategy (i.e., all values censored after the occurrence of the intercurrent event) were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were not imputed. Invalid BCVA values were excluded from analysis. 95% confidence interval (CI) is a rounding of 95.04% CI.
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96, and 100
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 315 | 313 | 312
Percentage of participants
  Week 4: number analyzed (Participants) | 310 | 308 | 306
  Week 4 | 1.9 [0.4 to 3.4] | 2.6 [0.9 to 4.3] | 1.6 [0.2 to 3.0]
  Week 8: number analyzed (Participants) | 309 | 308 | 304
  Week 8 | 2.0 [0.4 to 3.5] | 3.0 [1.1 to 4.8] | 2.0 [0.4 to 3.5]
  Week 12: number analyzed (Participants) | 305 | 303 | 302
  Week 12 | 1.6 [0.2 to 3.0] | 2.0 [0.5 to 3.5] | 1.6 [0.2 to 3.0]
  Week 16: number analyzed (Participants) | 296 | 296 | 299
  Week 16 | 0.7 [0.0 to 1.6] | 2.1 [0.5 to 3.7] | 1.6 [0.2 to 3.0]
  Week 20: number analyzed (Participants) | 294 | 292 | 296
  Week 20 | 1.3 [0.0 to 2.7] | 1.7 [0.3 to 3.2] | 1.7 [0.2 to 3.1]
  Week 24: number analyzed (Participants) | 292 | 293 | 294
  Week 24 | 0.7 [0.0 to 1.6] | 1.7 [0.3 to 3.2] | 1.7 [0.3 to 3.1]
  Week 28: number analyzed (Participants) | 283 | 287 | 284
  Week 28 | 1.4 [0.1 to 2.8] | 1.4 [0.1 to 2.8] | 1.4 [0.1 to 2.7]
  Week 32: number analyzed (Participants) | 267 | 268 | 275
  Week 32 | 1.1 [0.0 to 2.4] | 1.2 [0.0 to 2.4] | 1.8 [0.2 to 3.3]
  Week 36: number analyzed (Participants) | 268 | 268 | 268
  Week 36 | 1.6 [0.1 to 3.1] | 1.6 [0.1 to 3.1] | 1.5 [0.1 to 3.0]
  Week 40: number analyzed (Participants) | 275 | 269 | 263
  Week 40 | 1.5 [0.1 to 3.0] | 2.3 [0.5 to 4.1] | 1.5 [0.1 to 2.9]
  Week 44: number analyzed (Participants) | 268 | 269 | 266
  Week 44 | 3.1 [1.0 to 5.2] | 1.9 [0.3 to 3.6] | 1.4 [0.1 to 2.8]
  Week 48: number analyzed (Participants) | 264 | 266 | 266
  Week 48 | 1.6 [0.1 to 3.1] | 2.3 [0.5 to 4.1] | 1.8 [0.3 to 3.3]
  Week 52: number analyzed (Participants) | 264 | 267 | 253
  Week 52 | 2.0 [0.3 to 3.8] | 1.5 [0.1 to 3.0] | 1.5 [0.1 to 2.9]
  Week 56: number analyzed (Participants) | 260 | 263 | 256
  Week 56 | 1.5 [0.0 to 3.0] | 1.6 [0.1 to 3.1] | 1.9 [0.3 to 3.5]
  Week 60: number analyzed (Participants) | 270 | 261 | 261
  Week 60 | 1.9 [0.3 to 3.5] | 1.2 [0.0 to 2.5] | 1.4 [0.1 to 2.8]
  Week 64: number analyzed (Participants) | 259 | 263 | 263
  Week 64 | 1.2 [0.0 to 2.6] | 2.5 [0.6 to 4.3] | 1.8 [0.2 to 3.3]
  Week 68: number analyzed (Participants) | 251 | 257 | 253
  Week 68 | 1.3 [0.0 to 2.7] | 2.4 [0.6 to 4.3] | 1.8 [0.3 to 3.4]
  Week 72: number analyzed (Participants) | 253 | 257 | 251
  Week 72 | 1.3 [0.0 to 2.7] | 1.6 [0.1 to 3.1] | 1.5 [0.1 to 2.9]
  Week 76: number analyzed (Participants) | 247 | 253 | 251
  Week 76 | 0.9 [0.0 to 2.1] | 1.6 [0.1 to 3.2] | 3.4 [1.3 to 5.6]
  Week 80: number analyzed (Participants) | 247 | 259 | 251
  Week 80 | 0.9 [0.0 to 2.1] | 2.0 [0.3 to 3.8] | 3.0 [1.0 to 5.0]
  Week 84: number analyzed (Participants) | 248 | 260 | 252
  Week 84 | 0.9 [0.0 to 2.1] | 1.6 [0.1 to 3.2] | 1.0 [0.0 to 2.2]
  Week 88: number analyzed (Participants) | 245 | 256 | 247
  Week 88 | 1.3 [0.0 to 2.7] | 1.7 [0.1 to 3.2] | 2.0 [0.3 to 3.8]
  Week 92: number analyzed (Participants) | 248 | 258 | 248
  Week 92 | 2.2 [0.3 to 4.0] | 2.1 [0.4 to 3.9] | 2.8 [0.8 to 4.8]
  Week 96: number analyzed (Participants) | 242 | 259 | 245
  Week 96 | 1.7 [0.1 to 3.4] | 2.1 [0.3 to 3.8] | 0.9 [0.0 to 2.1]
  Week 100: number analyzed (Participants) | 254 | 258 | 247
  Week 100 | 2.5 [0.5 to 4.5] | 2.1 [0.3 to 3.8] | 1.2 [0.0 to 2.6]

31. Secondary Outcome: Percentage of Participants With BCVA Snellen Equivalent of 20/200 or Worse (BCVA ≤38 Letters) in the Study Eye Over Time, Treatment-Naive Population
Description: Best Corrected Visual Acuity (BCVA) was measured on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart at a starting distance of 4 meters. The BCVA letter score ranges from 0 to 100 (best score attainable), and a gain in BCVA letter score from baseline indicates an improvement in visual acuity. The weighted estimates of the percentage of participants were based on the Cochran-Mantel Haenszel (CMH) weights stratified by baseline BCVA (≥64 vs. <64 letters) and region (U.S. and Canada vs. rest of the world; Asia and rest of the world were combined). Treatment policy strategy (i.e., all observed values used) and hypothetical strategy (i.e., all values censored after the occurrence of the intercurrent event) were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were not imputed. Invalid BCVA values were excluded from analysis. 95% confidence interval (CI) is a rounding of 95.04% CI.
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96, and 100
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 238 | 245 | 242
Percentage of participants
  Week 4: number analyzed (Participants) | 234 | 241 | 236
  Week 4 | 1.7 [0.1 to 3.3] | 2.9 [0.8 to 4.9] | 1.3 [0.0 to 2.7]
  Week 8: number analyzed (Participants) | 232 | 240 | 234
  Week 8 | 2.2 [0.3 to 4.0] | 3.3 [1.1 to 5.5] | 2.1 [0.3 to 3.9]
  Week 12: number analyzed (Participants) | 230 | 235 | 235
  Week 12 | 1.3 [0.0 to 2.7] | 2.1 [0.3 to 3.9] | 1.7 [0.1 to 3.3]
  Week 16: number analyzed (Participants) | 222 | 229 | 232
  Week 16 | 0.5 [0.0 to 1.3] | 2.2 [0.3 to 4.0] | 1.7 [0.1 to 3.3]
  Week 20: number analyzed (Participants) | 223 | 227 | 229
  Week 20 | 1.3 [0.0 to 2.8] | 1.7 [0.1 to 3.4] | 1.7 [0.1 to 3.4]
  Week 24: number analyzed (Participants) | 219 | 228 | 228
  Week 24 | 0.5 [0.0 to 1.4] | 1.7 [0.1 to 3.4] | 1.3 [0.0 to 2.7]
  Week 28: number analyzed (Participants) | 212 | 224 | 217
  Week 28 | 1.0 [0.0 to 2.4] | 1.3 [0.0 to 2.9] | 1.3 [0.0 to 2.8]
  Week 32: number analyzed (Participants) | 195 | 205 | 209
  Week 32 | 1.1 [0.0 to 2.5] | 1.0 [0.0 to 2.3] | 1.9 [0.1 to 3.7]
  Week 36: number analyzed (Participants) | 194 | 205 | 205
  Week 36 | 1.7 [0.0 to 3.5] | 1.0 [0.0 to 2.4] | 1.5 [0.0 to 3.1]
  Week 40: number analyzed (Participants) | 202 | 204 | 200
  Week 40 | 1.6 [0.0 to 3.3] | 2.0 [0.1 to 3.9] | 1.4 [0.0 to 3.0]
  Week 44: number analyzed (Participants) | 199 | 209 | 202
  Week 44 | 2.7 [0.4 to 4.9] | 2.0 [0.1 to 3.8] | 1.4 [0.0 to 2.9]
  Week 48: number analyzed (Participants) | 195 | 210 | 203
  Week 48 | 1.6 [0.0 to 3.4] | 2.4 [0.3 to 4.5] | 1.9 [0.1 to 3.7]
  Week 52: number analyzed (Participants) | 197 | 209 | 196
  Week 52 | 2.7 [0.4 to 5.0] | 1.9 [0.1 to 3.8] | 1.4 [0.0 to 3.0]
  Week 56: number analyzed (Participants) | 194 | 207 | 198
  Week 56 | 1.0 [0.0 to 2.5] | 1.5 [0.0 to 3.1] | 2.0 [0.1 to 3.9]
  Week 60: number analyzed (Participants) | 200 | 198 | 199
  Week 60 | 2.1 [0.1 to 4.1] | 1.0 [0.0 to 2.4] | 1.9 [0.1 to 3.8]
  Week 64: number analyzed (Participants) | 191 | 202 | 200
  Week 64 | 1.6 [0.0 to 3.5] | 2.0 [0.1 to 4.0] | 1.9 [0.1 to 3.7]
  Week 68: number analyzed (Participants) | 187 | 197 | 193
  Week 68 | 1.1 [0.0 to 2.7] | 1.6 [0.0 to 3.3] | 1.9 [0.1 to 3.7]
  Week 72: number analyzed (Participants) | 186 | 196 | 189
  Week 72 | 1.7 [0.0 to 3.6] | 1.0 [0.0 to 2.4] | 1.4 [0.0 to 3.0]
  Week 76: number analyzed (Participants) | 180 | 195 | 189
  Week 76 | 1.2 [0.0 to 2.8] | 1.5 [0.0 to 3.2] | 3.5 [1.0 to 6.0]
  Week 80: number analyzed (Participants) | 177 | 203 | 190
  Week 80 | 1.2 [0.0 to 2.8] | 2.0 [0.1 to 4.0] | 3.5 [1.0 to 6.0]
  Week 84: number analyzed (Participants) | 181 | 203 | 192
  Week 84 | 1.2 [0.0 to 2.8] | 1.0 [0.0 to 2.4] | 1.4 [0.0 to 2.9]
  Week 88: number analyzed (Participants) | 179 | 196 | 185
  Week 88 | 1.7 [0.0 to 3.7] | 1.0 [0.0 to 2.4] | 2.1 [0.1 to 4.2]
  Week 92: number analyzed (Participants) | 180 | 199 | 188
  Week 92 | 2.4 [0.1 to 4.6] | 1.5 [0.0 to 3.3] | 2.6 [0.3 to 4.9]
  Week 96: number analyzed (Participants) | 174 | 201 | 187
  Week 96 | 1.3 [0.0 to 3.0] | 2.1 [0.1 to 4.0] | 0.6 [0.0 to 1.7]
  Week 100: number analyzed (Participants) | 185 | 199 | 186
  Week 100 | 2.3 [0.1 to 4.5] | 2.1 [0.1 to 4.1] | 1.1 [0.0 to 2.6]

32. Secondary Outcome: Percentage of Participants With a ≥2-Step Diabetic Retinopathy Severity Improvement From Baseline on the ETDRS Diabetic Retinopathy Severity Scale in the Study Eye Over Time, ITT Population
Description: The Early Treatment Diabetic Retinopathy Study (ETDRS) Diabetic Retinopathy Severity Scale (DRSS) classifies diabetic retinopathy into 12 severity steps ranging from absence of retinopathy to advanced proliferative diabetic retinopathy. Ocular imaging assessments were made independently by a central reading center. The weighted estimates of the percentage of participants were based on the Cochran-Mantel Haenszel (CMH) weights stratified by baseline BCVA (≥64 vs. <64 letters), prior IVT anti-VEGF therapy (yes vs. no), and region (U.S. and Canada vs. rest of the world; Asia and rest of the world regions were combined). Treatment policy strategy (i.e., all observed values used) and hypothetical strategy (i.e., all values censored after the occurrence of the intercurrent event) were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were not imputed. 95% confidence interval (CI) is a rounding of 95.04% CI.
Time Frame: Baseline, Weeks 16, 52, and 96
Population: ITT Population: all participants who were randomized in the study, grouped according to the treatment assigned at randomization. Only participants with non-missing, valid assessments at Baseline and each timepoint were included in the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 315 | 313 | 312
Percentage of participants
  Week 16: number analyzed (Participants) | 279 | 291 | 281
  Week 16 | 36.7 [31.2 to 42.3] | 35.0 [29.6 to 40.5] | 28.9 [23.9 to 34.0]
  Week 52: number analyzed (Participants) | 249 | 253 | 236
  Week 52 | 46.2 [40.0 to 52.3] | 42.3 [36.4 to 48.3] | 35.4 [29.6 to 41.2]
  Week 96: number analyzed (Participants) | 220 | 234 | 221
  Week 96 | 51.4 [44.8 to 57.9] | 42.8 [36.6 to 49.0] | 42.2 [35.9 to 48.5]

33. Secondary Outcome: Percentage of Participants With a ≥2-Step Diabetic Retinopathy Severity Improvement From Baseline on the ETDRS Diabetic Retinopathy Severity Scale in the Study Eye Over Time, Treatment-Naive Population
Description: The Early Treatment Diabetic Retinopathy Study (ETDRS) Diabetic Retinopathy Severity Scale (DRSS) classifies diabetic retinopathy into 12 severity steps ranging from absence of retinopathy to advanced proliferative diabetic retinopathy. Ocular imaging assessments were made independently by a central reading center. The weighted estimates of the percentage of participants were based on the Cochran-Mantel Haenszel (CMH) weights stratified by baseline BCVA (≥64 vs. <64 letters) and region (U.S. and Canada vs. rest of the world; Asia and rest of the world regions were combined). Treatment policy strategy (i.e., all observed values used) and hypothetical strategy (i.e., all values censored after the occurrence of the intercurrent event) were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were not imputed. 95% confidence interval (CI) is a rounding of 95.04% CI.
Time Frame: Baseline, Weeks 16, 52, and 96
Population: Treatment-Naive Population: all participants randomized in the study who had not received any intravitreal anti-VEGF agents in the study eye prior to randomization. Participants were grouped according to the treatment assigned at randomization. Only participants with non-missing, valid assessments at Baseline and each timepoint were included in the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 238 | 245 | 242
Percentage of participants
  Week 16: number analyzed (Participants) | 209 | 225 | 219
  Week 16 | 39.3 [32.7 to 45.8] | 39.5 [33.2 to 45.9] | 33.3 [27.1 to 39.4]
  Week 52: number analyzed (Participants) | 182 | 196 | 184
  Week 52 | 49.5 [42.3 to 56.8] | 47.4 [40.5 to 54.4] | 42.3 [35.3 to 49.3]
  Week 96: number analyzed (Participants) | 159 | 178 | 169
  Week 96 | 52.3 [44.6 to 60.1] | 47.0 [39.7 to 54.2] | 49.1 [41.7 to 56.6]

34. Secondary Outcome: Percentage of Participants With a ≥3-Step Diabetic Retinopathy Severity Improvement From Baseline on the ETDRS Diabetic Retinopathy Severity Scale in the Study Eye Over Time, ITT Population
Description: as for outcome 32
Time Frame: Baseline, Weeks 16, 52, and 96
Population: as for outcome 32
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 315 | 313 | 312
Percentage of participants
  Week 16: number analyzed (Participants) | 279 | 291 | 281
  Week 16 | 12.7 [8.8 to 16.5] | 12.8 [9.0 to 16.6] | 10.3 [6.8 to 13.8]
  Week 52: number analyzed (Participants) | 249 | 253 | 236
  Week 52 | 17.0 [12.3 to 21.6] | 15.3 [10.9 to 19.8] | 14.2 [10.0 to 18.5]
  Week 96: number analyzed (Participants) | 220 | 234 | 221
  Week 96 | 22.4 [16.9 to 27.8] | 14.6 [10.0 to 19.1] | 20.9 [15.8 to 26.0]

35. Secondary Outcome: Percentage of Participants With a ≥3-Step Diabetic Retinopathy Severity Improvement From Baseline on the ETDRS Diabetic Retinopathy Severity Scale in the Study Eye Over Time, Treatment-Naive Population
Description: as for outcome 33
Time Frame: Baseline, Weeks 16, 52, and 96
Population: as for outcome 33
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 238 | 245 | 242
Percentage of participants
  Week 16: number analyzed (Participants) | 209 | 225 | 219
  Week 16 | 14.4 [9.7 to 19.1] | 15.1 [10.4 to 19.8] | 10.4 [6.4 to 14.4]
  Week 52: number analyzed (Participants) | 182 | 196 | 184
  Week 52 | 19.5 [13.7 to 25.2] | 17.4 [12.1 to 22.8] | 16.4 [11.2 to 21.6]
  Week 96: number analyzed (Participants) | 159 | 178 | 169
  Week 96 | 23.9 [17.3 to 30.5] | 17.1 [11.5 to 22.6] | 25.3 [18.9 to 31.6]

36. Secondary Outcome: Percentage of Participants With a ≥4-Step Diabetic Retinopathy Severity Improvement From Baseline on the ETDRS Diabetic Retinopathy Severity Scale in the Study Eye Over Time, ITT Population
Description: as for outcome 32
Time Frame: Baseline, Weeks 16, 52, and 96
Population: as for outcome 32
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 315 | 313 | 312
Percentage of participants
  Week 16: number analyzed (Participants) | 279 | 291 | 281
  Week 16 | 3.6 [1.4 to 5.8] | 3.5 [1.4 to 5.6] | 3.9 [1.7 to 6.2]
  Week 52: number analyzed (Participants) | 249 | 253 | 236
  Week 52 | 5.8 [2.9 to 8.7] | 4.9 [2.2 to 7.7] | 4.5 [1.9 to 7.0]
  Week 96: number analyzed (Participants) | 220 | 234 | 221
  Week 96 | 5.9 [2.8 to 9.0] | 5.8 [2.8 to 8.8] | 6.0 [3.0 to 9.0]

37. Secondary Outcome: Percentage of Participants With a ≥4-Step Diabetic Retinopathy Severity Improvement From Baseline on the ETDRS Diabetic Retinopathy Severity Scale in the Study Eye Over Time, Treatment-Naive Population
Description: as for outcome 33
Time Frame: Baseline, Weeks 16, 52, and 96
Population: as for outcome 33
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 238 | 245 | 242
Percentage of participants
  Week 16: number analyzed (Participants) | 209 | 225 | 219
  Week 16 | 3.9 [1.3 to 6.4] | 3.5 [1.1 to 5.9] | 3.6 [1.2 to 6.1]
  Week 52: number analyzed (Participants) | 182 | 196 | 184
  Week 52 | 6.2 [2.7 to 9.7] | 5.1 [2.0 to 8.3] | 4.2 [1.4 to 7.0]
  Week 96: number analyzed (Participants) | 159 | 178 | 169
  Week 96 | 7.0 [3.0 to 11.0] | 6.8 [3.1 to 10.5] | 6.3 [2.8 to 9.8]

38. Secondary Outcome: Percentage of Participants Without Proliferative Diabetic Retinopathy (PDR) at Baseline Who Developed New PDR at Week 52, ITT and Treatment-Naive Populations
Description: The Early Treatment Diabetic Retinopathy Study (ETDRS) Diabetic Retinopathy Severity Scale (DRSS) classifies diabetic retinopathy into 12 severity steps ranging from absence of retinopathy to advanced proliferative diabetic retinopathy (PDR). PDR was defined as an ETDRS DRSS score of ≥61 on the 7-field/4-wide field color fundus photographs assessment by a central reading center. The weighted percentages of participants were based on the Cochran-Mantel Haenszel (CMH) weights stratified by baseline BCVA (≥64 vs. <64 letters), prior IVT anti-VEGF therapy (yes vs. no), and region (U.S. and Canada vs. rest of the world; Asia and rest of the world regions were combined). Treatment policy strategy (i.e., all observed values used) and hypothetical strategy (i.e., all values censored after the occurrence of the intercurrent event) were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were not imputed. 95% CI is a rounding of 95.04% CI.
Time Frame: Baseline and Week 52
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 219 | 224 | 214
Percentage of participants
  ITT Population | 0.9 [0.0 to 2.2] | 0.9 [0.0 to 2.2] | 0.5 [0.0 to 1.4]
  Treatment-Naive Population: number analyzed (Participants) | 158 | 172 | 168
  Treatment-Naive Population | 0.0 [0.0 to 0.0] | 1.2 [0.0 to 2.8] | 0.6 [0.0 to 1.9]
Statistical Analysis 1: Comparison: A: Faricimab 6 mg Q8W vs C: Aflibercept 2 mg Q8W; [analysis description as in outcome 23, analysis 1]; Test type: Other; Difference in CMH Weighted Percentage = 0.4, 95% CI 2-sided [-1.1 to 2.0]
Statistical Analysis 2: Comparison: B: Faricimab 6 mg PTI vs C: Aflibercept 2 mg Q8W; [analysis description as in outcome 23, analysis 2]; Test type: Other; Difference in CMH Weighted Percentage = 0.4, 95% CI 2-sided [-1.1 to 2.0]
Statistical Analysis 3: Comparison: A: Faricimab 6 mg Q8W vs C: Aflibercept 2 mg Q8W; [analysis description as in outcome 23, analysis 3]; Test type: Other; Difference in CMH Weighted Percentage = -0.6, 95% CI 2-sided [-1.9 to 0.6]
Statistical Analysis 4: Comparison: B: Faricimab 6 mg PTI vs C: Aflibercept 2 mg Q8W; [analysis description as in outcome 23, analysis 4]; Test type: Other; Difference in CMH Weighted Percentage = 0.5, 95% CI 2-sided [-1.5 to 2.5]

39. Secondary Outcome: Percentage of Participants Without High-Risk Proliferative Diabetic Retinopathy (PDR) at Baseline Who Developed High-Risk PDR at Week 52, ITT and Treatment-Naive Populations
Description: The Early Treatment Diabetic Retinopathy Study (ETDRS) Diabetic Retinopathy Severity Scale (DRSS) classifies diabetic retinopathy into 12 severity steps ranging from absence of retinopathy to advanced PDR. High-risk PDR was defined as an ETDRS DRSS score of ≥71 on the 7-field/4-wide field color fundus photographs assessment by a central reading center. The weighted estimates of the percentage of participants were based on the Cochran-Mantel Haenszel (CMH) weights stratified by baseline BCVA (≥64 vs. <64 letters), prior IVT anti-VEGF therapy (yes vs. no), and region (U.S. and Canada vs. rest of the world; Asia and rest of the world regions were combined). Treatment policy strategy (i.e., all observed values used) and hypothetical strategy (i.e., all values censored after the occurrence of the intercurrent event) were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were not imputed. 95% CI is a rounding of 95.04% CI.
Time Frame: Baseline and Week 52
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 237 | 241 | 227
Percentage of participants
  ITT Population | 0.4 [0.0 to 1.2] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
  Treatment-Naive Population: number analyzed (Participants) | 173 | 187 | 177
  Treatment-Naive Population | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
Statistical Analysis 1: Comparison: A: Faricimab 6 mg Q8W vs C: Aflibercept 2 mg Q8W; [analysis description as in outcome 23, analysis 1]; Test type: Other; Difference in CMH Weighted Percentage = 0.4, 95% CI 2-sided [-0.4 to 1.2]
Statistical Analysis 2: Comparison: B: Faricimab 6 mg PTI vs C: Aflibercept 2 mg Q8W; [analysis description as in outcome 23, analysis 2]; Test type: Other; Difference in CMH Weighted Percentage = 0.0, 95% CI 2-sided [0.0 to 0.0]
Statistical Analysis 3: Comparison: A: Faricimab 6 mg Q8W vs C: Aflibercept 2 mg Q8W; [analysis description as in outcome 23, analysis 3]; Test type: Other; Difference in CMH Weighted Percentage = 0.0, 95% CI 2-sided [0.0 to 0.0]
Statistical Analysis 4: Comparison: B: Faricimab 6 mg PTI vs C: Aflibercept 2 mg Q8W; [analysis description as in outcome 23, analysis 4]; Test type: Other; Difference in CMH Weighted Percentage = 0.0, 95% CI 2-sided [0.0 to 0.0]

40. Secondary Outcome: Percentage of Participants in the Faricimab 6 mg PTI Arm on a Once Every 4-Weeks, 8-Weeks, 12-Weeks, or 16-Weeks Treatment Interval at Week 52, ITT Population
Time Frame: Week 52
Population: ITT Population: all participants who were randomized in the study, grouped according to the treatment assigned at randomization. The number analyzed includes all participants in Arm B: Faricimab 6 mg PTI who had not discontinued the study prior to Week 52.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | B: Faricimab 6 mg PTI
Number analyzed (Participants) | 286
Percentage of participants
  Once Every 4 Weeks | 10.8 [7.2 to 14.4]
  Once Every 8 Weeks | 15.4 [11.2 to 19.6]
  Once Every 12 Weeks | 21.0 [16.3 to 25.7]
  Once Every 16 Weeks | 52.8 [47.0 to 58.6]

41. Secondary Outcome: Percentage of Participants in the Faricimab 6 mg PTI Arm on a Once Every 4-Weeks, 8-Weeks, 12-Weeks, or 16-Weeks Treatment Interval at Week 52, Treatment-Naive Population
Time Frame: Week 52
Population: Treatment-Naive Population: all participants randomized in the study who had not received any intravitreal anti-VEGF agents in the study eye prior to randomization. Participants were grouped according to the treatment assigned at randomization. The number analyzed includes all participants in Arm B: Faricimab 6 mg PTI who had not discontinued the study prior to Week 52.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | B: Faricimab 6 mg PTI
Number analyzed (Participants) | 222
Percentage of participants
  Once Every 4 Weeks | 9.0 [5.2 to 12.8]
  Once Every 8 Weeks | 14.4 [9.8 to 19.0]
  Once Every 12 Weeks | 22.1 [16.6 to 27.5]
  Once Every 16 Weeks | 54.5 [47.9 to 61.1]

42. Secondary Outcome: Percentage of Participants in the Faricimab 6 mg PTI Arm on a Once Every 4-Weeks, 8-Weeks, 12-Weeks, or 16-Weeks Treatment Interval at Week 96, ITT Population
Time Frame: Week 96
Population: ITT Population: all participants who were randomized in the study, grouped according to the treatment assigned at randomization. The number analyzed includes all participants in Arm B: Faricimab 6 mg PTI who had not discontinued the study prior to Week 96.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | B: Faricimab 6 mg PTI
Number analyzed (Participants) | 270
Percentage of participants
  Once Every 4 Weeks | 7.0 [4.0 to 10.1]
  Once Every 8 Weeks | 14.8 [10.6 to 19.1]
  Once Every 12 Weeks | 18.1 [13.5 to 22.8]
  Once Every 16 Weeks | 60.0 [54.1 to 65.9]

43. Secondary Outcome: Percentage of Participants in the Faricimab 6 mg PTI Arm on a Once Every 4-Weeks, 8-Weeks, 12-Weeks, or 16-Weeks Treatment Interval at Week 96, Treatment-Naive Population
Time Frame: Week 96
Population: Treatment-Naive Population: all participants randomized in the study who had not received any intravitreal anti-VEGF agents in the study eye prior to randomization. Participants were grouped according to the treatment assigned at randomization. The number analyzed includes all participants in Arm B: Faricimab 6 mg PTI who had not discontinued the study prior to Week 96.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | B: Faricimab 6 mg PTI
Number analyzed (Participants) | 208
Percentage of participants
  Once Every 4 Weeks | 7.2 [3.7 to 10.7]
  Once Every 8 Weeks | 11.1 [6.8 to 15.3]
  Once Every 12 Weeks | 16.8 [11.7 to 21.9]
  Once Every 16 Weeks | 64.9 [58.4 to 71.4]

44. Secondary Outcome: Percentage of Participants in the Faricimab 6 mg PTI Arm at Week 52 Who Achieved a Once Every 12-Weeks or 16-Weeks Treatment Interval Without an Interval Decrease Below Once Every 12 Weeks, ITT and Treatment-Naive Populations
Time Frame: From start of PTI (Week 12 or later) until Week 52
Population: ITT Population and Treatment-Naive Population. The number analyzed includes all participants in Arm B: Faricimab 6 mg PTI who had not discontinued the study prior to Week 52.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | B: Faricimab 6 mg PTI
Number analyzed (Participants) | 286
Percentage of participants
  ITT Population | 67.8 [62.4 to 73.3]
  Treatment-Naive Population: number analyzed (Participants) | 222
  Treatment-Naive Population | 71.6 [65.7 to 77.6]

45. Secondary Outcome: Percentage of Participants in the Faricimab 6 mg PTI Arm at Week 96 Who Achieved a Once Every 12-Weeks or 16-Weeks Treatment Interval Without an Interval Decrease Below Once Every 12 Weeks, ITT and Treatment-Naive Populations
Time Frame: From start of PTI (Week 12 or later) until Week 96
Population: ITT Population and Treatment-Naive Population. The number analyzed includes all participants in Arm B: Faricimab 6 mg PTI who had not discontinued the study prior to Week 96.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | B: Faricimab 6 mg PTI
Number analyzed (Participants) | 270
Percentage of participants
  ITT Population | 60.4 [54.5 to 66.2]
  Treatment-Naive Population: number analyzed (Participants) | 208
  Treatment-Naive Population | 64.4 [57.9 to 70.9]

46. Secondary Outcome: Change From Baseline in Central Subfield Thickness in the Study Eye Averaged Over Weeks 48, 52, and 56, ITT and Treatment-Naive Populations
Description: Central subfield thickness (CST) was defined as the distance between the internal limiting membrane (ILM) and Bruch's membrane (BM) as assessed by a central reading center. For the Mixed Model for Repeated Measures (MMRM) analysis, the model adjusted for treatment group, visit, visit-by-treatment group interaction, baseline CST (continuous), baseline BCVA (<64 vs. ≥64 letters), prior intravitreal anti-VEGF therapy (yes vs. no), and region of enrollment (U.S. and Canada vs. the rest of the world; Asia and rest of the world regions were combined). An unstructured covariance structure was used. Treatment policy strategy (i.e., all observed values used) and hypothetical strategy (i.e., all values censored after the occurrence of the intercurrent event) were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were implicitly imputed by MMRM. 95% confidence interval (CI) is a rounding of 95.04% CI.
Time Frame: From Baseline through Week 56
Population: ITT Population and Treatment-Naive Population
Measure: Mean (95% Confidence Interval); unit: microns
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 315 | 313 | 312
microns
  ITT Population | -206.6 [-214.7 to -198.4] | -196.5 [-204.7 to -188.4] | -170.3 [-178.5 to -162.2]
  Treatment-Naive Population: number analyzed (Participants) | 238 | 245 | 242
  Treatment-Naive Population | -204.6 [-213.5 to -195.7] | -197.5 [-206.2 to -188.8] | -173.6 [-182.3 to -164.8]
Statistical Analysis 1: Comparison: A: Faricimab 6 mg Q8W vs C: Aflibercept 2 mg Q8W; This is the adjusted mean difference for Arm A: Faricimab 6 mg Q8W minus Arm C: Aflibercept 2 mg Q8W in the ITT Population; Test type: Other; Adjusted mean difference = -36.2, 95% CI 2-sided [-47.8 to -24.7], Standard Error of Mean 5.88
Statistical Analysis 2: Comparison: B: Faricimab 6 mg PTI vs C: Aflibercept 2 mg Q8W; This is the adjusted mean difference for Arm B: Faricimab 6 mg PTI minus Arm C: Aflibercept 2 mg Q8W in the ITT Population; Test type: Other; Adjusted mean difference = -26.2, 95% CI 2-sided [-37.7 to -14.7], Standard Error of Mean 5.86
Statistical Analysis 3: Comparison: A: Faricimab 6 mg Q8W vs C: Aflibercept 2 mg Q8W; This is the adjusted mean difference for Arm A: Faricimab 6 mg Q8W minus Arm C: Aflibercept 2 mg Q8W in the Treatment-Naive Population; Test type: Other; Adjusted mean difference = -31.1, 95% CI 2-sided [-43.6 to -18.6], Standard Error of Mean 6.35
Statistical Analysis 4: Comparison: B: Faricimab 6 mg PTI vs C: Aflibercept 2 mg Q8W; This is the adjusted mean difference for Arm B: Faricimab 6 mg PTI minus Arm C: Aflibercept 2 mg Q8W in the Treatment-Naive Population; Test type: Other; Adjusted mean difference = -23.9, 95% CI 2-sided [-36.2 to -11.6], Standard Error of Mean 6.28

47. Secondary Outcome: Change From Baseline in Central Subfield Thickness in the Study Eye Over Time, ITT Population
Description: as for outcome 46
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96, and 100
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: microns
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 315 | 313 | 312
microns
  Week 4 | -118.4 [-128.5 to -108.2] | -124.9 [-135.0 to -114.8] | -111.0 [-121.2 to -100.8]
  Week 8 | -145.9 [-155.2 to -136.5] | -149.6 [-159.0 to -140.3] | -130.9 [-140.4 to -121.5]
  Week 12 | -165.6 [-174.3 to -156.9] | -168.4 [-177.1 to -159.8] | -144.7 [-153.4 to -136.0]
  Week 16 | -177.6 [-186.0 to -169.2] | -182.1 [-190.4 to -173.7] | -152.7 [-161.1 to -144.3]
  Week 20 | -184.6 [-193.2 to -176.1] | -174.6 [-183.1 to -166.0] | -159.0 [-167.6 to -150.4]
  Week 24 | -196.4 [-204.8 to -188.0] | -192.8 [-201.2 to -184.3] | -146.3 [-154.7 to -137.8]
  Week 28 | -174.6 [-184.4 to -164.9] | -193.7 [-203.4 to -184.0] | -163.8 [-173.6 to -154.0]
  Week 32 | -200.2 [-209.4 to -191.0] | -181.6 [-190.8 to -172.4] | -147.2 [-156.4 to -138.0]
  Week 36 | -179.4 [-188.9 to -169.8] | -201.0 [-210.6 to -191.5] | -166.0 [-175.7 to -156.4]
  Week 40 | -205.1 [-214.5 to -195.7] | -193.5 [-203.0 to -184.1] | -153.9 [-163.4 to -144.4]
  Week 44 | -187.5 [-197.4 to -177.5] | -189.2 [-199.1 to -179.3] | -172.6 [-182.6 to -162.6]
  Week 48 | -209.7 [-218.6 to -200.8] | -194.8 [-203.7 to -185.8] | -163.2 [-172.2 to -154.3]
  Week 52 | -191.0 [-200.6 to -181.4] | -193.0 [-202.6 to -183.4] | -179.2 [-188.9 to -169.5]
  Week 56 | -212.4 [-221.5 to -203.4] | -200.3 [-209.3 to -191.2] | -164.4 [-173.5 to -155.2]
  Week 60 | -197.8 [-207.4 to -188.2] | -196.3 [-205.9 to -186.6] | -182.0 [-191.7 to -172.3]
  Week 64 | -214.9 [-224.0 to -205.9] | -199.9 [-208.9 to -190.8] | -171.5 [-180.6 to -162.4]
  Week 68 | -201.1 [-210.0 to -192.3] | -200.9 [-209.7 to -192.1] | -186.8 [-195.7 to -177.9]
  Week 72 | -216.2 [-224.9 to -207.6] | -201.6 [-210.3 to -193.0] | -182.3 [-191.1 to -173.6]
  Week 76 | -206.0 [-215.1 to -197.0] | -200.7 [-209.8 to -191.7] | -188.4 [-197.6 to -179.3]
  Week 80 | -219.1 [-227.7 to -210.5] | -203.2 [-211.7 to -194.6] | -184.5 [-193.2 to -175.9]
  Week 84 | -211.8 [-221.1 to -202.5] | -204.9 [-214.1 to -195.7] | -186.2 [-195.5 to -176.9]
  Week 88 | -218.6 [-228.0 to -209.3] | -204.1 [-213.4 to -194.8] | -183.7 [-193.1 to -174.3]
  Week 92 | -210.9 [-220.1 to -201.7] | -202.4 [-211.4 to -193.3] | -193.9 [-203.2 to -184.7]
  Week 96 | -224.0 [-232.9 to -215.1] | -203.8 [-212.6 to -195.1] | -194.7 [-203.6 to -185.8]
  Week 100 | -213.1 [-221.8 to -204.3] | -207.3 [-216.0 to -198.6] | -200.2 [-209.0 to -191.4]

48. Secondary Outcome: Change From Baseline in Central Subfield Thickness in the Study Eye Over Time, Treatment-Naive Population
Description: Central subfield thickness (CST) was defined as the distance between the internal limiting membrane (ILM) and Bruch's membrane (BM) as assessed by a central reading center. For the Mixed Model for Repeated Measures (MMRM) analysis, the model adjusted for treatment group, visit, visit-by-treatment group interaction, baseline CST (continuous), baseline BCVA (<64 vs. ≥64 letters), and region of enrollment (U.S. and Canada vs. the rest of the world; Asia and rest of the world regions were combined). An unstructured covariance structure was used. Treatment policy strategy (i.e., all observed values used) and hypothetical strategy (i.e., all values censored after the occurrence of the intercurrent event) were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were implicitly imputed by MMRM. 95% confidence interval (CI) is a rounding of 95.04% CI.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96, and 100
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: microns
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 238 | 245 | 242
microns
  Week 4 | -116.1 [-127.0 to -105.2] | -121.5 [-132.1 to -110.9] | -110.1 [-120.9 to -99.3]
  Week 8 | -142.9 [-153.0 to -132.8] | -147.4 [-157.3 to -137.5] | -131.5 [-141.5 to -121.5]
  Week 12 | -162.8 [-171.9 to -153.6] | -166.7 [-175.7 to -157.8] | -147.4 [-156.4 to -138.3]
  Week 16 | -175.1 [-183.8 to -166.3] | -181.7 [-190.3 to -173.1] | -155.9 [-164.5 to -147.2]
  Week 20 | -182.9 [-192.0 to -173.8] | -178.1 [-187.0 to -169.2] | -161.6 [-170.6 to -152.6]
  Week 24 | -194.2 [-203.4 to -184.9] | -191.1 [-200.2 to -182.0] | -149.7 [-158.9 to -140.6]
  Week 28 | -177.4 [-188.1 to -166.7] | -194.0 [-204.4 to -183.5] | -167.5 [-178.0 to -156.9]
  Week 32 | -196.4 [-206.6 to -186.2] | -183.7 [-193.7 to -173.8] | -150.2 [-160.3 to -140.2]
  Week 36 | -181.9 [-191.9 to -171.9] | -203.6 [-213.3 to -193.8] | -168.7 [-178.6 to -158.9]
  Week 40 | -198.9 [-209.7 to -188.1] | -192.1 [-202.8 to -181.4] | -157.4 [-168.2 to -146.5]
  Week 44 | -187.3 [-198.5 to -176.1] | -189.3 [-200.2 to -178.3] | -172.9 [-184.0 to -161.8]
  Week 48 | -207.3 [-217.3 to -197.3] | -194.9 [-204.7 to -185.1] | -165.0 [-174.9 to -155.1]
  Week 52 | -191.1 [-201.7 to -180.5] | -196.2 [-206.5 to -185.9] | -181.1 [-191.6 to -170.5]
  Week 56 | -210.4 [-220.0 to -200.8] | -200.9 [-210.3 to -191.5] | -171.0 [-180.6 to -161.4]
  Week 60 | -195.0 [-205.6 to -184.4] | -198.0 [-208.4 to -187.5] | -185.1 [-195.6 to -174.5]
  Week 64 | -213.7 [-223.5 to -203.9] | -199.2 [-208.8 to -189.6] | -175.3 [-184.9 to -165.6]
  Week 68 | -201.5 [-211.2 to -191.7] | -201.7 [-211.2 to -192.1] | -189.1 [-198.8 to -179.5]
  Week 72 | -215.9 [-225.5 to -206.4] | -203.2 [-212.5 to -193.9] | -184.1 [-193.5 to -174.6]
  Week 76 | -204.8 [-214.8 to -194.9] | -202.1 [-211.8 to -192.4] | -189.8 [-199.7 to -180.0]
  Week 80 | -217.3 [-227.0 to -207.5] | -202.2 [-211.6 to -192.7] | -186.2 [-195.9 to -176.6]
  Week 84 | -211.0 [-221.6 to -200.4] | -202.9 [-213.2 to -192.7] | -185.7 [-196.1 to -175.2]
  Week 88 | -215.9 [-226.4 to -205.5] | -205.2 [-215.3 to -195.0] | -186.4 [-196.7 to -176.1]
  Week 92 | -208.8 [-218.9 to -198.7] | -202.2 [-212.0 to -192.5] | -195.9 [-205.9 to -186.0]
  Week 96 | -221.0 [-231.4 to -210.7] | -199.0 [-209.0 to -189.1] | -196.7 [-206.9 to -186.6]
  Week 100 | -213.4 [-222.7 to -204.1] | -206.7 [-215.7 to -197.7] | -201.3 [-210.5 to -192.1]

49. Secondary Outcome: Percentage of Participants With Absence of Diabetic Macular Edema in the Study Eye Averaged Over Weeks 48, 52, and 56, ITT and Treatment-Naive Populations
Description: Absence of diabetic macular edema was defined as achieving a central subfield thickness (CST) of <325 microns in the study eye. CST was defined as the distance between the internal limiting membrane and Bruch's membrane. For each participant, an average CST value was calculated across the three visits, and this averaged value was then used to determine if the endpoint was met. The results were summarized as the percentage of participants per treatment arm who met the endpoint. The weighted estimates of the percentage of participants were based on the Cochran-Mantel Haenszel (CMH) weights stratified by baseline BCVA (≥64 vs. <64 letters), prior IVT anti-VEGF therapy (yes vs. no), and region (U.S. and Canada vs. rest of the world). Treatment policy strategy and hypothetical strategy were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were not imputed. 95% confidence interval (CI) is a rounding of 95.04% CI.
Time Frame: Average of Weeks 48, 52, and 56
Population: as for outcome 23
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 272 | 276 | 275
Percentage of participants
  ITT Population | 81.3 [76.8 to 85.9] | 78.0 [73.1 to 82.8] | 65.4 [59.9 to 70.8]
  Treatment-Naive Population: number analyzed (Participants) | 201 | 215 | 211
  Treatment-Naive Population | 83.5 [78.4 to 88.5] | 80.4 [75.1 to 85.7] | 68.3 [62.1 to 74.4]
Statistical Analysis 1: Comparison: A: Faricimab 6 mg Q8W vs C: Aflibercept 2 mg Q8W; [analysis description as in outcome 23, analysis 1]; Test type: Other; Difference in CMH Weighted Percentage = 16.0, 95% CI 2-sided [8.9 to 23.1]
Statistical Analysis 2: Comparison: B: Faricimab 6 mg PTI vs C: Aflibercept 2 mg Q8W; [analysis description as in outcome 23, analysis 2]; Test type: Other; Difference in CMH Weighted Percentage = 12.7, 95% CI 2-sided [5.4 to 20.0]
Statistical Analysis 3: Comparison: A: Faricimab 6 mg Q8W vs C: Aflibercept 2 mg Q8W; [analysis description as in outcome 23, analysis 3]; Test type: Other; Difference in CMH Weighted Percentage = 15.2, 95% CI 2-sided [7.3 to 23.2]
Statistical Analysis 4: Comparison: B: Faricimab 6 mg PTI vs C: Aflibercept 2 mg Q8W; [analysis description as in outcome 23, analysis 4]; Test type: Other; Difference in CMH Weighted Percentage = 12.5, 95% CI 2-sided [4.4 to 20.6]

50. Secondary Outcome: Percentage of Participants With Absence of Diabetic Macular Edema in the Study Eye Over Time, ITT Population
Description: Absence of diabetic macular edema was defined as achieving a central subfield thickness of <325 microns in the study eye. Central subfield thickness was defined as the distance between the internal limiting membrane (ILM) and Bruch's membrane (BM) as assessed by a central reading center. The weighted estimates of the percentage of participants were based on the Cochran-Mantel Haenszel (CMH) weights stratified by baseline BCVA (≥64 vs. <64 letters), prior IVT anti-VEGF therapy (yes vs. no), and region (U.S. and Canada vs. rest of the world; Asia and rest of the world regions were combined). Treatment policy strategy (i.e., all observed values used) and hypothetical strategy (i.e., all values censored after the occurrence of the intercurrent event) were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were not imputed. 95% confidence interval (CI) is a rounding of 95.04% CI.
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96, and 100
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 315 | 313 | 312
Percentage of participants
  Week 4: number analyzed (Participants) | 309 | 307 | 303
  Week 4 | 36.1 [30.8 to 41.4] | 41.3 [35.9 to 46.8] | 35.0 [29.7 to 40.4]
  Week 8: number analyzed (Participants) | 309 | 309 | 303
  Week 8 | 48.4 [42.9 to 54.0] | 52.7 [47.2 to 58.2] | 42.6 [37.1 to 48.2]
  Week 12: number analyzed (Participants) | 303 | 301 | 301
  Week 12 | 60.9 [55.4 to 66.4] | 67.4 [62.1 to 72.6] | 49.6 [44.0 to 55.2]
  Week 16: number analyzed (Participants) | 293 | 293 | 299
  Week 16 | 67.2 [61.8 to 72.5] | 72.0 [66.9 to 77.0] | 58.6 [53.1 to 64.1]
  Week 20: number analyzed (Participants) | 294 | 291 | 294
  Week 20 | 71.1 [65.9 to 76.2] | 70.7 [65.6 to 75.8] | 58.9 [53.4 to 64.5]
  Week 24: number analyzed (Participants) | 290 | 289 | 291
  Week 24 | 76.5 [71.7 to 81.4] | 81.3 [76.8 to 85.8] | 53.7 [48.1 to 59.4]
  Week 28: number analyzed (Participants) | 281 | 284 | 283
  Week 28 | 71.4 [66.2 to 76.5] | 79.3 [74.6 to 84.0] | 62.5 [57.0 to 68.0]
  Week 32: number analyzed (Participants) | 265 | 265 | 270
  Week 32 | 79.0 [74.2 to 83.8] | 72.1 [66.8 to 77.4] | 55.8 [50.1 to 61.5]
  Week 36: number analyzed (Participants) | 265 | 266 | 264
  Week 36 | 70.9 [65.6 to 76.1] | 81.7 [77.1 to 86.3] | 63.1 [57.4 to 68.8]
  Week 40: number analyzed (Participants) | 275 | 267 | 262
  Week 40 | 82.3 [77.9 to 86.7] | 80.8 [76.1 to 85.5] | 58.8 [53.0 to 64.7]
  Week 44: number analyzed (Participants) | 266 | 268 | 266
  Week 44 | 74.7 [69.6 to 79.9] | 79.0 [74.3 to 83.8] | 67.6 [62.1 to 73.1]
  Week 48: number analyzed (Participants) | 263 | 261 | 261
  Week 48 | 86.5 [82.5 to 90.5] | 81.5 [76.8 to 86.1] | 64.0 [58.3 to 69.7]
  Week 52: number analyzed (Participants) | 262 | 266 | 252
  Week 52 | 77.4 [72.4 to 82.4] | 78.3 [73.4 to 83.1] | 71.1 [65.6 to 76.7]
  Week 56: number analyzed (Participants) | 260 | 262 | 251
  Week 56 | 86.5 [82.4 to 90.7] | 81.3 [76.6 to 86.0] | 65.0 [59.2 to 70.8]
  Week 60: number analyzed (Participants) | 267 | 260 | 257
  Week 60 | 78.8 [74.0 to 83.6] | 79.4 [74.6 to 84.3] | 72.3 [66.9 to 77.7]
  Week 64: number analyzed (Participants) | 257 | 260 | 261
  Week 64 | 88.3 [84.4 to 92.2] | 80.0 [75.2 to 84.8] | 67.7 [62.1 to 73.3]
  Week 68: number analyzed (Participants) | 250 | 256 | 249
  Week 68 | 83.5 [79.0 to 88.1] | 84.1 [79.7 to 88.5] | 74.8 [69.4 to 80.1]
  Week 72: number analyzed (Participants) | 254 | 256 | 245
  Week 72 | 88.0 [84.0 to 92.0] | 85.2 [81.0 to 89.5] | 70.2 [64.5 to 75.9]
  Week 76: number analyzed (Participants) | 247 | 251 | 245
  Week 76 | 85.6 [81.3 to 89.8] | 84.9 [80.5 to 89.2] | 76.0 [70.7 to 81.2]
  Week 80: number analyzed (Participants) | 249 | 257 | 248
  Week 80 | 88.5 [84.5 to 92.4] | 81.9 [77.3 to 86.6] | 73.2 [67.7 to 78.7]
  Week 84: number analyzed (Participants) | 247 | 258 | 250
  Week 84 | 85.1 [80.7 to 89.5] | 86.1 [82.0 to 90.3] | 74.9 [69.5 to 80.3]
  Week 88: number analyzed (Participants) | 246 | 253 | 245
  Week 88 | 90.4 [86.8 to 94.0] | 83.2 [78.7 to 87.7] | 74.2 [68.7 to 79.6]
  Week 92: number analyzed (Participants) | 247 | 257 | 244
  Week 92 | 86.5 [82.3 to 90.7] | 78.2 [73.2 to 83.3] | 78.2 [73.1 to 83.3]
  Week 96: number analyzed (Participants) | 239 | 257 | 245
  Week 96 | 91.8 [88.4 to 95.3] | 83.7 [79.2 to 88.2] | 77.3 [72.1 to 82.4]
  Week 100: number analyzed (Participants) | 247 | 257 | 243
  Week 100 | 89.5 [85.7 to 93.4] | 85.9 [81.7 to 90.1] | 81.0 [76.1 to 86.0]

51. Secondary Outcome: Percentage of Participants With Retinal Dryness in the Study Eye Over Time, ITT Population
Description: Retinal dryness was defined as achieving a central subfield thickness (ILM-BM) of <280 microns. Central subfield thickness was defined as the distance between the internal limiting membrane (ILM) and Bruch's membrane (BM) as assessed by a central reading center. The weighted estimates of the percentage of participants was based on the Cochran-Mantel Haenszel (CMH) weights stratified by baseline BCVA (≥64 vs. <64 letters), prior IVT anti-VEGF therapy (yes vs. no), and region (U.S. and Canada vs. rest of the world; Asia and rest of the world regions were combined). Treatment policy strategy (i.e., all observed values used) and hypothetical strategy (i.e., all values censored after the occurrence of the intercurrent event) were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were not imputed. 95% confidence interval (CI) is a rounding of 95.04% CI.
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96, and 100
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 315 | 313 | 312
Percentage of participants
  Week 4: number analyzed (Participants) | 309 | 307 | 303
  Week 4 | 15.4 [11.5 to 19.4] | 16.0 [12.0 to 19.9] | 12.6 [8.9 to 16.3]
  Week 8: number analyzed (Participants) | 309 | 309 | 303
  Week 8 | 24.2 [19.6 to 28.8] | 24.6 [19.9 to 29.3] | 16.2 [12.1 to 20.3]
  Week 12: number analyzed (Participants) | 303 | 301 | 301
  Week 12 | 32.4 [27.3 to 37.5] | 34.1 [28.9 to 39.4] | 22.1 [17.4 to 26.7]
  Week 16: number analyzed (Participants) | 293 | 293 | 299
  Week 16 | 38.4 [33.0 to 43.9] | 42.5 [36.9 to 48.0] | 23.2 [18.5 to 27.9]
  Week 20: number analyzed (Participants) | 294 | 291 | 294
  Week 20 | 45.9 [40.3 to 51.5] | 40.6 [35.0 to 46.1] | 29.7 [24.5 to 34.8]
  Week 24: number analyzed (Participants) | 290 | 289 | 291
  Week 24 | 53.0 [47.3 to 58.7] | 48.1 [42.4 to 53.8] | 26.6 [21.6 to 31.6]
  Week 28: number analyzed (Participants) | 281 | 284 | 283
  Week 28 | 45.9 [40.1 to 51.7] | 50.2 [44.4 to 55.9] | 34.3 [28.8 to 39.8]
  Week 32: number analyzed (Participants) | 265 | 265 | 270
  Week 32 | 55.0 [49.1 to 60.8] | 43.2 [37.3 to 49.0] | 30.6 [25.1 to 36.1]
  Week 36: number analyzed (Participants) | 265 | 266 | 264
  Week 36 | 48.5 [42.5 to 54.5] | 54.3 [48.4 to 60.3] | 39.2 [33.4 to 45.1]
  Week 40: number analyzed (Participants) | 275 | 267 | 262
  Week 40 | 57.5 [51.8 to 63.2] | 51.3 [45.3 to 57.3] | 32.2 [26.7 to 37.7]
  Week 44: number analyzed (Participants) | 266 | 268 | 266
  Week 44 | 51.5 [45.7 to 57.4] | 51.9 [46.1 to 57.8] | 37.1 [31.4 to 42.8]
  Week 48: number analyzed (Participants) | 263 | 261 | 261
  Week 48 | 63.2 [57.4 to 69.0] | 50.1 [44.2 to 56.0] | 36.2 [30.4 to 42.0]
  Week 52: number analyzed (Participants) | 262 | 266 | 252
  Week 52 | 57.8 [51.9 to 63.7] | 54.7 [48.7 to 60.6] | 42.3 [36.2 to 48.4]
  Week 56: number analyzed (Participants) | 260 | 262 | 251
  Week 56 | 66.3 [60.6 to 72.0] | 56.9 [51.0 to 62.9] | 41.2 [35.1 to 47.2]
  Week 60: number analyzed (Participants) | 267 | 260 | 257
  Week 60 | 60.2 [54.4 to 66.0] | 54.0 [48.0 to 60.0] | 47.7 [41.6 to 53.7]
  Week 64: number analyzed (Participants) | 257 | 260 | 261
  Week 64 | 68.5 [62.8 to 74.1] | 55.4 [49.4 to 61.3] | 47.4 [41.3 to 53.4]
  Week 68: number analyzed (Participants) | 250 | 256 | 249
  Week 68 | 61.3 [55.3 to 67.3] | 57.7 [51.7 to 63.8] | 52.3 [46.1 to 58.5]
  Week 72: number analyzed (Participants) | 254 | 256 | 245
  Week 72 | 65.8 [60.1 to 71.5] | 58.5 [52.6 to 64.3] | 47.7 [41.4 to 53.9]
  Week 76: number analyzed (Participants) | 247 | 251 | 245
  Week 76 | 65.9 [60.1 to 71.8] | 54.8 [48.6 to 60.9] | 53.9 [47.7 to 60.1]
  Week 80: number analyzed (Participants) | 249 | 257 | 248
  Week 80 | 70.1 [64.5 to 75.8] | 54.7 [48.7 to 60.6] | 51.1 [44.8 to 57.3]
  Week 84: number analyzed (Participants) | 247 | 258 | 250
  Week 84 | 67.1 [61.3 to 72.9] | 61.2 [55.5 to 67.0] | 56.0 [49.9 to 62.2]
  Week 88: number analyzed (Participants) | 246 | 253 | 245
  Week 88 | 72.2 [66.7 to 77.7] | 58.0 [52.1 to 64.0] | 54.2 [48.0 to 60.5]
  Week 92: number analyzed (Participants) | 247 | 257 | 244
  Week 92 | 66.2 [60.5 to 72.0] | 58.0 [52.2 to 63.8] | 57.9 [51.7 to 64.0]
  Week 96: number analyzed (Participants) | 239 | 257 | 245
  Week 96 | 72.7 [67.2 to 78.2] | 61.4 [55.6 to 67.2] | 58.0 [51.8 to 64.2]
  Week 100: number analyzed (Participants) | 247 | 257 | 243
  Week 100 | 71.4 [65.9 to 76.8] | 60.5 [54.5 to 66.4] | 60.7 [54.5 to 66.8]

52. Secondary Outcome: Percentage of Participants With Absence of Intraretinal Fluid in the Study Eye Over Time, ITT Population
Description: Intraretinal fluid was measured using optical coherence tomography (OCT) in the central subfield (center 1 mm). The weighted estimates of the percentage of participants were based on the Cochran-Mantel Haenszel (CMH) weights stratified by baseline BCVA (≥64 vs. <64 letters), prior IVT anti-VEGF therapy (yes vs. no), and region (U.S. and Canada vs. rest of the world); Asia and rest of the world regions were combined due to a small number of enrolled participants. Treatment policy strategy (i.e., all observed values used) and hypothetical strategy (i.e., all values censored after the occurrence of the intercurrent event) were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were not imputed. 95% confidence interval (CI) is a rounding of 95.04% CI.
Time Frame: Baseline, Weeks 16, 48, 52, 56, 92, 96, and 100
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 315 | 313 | 312
Percentage of participants
  Week 16: number analyzed (Participants) | 289 | 293 | 298
  Week 16 | 16.3 [12.0 to 20.5] | 21.9 [17.1 to 26.6] | 13.4 [9.6 to 17.3]
  Week 48: number analyzed (Participants) | 262 | 261 | 263
  Week 48 | 45.6 [39.7 to 51.6] | 33.2 [27.5 to 38.9] | 21.9 [17.0 to 26.9]
  Week 52: number analyzed (Participants) | 262 | 261 | 249
  Week 52 | 42.1 [36.3 to 47.9] | 38.8 [32.9 to 44.7] | 25.5 [20.2 to 30.8]
  Week 56: number analyzed (Participants) | 254 | 256 | 254
  Week 56 | 49.3 [43.3 to 55.3] | 42.7 [36.7 to 48.7] | 23.7 [18.5 to 28.9]
  Week 92: number analyzed (Participants) | 242 | 251 | 241
  Week 92 | 58.5 [52.3 to 64.7] | 43.2 [37.1 to 49.3] | 33.2 [27.4 to 39.1]
  Week 96: number analyzed (Participants) | 232 | 254 | 241
  Week 96 | 63.1 [57.0 to 69.2] | 47.6 [41.5 to 53.7] | 34.6 [28.7 to 40.6]
  Week 100: number analyzed (Participants) | 238 | 251 | 237
  Week 100 | 61.4 [55.2 to 67.5] | 44.5 [38.4 to 50.7] | 37.6 [31.5 to 43.6]

53. Secondary Outcome: Percentage of Participants With Absence of Subretinal Fluid in the Study Eye Over Time, ITT Population
Description: Subretinal fluid was measured using optical coherence tomography (OCT) in the central subfield (center 1 mm). The weighted estimates of the percentage of participants were based on the Cochran-Mantel Haenszel (CMH) weights stratified by baseline BCVA (≥64 vs. <64 letters), prior IVT anti-VEGF therapy (yes vs. no), and region (U.S. and Canada vs. rest of the world); Asia and rest of the world regions were combined due to a small number of enrolled participants. Treatment policy strategy (i.e., all observed values used) and hypothetical strategy (i.e., all values censored after the occurrence of the intercurrent event) were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were not imputed. 95% confidence interval (CI) is a rounding of 95.04% CI.
Time Frame: Baseline, Weeks 16, 48, 52, 56, 92, 96, and 100
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 315 | 313 | 312
Percentage of participants
  Week 16: number analyzed (Participants) | 294 | 294 | 297
  Week 16 | 95.3 [92.9 to 97.7] | 94.5 [92.0 to 97.1] | 95.9 [93.7 to 98.2]
  Week 48: number analyzed (Participants) | 263 | 266 | 261
  Week 48 | 97.0 [95.0 to 99.0] | 95.5 [93.1 to 97.9] | 96.2 [93.8 to 98.5]
  Week 52: number analyzed (Participants) | 263 | 264 | 252
  Week 52 | 95.8 [93.3 to 98.2] | 95.4 [92.9 to 97.9] | 98.0 [96.2 to 99.7]
  Week 56: number analyzed (Participants) | 258 | 260 | 255
  Week 56 | 97.0 [95.0 to 99.0] | 97.0 [95.0 to 99.0] | 97.3 [95.3 to 99.3]
  Week 92: number analyzed (Participants) | 246 | 255 | 243
  Week 92 | 94.8 [92.1 to 97.6] | 94.5 [91.7 to 97.3] | 96.7 [94.5 to 99.0]
  Week 96: number analyzed (Participants) | 237 | 256 | 242
  Week 96 | 97.0 [94.8 to 99.1] | 94.1 [91.3 to 97.0] | 96.7 [94.5 to 98.9]
  Week 100: number analyzed (Participants) | 246 | 257 | 244
  Week 100 | 94.3 [91.4 to 97.2] | 97.3 [95.4 to 99.2] | 97.1 [95.0 to 99.2]

54. Secondary Outcome: Percentage of Participants With Absence of Intraretinal Fluid and Subretinal Fluid in the Study Eye Over Time, ITT Population
Description: Intraretinal fluid and subretinal fluid were measured using optical coherence tomography (OCT) in the central subfield (center 1 mm). The weighted estimates of the percentage of participants were based on the Cochran-Mantel Haenszel (CMH) weights stratified by baseline BCVA (≥64 vs. <64 letters), prior IVT anti-VEGF therapy (yes vs. no), and region (U.S. and Canada vs. rest of the world); Asia and rest of the world regions were combined due to a small number of enrolled participants. Treatment policy strategy (i.e., all observed values used) and hypothetical strategy (i.e., all values censored after the occurrence of the intercurrent event) were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were not imputed. 95% confidence interval (CI) is a rounding of 95.04% CI.
Time Frame: Baseline, Weeks 16, 48, 52, 56, 92, 96, and 100
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 315 | 313 | 312
Percentage of participants
  Week 16: number analyzed (Participants) | 290 | 293 | 298
  Week 16 | 15.9 [11.7 to 20.1] | 21.9 [17.1 to 26.6] | 13.1 [9.3 to 16.9]
  Week 48: number analyzed (Participants) | 262 | 261 | 263
  Week 48 | 45.2 [39.3 to 51.2] | 32.4 [26.8 to 38.1] | 21.9 [17.0 to 26.9]
  Week 52: number analyzed (Participants) | 262 | 261 | 249
  Week 52 | 42.1 [36.3 to 47.9] | 38.0 [32.2 to 43.8] | 25.5 [20.2 to 30.8]
  Week 56: number analyzed (Participants) | 254 | 256 | 254
  Week 56 | 47.0 [41.0 to 53.0] | 42.4 [36.4 to 48.3] | 23.7 [18.5 to 28.9]
  Week 92: number analyzed (Participants) | 242 | 251 | 241
  Week 92 | 57.2 [51.0 to 63.4] | 41.3 [35.2 to 47.3] | 32.0 [26.3 to 37.8]
  Week 96: number analyzed (Participants) | 232 | 254 | 241
  Week 96 | 62.4 [56.2 to 68.5] | 46.0 [39.8 to 52.1] | 34.2 [28.3 to 40.1]
  Week 100: number analyzed (Participants) | 238 | 251 | 238
  Week 100 | 59.3 [53.0 to 65.5] | 43.8 [37.6 to 49.9] | 37.4 [31.4 to 43.5]

55. Secondary Outcome: Change From Baseline in the National Eye Institute Visual Functioning Questionnaire-25 (NEI VFQ-25) Composite Score Over Time, ITT Population
Description: The NEI VFQ-25 captures a patient's perception of vision-related functioning and quality of life. The core measure includes 25 items that comprise 11 vision-related subscales and one item on general health. The composite score ranges from 0 to 100, with higher scores, or a positive change from baseline, indicating better vision-related functioning. For the Mixed Model for Repeated Measures (MMRM) analysis, the model adjusted for treatment arm, visit, visit-by-treatment arm interaction, baseline NEI VFQ-25 Composite Score (continuous), baseline BCVA (<64 vs. ≥64 letters), prior intravitreal anti-VEGF therapy (yes vs. no), and region of enrollment. An unstructured covariance structure was used. Treatment policy strategy and hypothetical strategy were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were implicitly imputed by MMRM. 95% CI is a rounding of 95.04% CI.
Time Frame: Baseline, Weeks 24, 52, and 100
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 315 | 313 | 312
score on a scale
  Week 24 | 6.0 [4.8 to 7.2] | 6.9 [5.7 to 8.1] | 6.0 [4.8 to 7.2]
  Week 52 | 7.3 [5.9 to 8.6] | 7.9 [6.6 to 9.3] | 7.5 [6.1 to 8.9]
  Week 100 | 8.0 [6.6 to 9.4] | 7.4 [6.0 to 8.8] | 7.6 [6.1 to 9.0]

56. Secondary Outcome: Percentage of Participants With at Least One Adverse Event
Description: This analysis of adverse events (AEs) includes both ocular and non-ocular (systemic) AEs. Investigators sought information on AEs at each contact with the participants. All AEs were recorded and the investigator made an assessment of seriousness, severity, and causality of each AE. AEs of special interest included the following: Cases of potential drug-induced liver injury that include an elevated ALT or AST in combination with either an elevated bilirubin or clinical jaundice, as defined by Hy's Law; Suspected transmission of an infectious agent by the study drug; Sight-threatening AEs that cause a drop in visual acuity (VA) score ≥30 letters lasting more than 1 hour, require surgical or medical intervention to prevent permanent loss of sight, or are associated with severe intraocular inflammation.
Time Frame: From first dose of study drug through end of study (up to 2 years)
Population: The safety-evaluable population comprised all participants who received at least one injection of active study drug (faricimab or aflibercept) in the study eye.
Measure: Number; unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 313 | 313 | 311
Percentage of participants
  Adverse Event (AE) | 92.7 | 91.4 | 89.1
  Serious AE (SAE) | 35.5 | 37.4 | 29.9
  AE Leading to Withdrawal from Study Treatment | 2.6 | 2.9 | 1.6
  AE of Special Interest (AESI) | 6.1 | 7.0 | 4.8

57. Secondary Outcome: Percentage of Participants With at Least One Ocular Adverse Event in the Study Eye or the Fellow Eye
Description: This analysis of adverse events (AEs) only includes ocular AEs, which are categorized as having occurred either in the study eye or the fellow eye. Investigators sought information on AEs at each contact with the participants. All AEs were recorded and the investigator made an assessment of seriousness, severity, and causality of each AE. Ocular AEs of special interest included the following: Suspected transmission of an infectious agent by the study drug; Sight-threatening AEs that cause a drop in visual acuity (VA) score ≥30 letters lasting more than 1 hour, require surgical or medical intervention to prevent permanent loss of sight, or are associated with severe intraocular inflammation.
Time Frame: From first dose of study drug through end of study (up to 2 years)
Population: as for outcome 56
Measure: Number; unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 313 | 313 | 311
Percentage of participants
  Study Eye: Adverse Event (AE) | 47.0 | 46.6 | 46.3
  Study Eye: Serious AE (SAE) | 3.8 | 4.5 | 2.3
  Study Eye: AE Leading to Withdrawal from Treatment | 1.3 | 1.9 | 0.3
  Study Eye: Treatment-related AE | 3.2 | 2.2 | 1.9
  Study Eye: Treatment-related SAE | 0.0 | 1.3 | 0.0
  Study Eye: AE of Special Interest (AESI) | 3.5 | 4.2 | 2.6
  Study Eye: AESI, Drop in VA Score ≥30 Letters | 2.6 | 2.2 | 2.3
  Study Eye: AESI, Associated with Severe IOI | 0.6 | 1.6 | 0.0
  Study Eye: AESI, Intervention Req. to Prevent Permanent Vision Loss | 1.0 | 1.3 | 0.3
  Fellow Eye: AE | 40.3 | 42.2 | 46.3
  Fellow Eye: SAE | 2.9 | 3.5 | 2.3
  Fellow Eye: AESI | 2.9 | 2.9 | 2.3
  Fellow Eye: AESI, Drop in VA Score ≥30 Letters | 2.2 | 1.9 | 1.3
  Fellow Eye: AESI, Associated with Severe IOI | 0.0 | 0.3 | 0.0
  Fellow Eye: AESI, Intervention Req. to Prevent Permanent Vision Loss | 1.0 | 1.3 | 1.0

58. Secondary Outcome: Percentage of Participants With at Least One Non-Ocular Adverse Event
Description: This analysis of adverse events (AEs) only includes non-ocular (systemic) AEs. Investigators sought information on adverse events (AEs) at each contact with the participants. All AEs were recorded and the investigator made an assessment of seriousness, severity, and causality of each AE. The non-ocular AE of special interest was: Cases of potential drug-induced liver injury that include an elevated ALT or AST in combination with either an elevated bilirubin or clinical jaundice, as defined by Hy's Law.
Time Frame: From first dose of study drug through end of study (up to 2 years)
Population: as for outcome 56
Measure: Number; unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 313 | 313 | 311
Percentage of participants
  Adverse Event (AE) | 76.7 | 80.2 | 77.8
  Serious AE (SAE) | 31.6 | 31.0 | 27.0
  AE Leading to Withdrawal from Study Treatment | 1.3 | 1.0 | 1.3
  AE of Special Interest (AESI) | 0.0 | 0.0 | 0.3
  AESI, Elevated ALT or AST with Either Elevated Bilirubin or Clinical Jaundice | 0.0 | 0.0 | 0.3

59. Secondary Outcome: Plasma Concentration of Faricimab Over Time
Description: Faricimab concentration in plasma was determined using a validated immunoassay method.
Time Frame: Pre-dose on Day 1 (Baseline); Weeks 4, 28, 52, 76, and 100
Population: This analysis only included participants in Arms A and B who received treatment with faricimab and with at least one plasma sample, provided sufficient dosing information (dose and dosing time) was available. The number of participants analyzed at a given timepoint includes those with an available plasma sample and dosing information at that timepoint.
Measure: Mean (Standard Deviation); unit: micrograms per millilitre (μg/mL)
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI
Number analyzed (Participants) | 313 | 311
micrograms per millilitre (μg/mL)
  Baseline: number analyzed (Participants) | 299 | 305
  Baseline | 0.0000 (0.0001) | 0.0000 (0.0001)
  Week 4: number analyzed (Participants) | 295 | 292
  Week 4 | 0.0211 (0.0337) | 0.0181 (0.0139)
  Week 28: number analyzed (Participants) | 261 | 266
  Week 28 | 0.0033 (0.0053) | 0.0089 (0.0145)
  Week 52: number analyzed (Participants) | 251 | 255
  Week 52 | 0.0052 (0.0104) | 0.0100 (0.0132)
  Week 76: number analyzed (Participants) | 229 | 228
  Week 76 | 0.0048 (0.0085) | 0.0068 (0.0255)
  Week 100: number analyzed (Participants) | 246 | 243
  Week 100 | 0.0052 (0.0087) | 0.0077 (0.0126)

60. Secondary Outcome: Percentage of Participants Who Test Positive for Treatment-Emergent Anti-Drug Antibodies Against Faricimab During the Study
Description: Anti-drug antibodies (ADAs) against fariciamb were detected in plasma using a validated bridging enzyme-linked immunosorbent assay (ELISA). The percentage of participants with treatment-emergent ADA-positive samples includes post-baseline evaluable participants with at least one treatment-induced (defined as having an ADA-negative sample or missing sample at baseline and any positive post-baseline sample) or treatment-boosted (defined as having an ADA-positive sample at baseline and any positive post-baseline sample with a titer that is equal to or greater than 4-fold baseline titer) ADA-positive sample during the study treatment period.
Time Frame: Baseline, Weeks 4, 28, 52, 76, and 100
Population: The analysis population consisted of all participants receiving faricimab with at least one determinant post-baseline ADA assessment.
Measure: Number; unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI
Number analyzed (Participants) | 310 | 311
Percentage of participants
  Total Treatment-Emergent ADA-Positive | 12.6 | 10.6
  Treatment-Induced ADA-Positive | 12.6 | 10.3
  Treatment-Boosted ADA-Positive | 0.0 | 0.3

ADVERSE EVENTS:
Time Frame: From Baseline until Week 100
Description: Adverse events (AEs) are reported for the safety population, which includes all participants who received at least one injection of active study drug (faricimab or aflibercept) in the study eye. For ocular AEs, the number of participants and events reported per term are combined totals of AEs that occurred in the study eye or the fellow eye.
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
All-Cause Mortality (participants affected / at risk) | 16/313 | 21/313 | 13/311
Serious Adverse Events (participants affected / at risk) | 111/313 | 117/313 | 93/311
Other Adverse Events (participants affected / at risk) | 161/313 | 163/313 | 163/311
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A: Faricimab 6 mg Q8W (N=313) | B: Faricimab 6 mg PTI (N=313) | C: Aflibercept 2 mg Q8W (N=311)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (5) | 2 (2)
Acute left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 5 (5) | 3 (3) | 4 (4)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2)
Arrhythmia (Cardiac disorders) | 1 (1) | 2 (2) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 3 (3) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 7 (12) | 3 (4) | 5 (6)
Cardiovascular disorder (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic left ventricular failure (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 2 (2) | 5 (5) | 4 (4)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 5 (5) | 5 (5)
Myocardial ischaemia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ventricular tachyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sudden hearing loss (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Vestibular disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Angle closure glaucoma (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 4 (4) | 3 (3) | 3 (3)
Diabetic retinal oedema (Eye disorders) | 2 (5) | 2 (2) | 2 (2)
Diabetic retinopathy (Eye disorders) | 4 (4) | 2 (2) | 2 (2)
Glaucoma (Eye disorders) | 2 (2) | 1 (1) | 0 (0)
Macular fibrosis (Eye disorders) | 0 (0) | 2 (2) | 1 (1)
Macular oedema (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Narrow anterior chamber angle (Eye disorders) | 1 (2) | 0 (0) | 0 (0)
Ocular hypertension (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Retinal artery occlusion (Eye disorders) | 0 (0) | 0 (0) | 2 (2)
Retinal haemorrhage (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Retinal neovascularisation (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Retinal tear (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Rhegmatogenous retinal detachment (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Uveitic glaucoma (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Uveitis (Eye disorders) | 0 (0) | 4 (5) | 0 (0)
Visual acuity reduced (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 3 (4) | 1 (1) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Diabetic gastroparesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 2 (2) | 0 (0) | 2 (2)
Death (General disorders) | 3 (3) | 5 (5) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) | 0 (0)
Generalised oedema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Ill-defined disorder (General disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Biliary dyskinesia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (2) | 0 (0) | 1 (1)
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 5 (5) | 10 (10) | 4 (4)
Cellulitis (Infections and infestations) | 4 (4) | 5 (5) | 4 (4)
Cellulitis gangrenous (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Cholecystitis infective (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Chorioretinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Complicated appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Diabetic foot infection (Infections and infestations) | 0 (0) | 1 (1) | 3 (3)
Diabetic gangrene (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Endophthalmitis (Infections and infestations) | 0 (0) | 4 (4) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infected bite (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Keratouveitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Kidney infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 3 (3) | 1 (1) | 7 (7)
Pneumonia (Infections and infestations) | 8 (10) | 4 (4) | 7 (7)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia escherichia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pseudomonal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 6 (6) | 0 (0) | 7 (7)
Sepsis syndrome (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (4) | 1 (1) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral keratouveitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cataract traumatic (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Corneal abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Ilium fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Blood potassium increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood testosterone increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Influenza A virus test positive (Investigations) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Diabetic complication (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (4) | 1 (1) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 4 (5) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 3 (3)
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Tumour invasion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 4 (6) | 4 (4)
Coma (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Hypertensive encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 4 (4) | 2 (2) | 2 (3)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 2 (3) | 1 (2) | 3 (3)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo CNS origin (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Device dislocation (Product Issues) | 1 (1) | 0 (0) | 0 (0)
Completed suicide (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Delusional disorder, unspecified type (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Disorientation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 2 (2) | 4 (4)
Chronic kidney disease (Renal and urinary disorders) | 2 (2) | 0 (0) | 4 (4)
End stage renal disease (Renal and urinary disorders) | 3 (3) | 0 (0) | 2 (2)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 5 (6) | 1 (1) | 3 (3)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 3 (3)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 3 (3)
Aortic stenosis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Blood pressure inadequately controlled (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 3 (4)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Varicose vein (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Anaemia of chronic disease (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Blood loss anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular block (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Congestive cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cataract subcapsular (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Ocular ischaemic syndrome (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Retinal vein occlusion (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Tractional retinal detachment (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Complication associated with device (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cyst (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperpyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 3 (3) | 3 (3)
Coronavirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gangrene (Infections and infestations) | 1 (1) | 4 (4) | 2 (2)
Norovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Suspected COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Foreign body in throat (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Posterior capsule rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Skull fractured base (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 2 (2) | 0 (0)
Hyperosmolar state (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Cerebral microinfarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Lacunar infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Ruptured cerebral aneurysm (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Toxic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Device malfunction (Product Issues) | 1 (1) | 0 (0) | 0 (0)
Delusion (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Coronary artery bypass (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Circulatory collapse (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertensive urgency (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral artery aneurysm (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral artery stenosis (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A: Faricimab 6 mg Q8W (N=313) | B: Faricimab 6 mg PTI (N=313) | C: Aflibercept 2 mg Q8W (N=311)
Cataract (Eye disorders) | 58 (84) | 47 (65) | 55 (82)
Conjunctival haemorrhage (Eye disorders) | 25 (35) | 33 (41) | 24 (32)
Diabetic retinal oedema (Eye disorders) | 20 (27) | 29 (37) | 33 (40)
Vitreous detachment (Eye disorders) | 20 (25) | 23 (28) | 13 (16)
Nasopharyngitis (Infections and infestations) | 27 (31) | 18 (23) | 30 (39)
Hypertension (Vascular disorders) | 22 (27) | 32 (34) | 36 (38)
Vitreous floaters (Eye disorders) | 17 (25) | 11 (13) | 10 (13)
Urinary tract infection (Infections and infestations) | 14 (23) | 15 (17) | 19 (22)
Fall (Injury, poisoning and procedural complications) | 16 (16) | 19 (20) | 9 (9)
Intraocular pressure increased (Investigations) | 17 (28) | 13 (25) | 11 (13)

LIMITATIONS AND CAVEATS:
All secondary outcome measures were unpowered for statistical analysis, and the results should be interpreted with caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2019-06-20): https://cdn.clinicaltrials.gov/large-docs/80/NCT03622580/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-15): https://cdn.clinicaltrials.gov/large-docs/80/NCT03622580/SAP_001.pdf